Official Title:

An Open-Label, Multinational, Multicenter, Phase IIIB Study to Assess Safety of Rituximab Following Subcutaneous Administration in Patients With CD20+ DLBCL or CD20+ Follicular NHL Grade 1 to

3A

NCT Number: NCT02406092

**Document Date:** SAP Version 1: 04-January-2022

#### STATISTICAL ANALYSIS PLAN

TITLE: AN OPEN-LABEL, MULTINATIONAL, MULTICENTER,

PHASE IIIB STUDY TO ASSESS SAFETY OF RITUXIMAB FOLLOWING SUBCUTANEOUS ADMINISTRATION IN PATIENTS WITH CD20+ DLBCL OR CD20+ FOLLICULAR

**NHL GRADE 1 TO 3A** 

PROTOCOL NUMBER: ML28964

STUDY DRUG: Rituximab

**VERSION NUMBER:** 1.0

IND NUMBER: N/A

**EUDRACT NUMBER:** N/A

**SPONSOR:** Roche Algeria

PLAN PREPARED BY:

SPARC Consulting (on behalf of IQVIA), Milan - Italy

**DATE FINAL:** See electronic date stamp below

**DATE(S) AMENDED:** N/A

STATISTICAL ANALYSIS PLAN APPROVAL

[This space is reserved for the electronic signature]

#### **CONFIDENTIAL**

This is F. Hoffmann-La Roche Ltd local affiliates document that contains confidential information. Nothing herein is to be disclosed without written consent from F. Hoffmann-La Roche Ltd.

Rituximab - Roche North Africa (Algeria, Morocco & Tunisia) Mabrella ML28964 Daughter Protocol Statistical Analysis Plan ML28964

# STATISTICAL ANALYSIS PLAN HISTORY

| Version | Date Release |
|---------|--------------|
| 0.1 | 15DEC2021 |
| 0.2 | 22DEC2021 |
| 1.0 | 04JAN2022 |

# **TABLE OF CONTENTS**

| ST | ATISTICAL A | ANALYSIS PLAN HISTORY | 2 |
|----|-------------|-------------------------------------------------|----|
| 1. | BACKGRO | OUND | 21 |
| 2. | STUDY DE | ESIGN | 21 |
| | 2.1 | Protocol Synopsis | 22 |
| | 2.2 | Outcome Measures | 22 |
| | 2.2.1 | Safety Outcome Measures | 22 |
| | 2.2.2 | Efficacy Outcome Measures | 22 |
| | 2.2.3 | Exploratory Outcome Measures | 23 |
| | 2.2.4 | Pharmacokinetic Outcome Measures | 23 |
| | 2.3 | Determination of Sample Size | 23 |
| | 2.3.1 | Sample Size for the China Extension Period | 23 |
| | 2.4 | Analysis Timing | 24 |
| | 2.4.1 | Analysis Timing for the China Subgroup Analysis | 24 |
| 3. | STUDY CO | ONDUCT | 24 |
| | 3.1 | Randomization | 24 |
| | 3.2 | Independent Review Facility | 24 |
| | 3.3 | Data Monitoring | 24 |
| 4. | STATISTIC | CAL METHODS | 24 |
| | 4.1 | Analysis Populations | 25 |
| | 4.1.1 | Randomized Population | 25 |
| | 4.1.2 | Per Protocol Population | 25 |
| | 4.1.3 | Pharmacokinetic-Evaluable Population | 25 |
| | 4.1.4 | Safety Population | 25 |
| | 4.1.5 | Intent-To-Treat Population | 26 |
| | 4.2 | Analysis of Study Conduct | 26 |
| | 4.2.1 | Definition of Baseline | 26 |
| | 4.3 | Analysis of Treatment Group Comparability | 26 |
| | 4.3.1 | Medical History | 26 |
| | 4.3.2 | Surgery and Procedures History | 27 |
| | 4.3.3 | Physical Examination | 27 |

| | 4.3.4 | Previous and Concomitant Therapies | 27 |
|---|---|---|---|
| | 4.3.5 | Viral Serology | 28 |
| | 4.4 | Efficacy Analysis | 28 |
| | 4.4.1 | Primary Efficacy Endpoint | 29 |
| | 4.4.2 | Secondary Efficacy Endpoints | 29 |
| | 4.4.3 | Exploratory Efficacy Endpoints | 30 |
| | 4.4.4 | Sensitivity Analyses | 30 |
| | 4.4.5 | Subgroup Analyses | 30 |
| | 4.5 | Pharmacokinetic and Pharmacodynamic Analyses | 30 |
| | 4.6 | Patient-Reported Outcome Analyses | 30 |
| | 4.7 | Healthcare Professional Reported Outcome Analyses | 31 |
| | 4.8 | Safety Analyses | 32 |
| | 4.8.1 | Exposure of Study Medication | 32 |
| | 4.8.2 | Adverse Events | 32 |
| | 4.8.3 | Laboratory Data | 36 |
| | 4.8.4 | Vital Signs | 36 |
| | 4.8.5 | ECOG Performance Status | 36 |
| | 4.9 | Missing Data | 36 |
| | 4.10 | Interim Analyses | 37 |
| 5. | CHINA SUB | GROUP ANALYSIS | 38 |
| 6. | REFERENC | ES | 39 |
| | Appendix 1 - | - Protocol Synopsis | 46 |
| | Appendix 2 - | - Schedule of Assessments | 54 |
| | Appendix 3 - | - Table and Listing Shells | 60 |
| | TABLE 14. | 1.1. ENROLLED BY COUNTRY AND SITE (ITT POPULATION) | 61 |
| | TABLE 14. | 1.2. SUMMARY OF PATIENT DISPOSITION (ITT POPULATION) | 62 |
| | TABLE 14. | 1.3. SUMMARY OF PROTOCOL DEVIATIONS (ITT POPULATION) | 63 |
| | TABLE 14. | 1.4. SUMMARY OF DEMOGRAPHICS (ITT POPULATION) | 64 |

| TABLE | 14.1.5. SERUM PREGNANCY TEST AT SCREENING (SAFETY POPULATION) | . 65 |
|---|---|---|
| TABLE | 14.1.6. SUMMARY OF BASELINE CHARACTERISTICS - PART #1 (ITT POPULATION) | . 66 |
| TABLE | 14.1.7. SUMMARY OF BASELINE CHARACTERISTICS - PART #2 (ITT POPULATION) | . 67 |
| TABLE | 14.1.8. DLBCL DIAGNOSIS (SAFETY POPULATION) | . 68 |
| TABLE | 14.1.9. FOLLICULAR LYMPHOMA DIAGNOSIS (SAFETY POPULATION) | . 69 |
| TABLE | 14.1.10. SUMMARY OF BONE MARROW AT BASELINE (ITT POPULATION) | . 70 |
| TABLE | 14.1.11. LEAD ECG AT SCREENING (SAFETY POPULATION) | . 71 |
| TABLE | 14.1.12. VIRAL SEROLOGY AT SCREENING (SAFETY POPULATION) | |
| TABLE | 14.1.13. SUMMARY OF PREVIOUS DISEASE (ITT POPULATION) | |
| TABLE | 14.1.14. SUMMARY OF CONCOMITANT DISEASE (ITT POPULATION) | |
| TABLE | 14.1.15. SUMMARY OF PHYSICAL EXAMINATION (SAFETY POPULATION) | |
| TABLE | 14.1.16. SUMMARY OF PREVIOUS THERAPIES (SAFETY POPULATION) | |
| TABLE | 14.1.17. SUMMARY OF CONCOMITANT THERAPIES (SAFETY POPULATION) | |
| TABLE | 14.1.18. SUMMARY OF PREVIOUS IV RITUXIMAB DOSE FOR DLBCL (SAFETY POPULATION) | |
| TABLE | 14.1.19. SUMMARY OF PREVIOUS IV RITUXIMAB DOSE FOR FL (SAFETY POPULATION) | |
| TABLE | 14.1.20. EXPOSURE TO RITUXIMAB SC - ADMINISTRATION SUMMARY (SAFETY | . , . |
| m 7 - 7 - 7 | POPULATION) | . 80 |
| TABLE | 14.1.21. EXPOSURE TO RITUXIMAB SC - ADMINISTRATION DETAILS (SAFETY POPULATION) | 81 |

| TABLE 14.1.22. EXPOSURE TO RITUXIMAB SC - ADMINISTRATION DETAILS (SAFETY | |
|---|---|
| POPULATION) | 82 |
| TABLE 14.1.23. TYPE OF CHEMOTHERAPY (SAFETY POPULATION) | 83 |
| TABLE 14.1.24. EXPOSURE TO CHEMOTHERAPY (SAFETY POPULATION) | 84 |
| TABLE 14.1.25. EXPOSURE TO NEW ANTI - LYMPHOMA TREATMENT CHEMO/IMMUNO THERAPY (SAFETY POPULATION) | 85 |
| TABLE 14.1.26. INITIAL CHOP REGIMEN DOSAGE (SAFETY POPULATION) | 86 |
| TABLE 14.1.27. INITIAL CVP REGIMEN DOSAGE (SAFETY POPULATION) | 87 |
| TABLE 14.1.28. INITIAL FLUDARABINE DOSAGE (SAFETY POPULATION) | 88 |
| TABLE 14.1.29. EXPOSURE TO NEW ANTI - LYMPHOMA TREATMENT RADIOTHERAPY (SAFETY POPULATION) | 89 |
| TABLE 14.2.1. OVERALL SUMMARY OF PATIENTS EXPERIENCING EACH CLASS OF TREATMENT EMERGENT ADVERSE EVENT (SAFETY POPULATION) | 90 |
| TABLE 14.2.2. PROPORTION OF TREATMENT EMERGENT ADVERSE EVENT BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 91 |
| TABLE 14.2.3. PROPORTION OF SERIOUS TREATMENT EMERGENT ADVERSE EVENT BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 92 |
| TABLE 14.2.4. PROPORTION OF LOCALIZED ADMINISTRATION ASSOCIATED REACTIONS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | |
| TABLE 14.2.5. PROPORTION OF NON-LOCALIZED ADMINISTRATION ASSOCIATED REACTIONS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 94 |

| 95 | TABLE 14.2.6. PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ AES BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) |
|---|---|
| | TABLE 14.2.7. PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ SAES BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) |
| 97 | TABLE 14.2.8. PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ AARS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) |
| 98 | TABLE 14.2.9. PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO RITUXIMAB DRUG INTERRUPTED/DRUG DELAYED BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) |
| | TABLE 14.2.10. PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO RITUXIMAB DOSE DISCONTINUATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) |
| 100 | TABLE 14.2.11. PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO CHEMOTHERAPY DOSE MODIFICATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) |
| 101 | TABLE 14.2.12. PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO CHEMOTHERAPY DOSE DISCONTINUATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) |
| 102 | TABLE 14.2.13. PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO DEATH BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) |
| 103 | TABLE 14.2.14. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) |
| | TABLE 14.2. <b>15</b> . SUMMARY OF SERIOUS TREATMENT-<br>EMERGENT ADVERSE EVENTS BY SYSTEM |

| | ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 104 |
|---|---|---|
| TABLE | 14.2.16. SUMMARY OF ADVERSE EVENTS OF SPECIAL INTEREST BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 105 |
| TABLE | 14.2.17. SUMMARY OF ADMINISTRATION ASSOCIATED REACTIONS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 106 |
| TABLE | 14.2.18. SUMMARY OF INFUSION/INJECTION-<br>RELATED REACTIONS BY SYSTEM ORGAN<br>CLASS AND PREFERRED TERM (SAFETY<br>POPULATION) | 107 |
| TABLE | 14.2.19. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ AES BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 108 |
| TABLE | 14.2.20. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ SAES BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 109 |
| TABLE | 14.2.21. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ AESI BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 110 |
| TABLE | 14.2.22. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ AARS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 111 |
| TABLE | 14.2.23. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ IIRRS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 112 |
| TABLE | 14.2.24. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITHIN THE MEDDRA SMQ `ANAPHYLACTIC REACTIONS' (WIDE) BY SYSTEM ORGAN CLASS AND PREFERRED | 440 |
| TABLE | TERM (SAFETY POPULATION) | 113 |

Rituximab - Roche North Africa (Algeria, Morocco & Tunisia) Mabrella ML28964 Daughter Protocol 8/Statistical Analysis Plan ML28964

| | SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 114 |
|---|---|---|
| TABLE | 14.2.26. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO RITUXIMAB DOSE DISCONTINUATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 115 |
| TABLE | 14.2.27. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO CHEMOTHERAPY DOSE MODIFICATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 116 |
| TABLE | 14.2.28. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO CHEMOTHERAPY DOSE DISCONTINUATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 117 |
| TABLE | 14.2.29. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO DEATH BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 118 |
| TABLE | 14.2.30. SUMMARY OF CUTANEOUS AND SOFT TISSUE AARS (LOCALIZED) BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 119 |
| TABLE | 14.2.31. SUMMARY OF CUTANEOUS AND SOFT TISSUE AARS (NON-LOCALIZED) BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 120 |
| TABLE | 14.2.32. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH AN INCIDENCE OF >=5% BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION) | 121 |
| TABLE | 14.2.33. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM AND MAXIMUM SEVERITY (SAFETY POPULATION) | 122 |
| TABLE | 14.2.34. SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM AND STRONGEST RELATIONSHIP (SAFETY POPULATION) | |

| TABLE | 14.2.35. SUMMARY OF NON-SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS WITH AN INCIDENCE OF >=5% BY SYSTEM ORGAN CLASS AND PREFERRED TERM | |
|---|---|---|
| | (SAFETY POPULATION) | 124 |
| TABLE | 14.2.36. SUMMARY OF PATIENTS DEAD OVER THE STUDY (SAFETY POPULATION) | 125 |
| TABLE | 14.3.1. SUMMARY OF HEMATOLOGY PARAMETERS OVER THE STUDY (SAFETY POPULATION) | 126 |
| TABLE | 14.3.2. SUMMARY OF BLOOD CHEMISTRY PARAMETERS OVER THE STUDY (SAFETY POPULATION) | 127 |
| TABLE | 14.3.3. SUMMARY OF COAGULATION TESTS OVER THE STUDY (SAFETY POPULATION) | 128 |
| TABLE | 14.3.4. SHIFT TABLE OF HEMATOLOGY PARAMETERS ACCORDING TO NCI CTCAE WORST GRADE RECORDED DURING THE TREATMENT PERIOD (SAFETY POPULATION) | 129 |
| TABLE | 14.3.5. SHIFT TABLE OF BLOOD CHEMISTRY PARAMETERS ACCORDING TO NCI CTCAE WORST GRADE RECORDED DURING THE TREATMENT PERIOD (SAFETY POPULATION) | 130 |
| TABLE | 14.3.6. SHIFT TABLE OF COAGULATION TESTS ACCORDING TO NCI CTCAE WORST GRADE RECORDED DURING THE TREATMENT PERIOD (SAFETY POPULATION) | 131 |
| TABLE | 14.3.7. SUMMARY OF VITAL SIGNS OVER THE STUDY (SAFETY POPULATION) | |
| TABLE | 14.3.8. ECOG PERFORMANCE STATUS (SAFETY POPULATION) | 133 |
| TABLE | 14.4.1. TARGET LESION ASSESSMENT AT SCREENING (PART #1) (SAFETY POPULATION) | 134 |
| TABLE | 14.4.2. TARGET LESION ASSESSMENT AT SCREENING (PART #2) (SAFETY POPULATION) | 135 |
| TABLE | 14.4.3. POST-SCREENING TARGET LESION ASSESSMENT (PART #1) (SAFETY POPULATION) | |

| | 14.4.4. POST-SCREENING TARGET LESION ASSESSMENT (PART #2) (SAFETY | TABLE |
|---|---|---|
| | POPULATION) | |
| | 14.4.5. OVERALL LESION ASSESSMENT (SAFETY POPULATION) | TABLE |
| 139 | 14.5.1. OVERALL SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV (ITT POPULATION) | TABLE |
| 140 | 14.5.2. OVERALL SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION (ITT POPULATION) | TABLE |
| 141 | 14.5.3. OVERALL SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION CURVE FOR ALL SUBJECTS (ITT POPULATION) | TABLE |
| 142 | 14.5.4. OVERALL SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION CURVE by TYPE OF LYMPHOMA (ITT POPULATION) | TABLE |
| 143 | 14.5.5. PROGRESSION FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV (ITT POPULATION) | TABLE |
| 144 | 14.5.6. PROGRESSION FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION (ITT POPULATION) | TABLE |
| 145 | 14.5.7. PROGRESSION FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION CURVE FOR ALL SUBJECTS (ITT POPULATION) | TABLE |
| 146 | 14.5.8. PROGRESSION FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION CURVE by TYPE OF LYMPHOMA (ITT POPULATION) | TABLE |
| 147 | 14.5.9. DISEASE FREE SURVIVAL (ITT POPULATION) | TABLE |
| | 14.5.10. DISEASE FREE SURVIVAL: DISTRIBUCTION FUNCTION (ITT POPULATION) | TABLE |
| | 14.5.11. DISEASE FREE SURVIVAL: DISTRIBUCTION FUNCTION CURVE FOR ALL SUBJECTS (ITT POPULATION) | TABLE |

| 150 | 14.5.12. DISEASE FREE SURVIVAL: DISTRIBUCTION FUNCTION CURVE by TYPE OF LYMPHOMA (ITT POPULATION) | TABLE |
|---|---|---|
| , | 14.5.13. EVENT FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV (ITT POPULATION | TABLE |
| | 14.5.14. EVENT FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION (ITT POPULATION) | TABLE |
| 450 | 14.5.15. EVENT FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION CURVE FOR ALL SUBJECTS (ITT | TABLE |
| | POPULATION) | TABLE |
| | (ITT POPULATION) | TABLE |
| | 14.6.1. RITUXIMAB IV ADMINISTRATION SATIFICATION QUESTIONNAIRE - ITEMS FREQUENCY ANALYSIS (SAFETY POPULATION) | TABLE |
| 157 | 14.6.2. RITUXIMAB SC ADMINISTRATION SATIFICATION QUESTIONNAIRE - ITEMS FREQUENCY ANALYSIS (SAFETY POPULATION) | TABLE |
| 158 | 14.6.3. SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE IV MEAN SCORES (SAFETY POPULATION) | TABLE |
| 159 | 14.6.4. SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE IV MEAN SCORES (SAFETY POPULATION) | TABLE |
| 160 | 14.6.5. SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE IV MEAN SCORES (SAFETY | TABLE |

| TABLE 14.6.6. SUMMARY OF RITUXIMAE ADMINISTRATION SATISFAC | TION | |
|---|---|---|
| QUESTIONNAIRE IV MEAN S POPULATION) | • | 31 |
| TABLE 14.6.7. SUMMARY OF RITUXIMAE ADMINISTRATION SATISFAC QUESTIONNAIRE IV MEAN S POPULATION) | TION<br>CORES (SAFETY | 32 |
| TABLE 14.6.8. SUMMARY OF RITUXIMAE ADMINISTRATION SATISFAC QUESTIONNAIRE SC MEAN S POPULATION) | TION<br>CORES (SAFETY | 33 |
| TABLE 14.6.9. SUMMARY OF RITUXIMAE ADMINISTRATION SATISFAC QUESTIONNAIRE SC MEAN S POPULATION) | TION<br>CORES (SAFETY | 64 |
| TABLE 14.6.10. SUMMARY OF RITUXIMA ADMINISTRATION SATISFAC QUESTIONNAIRE SC MEAN S POPULATION) | TION<br>CORES (SAFETY | 35 |
| TABLE 14.6.11. SUMMARY OF RITUXIMA ADMINISTRATION SATISFAC QUESTIONNAIRE SC MEAN S POPULATION) | TION<br>CORES (SAFETY | 36 |
| TABLE 14.6.12. SUMMARY OF RITUXIMA ADMINISTRATION SATISFAC QUESTIONNAIRE SC MEAN S POPULATION) | TION<br>CORES (SAFETY | 67 |
| TABLE 14.6.13. HEALTHCARE PROFESSI QUESTIONNAIRE (PART #1) | | 38 |
| TABLE 14.6.14. HEALTHCARE PROFESSI QUESTIONNAIRE (PART #2) | IONAL | |
| LISTING 16.2.1.1. ANALYSIS SETs | | |
| LISTING 16.2.1.2. INCLUSION/EXCLUS | | 71 |
| LISTING 16.2.2.1. MAJOR PROTOCOL I | | |
| LISTING 16.2.2.2. MINOR PROTOCOL I | | |
| LISTING 16.2.2.3. COVID-19 RELATED | | <b>.</b> . |
| DEVIATIONS | | |
| LISTING 16.2.3.1. STUDY DRUG DISCO | JNTINUATION11 | J |

| LISTING | 16.2.4.1. INFORMED CONSENT & DEMOGRAPHY | . 176 |
|---|---|---|
| LISTING | 16.2.4.2. MEDICAL HISTORY | . 177 |
| LISTING | 16.2.4.3. SURGERY AND PROCEDURES HISTORY (CANCER AND NON-CANCER RELATED) | 178 |
| LISTING | 16.2.4.4. DLBCL DIAGNOSIS | |
| | 16.2.4.5. FOLLICULAR LYMPHOMA DIAGNOSIS | |
| | 16.2.4.6. ECOG PERFORMANCE STATUS, FLIPI AND IPI SCORE | |
| LISTING | 16.2.4.7. VIRAL SEROLOGY AT SCREENING | |
| | 16.2.4.8. CONCOMITANT MEDICATIONS | |
| LISTING | 16.2.5.1. PREVIOUS IV RITUXIMAB DOSE - DLBCL | . 184 |
| LISTING | 16.2.5.2. PREVIOUS IV RITUXIMAB DOSE - FL | . 185 |
| LISTING | 16.2.5.3. INITIAL CHOP | |
| LISTING | 16.2.5.4. SUBSEQUENT CHOP | . 187 |
| LISTING | 16.2.5.5. SUBSEQUENT cvp | . 188 |
| LISTING | 16.2.5.6. SUBSEQUENT FLUDARABINE | . 189 |
| LISTING | 16.2.5.7. SUBSEQUENT CHEMOTHERAPY | . 190 |
| LISTING | 16.2.5.8. INITIAL CVP | . 191 |
| LISTING | 16.2.5.9. INITIAL FLUDARABINE | . 192 |
| LISTING | 16.2.5.10. OTHER CHEMOTHERAPY | . 193 |
| LISTING | 16.2.5.11. STUDY DRUG ADMINISTRATION | . 194 |
| LISTING | 16.2.5.12. ANTI-LYMPHOMA CHEMO/IMMUNO THERAPY TREATMENT | . 195 |
| LISTING | 16.2.5.13. ANTI-LYMPHOMA RADIOTHERAPY TREATMENT | . 196 |
| LISTING | 16.2.5.14. ANTI-LYMPHOMA TREATMENT | . 197 |
| LISTING | 16.2.5.15. CHEMOTHERAPY SELECTION | . 198 |
| LISTING | 16.2.6.1. PRE-TREATMENT ADVERSE EVENTS | . 199 |
| LISTING | 16.2.6.2. ADVERSE EVENTS | . 200 |
| LISTING | 16.2.6.3. SERIOUS ADVERSE EVENTS | . 201 |
| | 16.2.6.4. ADVERSE EVENTS OF SPECIAL INTEREST (AESI) | . 202 |

| LISTING | 16.2.6.5. ADMINISTERED ASSOCIATED | |
|---------|-----------------------------------------------------------|-----|
| | REACTIONS | 203 |
| LISTING | 16.2.6.6. GRADE 3+ ADVERSE EVENTS | 204 |
| LISTING | 16.2.6.7. ADVERSE EVENTS LEADING TO | |
| | RITUXIMAB DRUG INTERRUPTION OR DRUG DELAYED | 205 |
| LISTING | 16.2. <b>6</b> .8. ADVERSE EVENTS LEADING TO | |
| | CHEMOTHERAPY DOSE MODIFICATION | 206 |
| LISTING | 16.2.6.9. ADVERSE EVENTS LEADING TO | |
| | CHEMOTHERAPY DISCONTINUATION | 207 |
| LISTING | 16.2.6.10. ADVERSE EVENTS WITHIN THE | 200 |
| TTOMING | MEDDRA SMQ ANAPHYLACTIC REACTIONS | |
| | 16.2.6.11. INJECTION SITE REACTIONS | |
| | 16.2. <b>6</b> .12. DEATH | |
| | 16.2.7.1. HEMATOLOGY | |
| | 16.2.7.2 BIOCHEMISTRY | |
| | 16.2.7.3. COAGULATION TESTS | |
| | 16.2.8.1. VITAL SIGNS & BODY WEIGHT | |
| | 16.2.8.2. SERUM PREGNANCY TEST | |
| | 16.2.8.3. URINE PREGNANCY TEST | |
| | 16.2.8.4. PHYSICAL EXAMINATION | |
| LISTING | 16.2.8.5. 12-LEAD ECG | 218 |
| LISTING | 16.2.8.6. TARGET LESION ASSESSMENT AT SCREENING (PART #1) | 219 |
| LISTING | 16.2.8.7. TARGET LESION ASSESSMENT AT | |
| | SCREENING (PART #2) | 220 |
| LISTING | 16.2.8.8. TARGET LESION ASSESSMENT SUBSEQUENT (PART #1) | 221 |
| LISTING | 16.2.8.9. TARGET LESION ASSESSMENT SUBSEQUENT (PART #2) | 222 |
| LISTING | 16.2.8.10. OVERALL LESION ASSESSMENT | 223 |
| LISTING | 16.2.8.11. SURVIVAL STATUS | 224 |
| LISTING | 16.2.8.12. BONE MARROW ASSESSMENT | 225 |
| LISTING | 16.2.8.13. RASQ FOR IV ADMINISTRATION | 226 |
| LISTING | 16.2.8.14. RASO FOR SC ADMINISTRATION | 227 |

| LISTING | 16.2.8.15. | HEALTHCARE | PROFESSIONAL | |
|---------|------------|------------|--------------|-----|
| | OUESTION | INAIRE | | 228 |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|---|---|
| aalPl | Age-adjusted International Prognostic Index |
| AAR | Administration-associated reaction |
| AE | Adverse Event |
| ALT (SGPT) | alanine aminotransferase |
| aPTT | Activated Partial Thromboplastin Time |
| AST (SGOT) | Aspartate Aminotransferase |
| BSA<br>BUN | body surface area |
| CEC | Blood Urea Nitrogen Clinical Events Committee |
| CHO | Chinese hamster ovary |
| СНОР | cyclophosphamide, oncovine (vincristine), doxorubicin, prednisone/prednisolone |
| CHOP-21 | CHOP given every 21 days |
| CHOP-14 | CHOP given every 14 days |
| CHVP | cyclophosphamide, doxorubicin, etoposide, prednisone/prednisolone |
| CI | Confidence Interval |
| CLL | chronic lymphocytic leukaemia |
| CR | Complete Response |
| CRF | Case Report Form |
| CRu | complete response unconfirmed |
| CRO | contract research organization |
| CT | Computerised Tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| $C_{trough}$ | Minimal plasma concentration prior to next drug administration |
| CVP | cyclophosphamide, vincristine, prednisone/prednisolone |
| DFS | disease-free survival |
| DLBCL | diffuse large B-cell lymphoma |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| EFS | event-free survival |
| EGSG | East German Study Group |
| EU | European Union |
| FC | Fludarabine, cyclophosphamide |

Rituximab - Roche North Africa (Algeria, Morocco & Tunisia) Mabrella ML28964 Daughter Protocol 17/Statistical Analysis Plan ML28964

Abbreviation Definition

FC 28 FC given every 28 days

FDA Food and Drug Administration

FDG-PET [18F]deoxyglucose positron emission tomography

FFS failure-free survival FL follicular lymphoma

FLIPI Follicular Lymphoma International Prognostic Index

G-CSF granulocyte colony-stimulating factor

GELA Groupe d'Etude des Lymphomes de l'Adulte
GLSG German Low-Grade Lymphoma Study Group

HACA human antichimeric antibody
HAMA human anti-mouse antibody

HBV Hepatitis B Virus
HCV Hepatitis C Virus

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

IB Investigator's Brochure ICF informed consent form

ICH International Council for Harmonisation

iDMC Independent Data Monitoring Committee

IDSMB Independent Data Safety Monitoring Board

IFN interferon-α

IMP Investigational Medicinal Product
INR International Normalised ratio
IPI International Prognostic Index
IRC Independent Review Committee
IRF Independent Review Facility
IRR Infusion-related reaction

IIRR infusion/injection-related reaction

ITT Intent-to-treat IV Intravenous

IWG International Working Group
LDH Lactate Dehydrogenase
LPLV last patient, last visit

MCP mitoxantrone, chlorambucil, prednisone/prednisolone

MedDRA Medical Dictionary for Regulatory Activities

MInT MabThera international trial
MRI Magnetic Resonance Imaging

Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

Mabrella ML28964 Daughter Protocol 18/Statistical Analysis Plan ML28964

Abbreviation Definition

NCI National Cancer Institute

NCI CTCAE National Cancer Institute Common Terminology Criteria for

Adverse Events

NHL Non-Hodgkin's Lymphoma

NIMP Non-investigational medicinal product

ORR Objective Response Rate

OS Overall Survival

PD progressive disease (disease progression)

PD pharmacodynamics

PET positron emission tomography

PFS progression-free survival

PK Pharmacokinetic

PML Progressive Multifocal Leukoencephalopathy

PR Partial Response

PRP patient-reported outcome

PT Prothrombin Time
PT Preferred Term
RBC Red Blood Cells

RCR Roche Clinical Repository

R-CHOP rituximab plus CHOP chemotherapy

RCT randomized controlled trial

R-CVP rituximab plus CVP chemotherapy
R-CHVP rituximab plus CHVP chemotherapy
R-FC Rituximab plus FC chemotherapy
rHuPH20 recombinant human hyaluronidase

SAE Serious Adverse Event
SAP Statistical Analysis Plan

SAS Statistical Analysis System (software)

SC subcutaneous(ly)
SD Stable Disease

SEER Surveillance, Epidemiology, and End Results

SOC System Organ Class

SPD sum of the products of the greatest diameters

SUSAR Suspected Unexpected Serious Adverse Reactions

SWT Satisfaction with Therapy
TLS Tumour lysis syndrome

TNLT time to next lymphoma treatment

Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

Mabrella ML28964 Daughter Protocol 19/Statistical Analysis Plan ML28964

| Abbreviation | Definition |
|--------------|------------------------------|
| TTF | time to treatment failure |
| TTP | time to tumour progression |
| ULN | <b>Upper Limit of Normal</b> |
| WBC | White Blood Cells |
| WHO | World Health Organization |

#### LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

# 1. BACKGROUND

The purpose of the analyses outlined in this Statistical Analysis Plan (SAP) is to evaluate the safety of Rituximab following subcutaneous administration in patients with CD20+ DLBCL or CD20+ follicular NHL grade 1 to 3A.

This SAP is based on Section 6 (Statistical considerations and analysis plan) of the study protocol version 3.1, signed on February 25 h, 2016.

# 2. <u>STUDY DESIGN</u>

This is an open-label, single-arm study to evaluate the safety of rituximab SC administered during first line treatment for FL (Induction and/or Maintenance), or DLBCL (treatment plus 24 months of follow-up).

This study will include adult patients with CD20+ DLBCL or CD20+ follicular NHL (grade 1 to 3a; NHL), who have already received at least one full dose of IV rituximab during induction or maintenance. Patients receiving Induction therapy must be able to receive at least 4 cycles of rituximab SC in addition to standard chemotherapy. FL Patients receiving Maintenance therapy must be able to receive at least 6 cycles of rituximab SC.

During administration of rituximab SC, patients will be assessed for safety and efficacy as detailed in the Schedule of Assessments (see Appendix 1 of Study Protocol). RASQ (see Appendix 6 of Study Protocol) will be applied to patients at the end of the study after rituximab administration. Healthcare Professional (HCP) Questionnaire (see Appendix 7 of study Protocol) will be applied at the end of the study to health care professionals.

#### **Induction Therapy:**

Patients receiving Induction therapy prior to entry into the study must be eligible to receive at least four further cycles of rituximab SC (i.e., 4 additional months of Induction treatment). Patients with follicular NHL who will continue into Maintenance therapy (after staging at the end of Induction) can continue to receive rituximab SC during Maintenance (see below).

#### Maintenance Therapy (patients with follicular NHL):

Patients receiving Maintenance therapy prior to entry into the study must be eligible to receive at least six further cycles of rituximab SC (i.e., 12 additional months of Maintenance treatment). Patients who are continuing into Maintenance therapy following at least four cycles of rituximab SC during Induction Therapy must also be eligible to

receive at least six cycles of rituximab SC (i.e. 12 additional months of Maintenance treatment).

## Post-treatment Follow Up:

All patients will continue the study with 24 months of follow-up period.

#### 2.1 PROTOCOL SYNOPSIS

The Protocol Synopsis is in Appendix 1. For additional details, see the Schedule of Assessments in Appendix 2.

#### 2.2 OUTCOME MEASURES

This study will evaluate safety of Rituximab following subcutaneous administration in patients with CD20+ DLBCL or CD20+ follicular NHL grade 1 to 3A.

## 2.2.1 Safety Outcome Measures

Safety outcome measures will include AARs (defined as all related AEs occurring within 24 hours of rituximab SC administration, including IIRRs, injection-site reactions, administration site conditions and all symptoms thereof), grade  $\geq$  3 AEs and SAEs. Other safety assessments include routine safety laboratory tests, vital signs measurements, and changes in concomitant medications. All clinical AEs and SAEs as well as laboratory abnormalities will be recorded regardless of their intensity / grading. Grading will be completed according to the NCI CTCAE version 4.0 (see Appendix 5 of the protocol).

## 2.2.2 Efficacy Outcome Measures

The efficacy of rituximab will be evaluated at the end of induction treatment for FL patients and at the end of the last cycle for DLBCL patients in terms of EFS, PFS, OS, CR/CRu and DFS. The endpoints of EFS, PFS and OS will be defined and analysed twice using two different starting points for the time-to-event calculations. The first starting point will be first dose of rituximab IV and the second will be first dose of rituximab SC.

- EFS is defined as the time from first dose of rituximab (analysed using both first dose of IV and first dose of SC) to first occurrence of progression or relapse, according to the IWG response criteria (Cheson et al 1999, see Protocol Appendix 2) or other country standards, or initiation of a non-protocol-specified anti-lymphoma therapy or death, whichever occurs first.
- PFS is defined as the time from first dose of rituximab (analysed using both first dose of IV and first dose of SC) to the first occurrence of progression or relapse, according to the IWG response criteria (Cheson et al. 1999, see Protocol Appendix 2) or other country standards, or death from any cause.

- OS is defined as the time from first dose of rituximab (analysed using both first dose of IV and first dose of SC) until death from any cause.
- DFS will be assessed at the end of induction treatment in patients achieving CR/CRu and is defined as the period from the date of the initial CR/CRu until the date of relapse or death from any cause.
- CR/CRu: Response assessments 4 6 weeks after the last dose of Induction treatment will be based on the Investigator's assessment, completed according to the original International Working Group (IWG) response criteria for response assessment of lymphoma (Cheson et al. 1999; see Protocol Appendix 2).

Tumour assessments will be based on computed tomography (CT) scans of the neck, chest, abdomen and/or pelvis (if detectable by these techniques) or other diagnostic means (e.g., magnetic resonance imaging [MRI], PET/CT) where applicable. Other methods (e.g., MRI) are acceptable for patients in whom CT scans are contraindicated. The CT scan used for eligibility assessments may be performed up to 28 days prior to dosing.

# 2.2.3 <u>Exploratory Outcome Measures</u>

Not applicable.

# 2.2.4 Pharmacokinetic Outcome Measures

Not applicable.

#### 2.3 DETERMINATION OF SAMPLE SIZE

A sample size of 110 patients is deemed sufficient for this study. In this study, all planned statistical analysis will be exploratory in nature as the study will not be powered to address any pre-defined statements and only descriptive statistical evaluations will be carried out primarily for safety (and efficacy) parameters. Additionally, no published reference is available on administration-associated reactions (AARs) following multiple doses of subcutaneous (SC) rituximab during induction and/or maintenance therapy in patients with CD20+ follicular non-Hodgkin's lymphoma (NHL) or CD20+ diffuse large B-cell lymphoma (DLBCL). However, with 110 patients a 95% Clopper-Pearson CI for the incidence of AARs will be no wider than +/- 9.7%. This width of interval is deemed sufficiently precise to draw valid conclusions around the incidence of ARRs. Additionally, enrolment of more than 110 patients within the specified indications could also be difficult in participating countries. Due to the fact of exploratory nature of the study, drop out patients will not be replaced.

## 2.3.1 <u>Sample Size for the China Extension Period</u>

Not applicable for this study.

#### 2.4 ANALYSIS TIMING

This length of the study study is planned according to the type of lymphoma (either FL or DLBCL). Since assessments for FL patients are expected to be on-study longer, this portion of the study will be determinative for the length of the study. For FL patients the study is estimated to take approximately 6 years (68 months) based on an approximately 12 month of recruitment period, 8 months of induction and 24 months of maintenance treatment and 24 months of follow-up period.

On the other hand, DLBCL patients are expected to be on-study for a shorter period of time (approximately in 4 years), based on approximately 12 months recruitment, 8 months of treatment and 24 months follow up period with a recruitment period of approximately 18 months

The end of the study, defined as last patient last visit (LPLV), will occur 24 months after the last SC rituximab treatment for the last FL or DLBCL patient, whichever comes later.

The statistical analysis will be performed after all patients have completed the study.

An interim analysis in not planned.

## 2.4.1 Analysis Timing for the China Subgroup Analysis

Not applicable for this study.

# 3. <u>STUDY CONDUCT</u>

# 3.1 RANDOMIZATION

Not applicable. This is an open-label study, non-comparative single arm study.

#### 3.2 INDEPENDENT REVIEW FACILITY

Not applicable for this study.

#### 3.3 DATA MONITORING

Not applicable for this study.

## 4. STATISTICAL METHODS

This is not a hypothesis testing study but an exploratory study with predefined precision of estimates for key safety parameters for sample size determination; there are no formal statistical hypotheses tests to be tested, and there will be no adjustments for multiplicity of endpoints or within-subgroups comparisons.

Descriptive statistics will be provided in summary tables according to the type of variable using appropriate descriptive statistics.

Continuous variables will be summarized by descriptive statistics (number of cases, mean, standard deviation, median, minimum and maximum).

Categorical variables will be summarized using counts of patients and percentages; missing category will be displayed if appropriate.

Exposure to study treatment (rituximab) and chemotherapy, including the number of cycles administered, duration of treatment exposure (calculated from date of first treatment date to the last treatment date) and dosing information (e.g., dose interruptions, modifications and delays) will be summarized.

The number of patients who prematurely discontinue study treatment and the number of patients who withdrew from the study will be summarized and reasons for withdrawal will be displayed

All data collected will be presented in by-patient data listings.

All planned analyses identified in this Statistical Analysis Plan (SAP) will be performed by SPARC Consulting (Milan) on behalf of IQVIA following Sponsor Authorization of this SAP.

All statistical analyses and data processing will be performed using SAS® Software (release 9.4 or higher) under Windows 10 PRO operating system.

All medical history and AE terms will be assigned to a Low Level Term (LLT), Preferred Term (PT) and will be classified by the primary System Organ Class (SOC) according to the Medical Dictionary for Regulatory Activities (MedDRA) thesaurus, version 24.1, medications will be coded using the INN-1.0V Dictionary, and laboratory values converted in Standard Unit (SI) by TCS, Mumbai, India.

Unplanned visits have been foreseen in the study. Unplanned measurements will not be included in by-visit summaries. Listings will include planned and unplanned data.

#### 4.1 ANALYSIS POPULATIONS

## 4.1.1 Randomized Population

Not applicable for this study.

# 4.1.2 <u>Per Protocol Population</u>

Not defined for this study.

# 4.1.3 <u>Pharmacokinetic-Evaluable Population</u>

Not applicable for this study.

## 4.1.4 <u>Safety Population</u>

The Safety data will be summarized based on the safety population (SAF), defined as all patients who have received at least one dose of rituximab.

## 4.1.5 <u>Intent-To-Treat Population</u>

The efficacy endpoints will be summarized based on the ITT population (ITT) defined as all patients enrolled into the study.

#### 4.2 ANALYSIS OF STUDY CONDUCT

Enrolment, patients' disposition, and discontinuation from the study will be summarized for the ITT population overall and for patients with Diffuse Large B-Cell Lymphoma (DLBCL) and patients with follicular Non-Hodgkin's Lymphoma (FL), separately. The reasons for study drug discontinuation will also be tabulated. Protocol deviations, including major deviations with regards to the inclusion and exclusion criteria and major deviations due to Covid-19 pandemic, will be summarized by deviation category for the ITT population. A line listing with all protocol deviations reported over the study will be also provided.

Deviations from the protocol including violations of inclusion/exclusion criteria will be assessed definitely as "minor" or "major" by the study clinical team prior to closure of the study database.

## 4.2.1 Definition of Baseline

Baseline is defined as the screening visit. Thus, change from baseline to a specific timepoint of a study parameter is calculated as follows:

Change from baseline to time X = (value at time X) - (baseline value).

#### 4.3 ANALYSIS OF TREATMENT GROUP COMPARABILITY

Demographic and other baseline characteristics (including age, sex, ethnicity, and baseline disease characteristics, e.g., DLBCL Diagnosis), as well as the demographic profile (height, weight, and BMI), IPI score (according to Shipp et al. 1993) and/or FLIPI score and serum pregnancy test at Screening/Baseline will be summarized using means, standard deviations, medians, and ranges for continuous variables and proportions for categorical variables, as appropriate.

Summaries will be presented overall and for patients with DLBCL and patients with FL separately for ITT population.

A summary analysis of the DLBCL and FL diagnosis will be presented for the SAF population.

The overall evaluation of a 12-lead ECG tracing at screening will be presented by means of a summary analysis on SAF population.

#### 4.3.1 Medical History

Data from "Medical History" form will be summarized for ITT population with descriptive statistics.

All verbatim terms reported will be assigned to a PT and will be classified by the primary SOC.

Previous diseases are those reported in the "Medical History" form of the eCRF not flagged as "Ongoing at study entry".

Concomitant diseases are those flagged as "Ongoing at study entry".

The following data will be presented:

- A default frequency table showing the number and percentage of patients who exhibited at least one previous disease and the previous diseases by primary SOC and PT;
- A default frequency table showing the number and percentage of patients who exhibited at least one concomitant disease and the concomitant diseases by primary SOC and PT.

Any previous diseases as well as concomitant diseases will be listed.

## 4.3.2 <u>Surgery and Procedures History</u>

Data from "Surgery and Procedures history (cancer and non-cancer related)" form will be summarized for ITT population with descriptive statistics.

All verbatim terms reported will be assigned to a PT and will be classified by the primary SOC.

The following data will be presented:

• A default frequency table showing the number and percentage of patients who exhibited at least one surgery and the surgery by primary SOC and PT;

All surgery and procedures will be listed.

# 4.3.3 **Physical Examination**

Physical Examinations details for each body system will be summarized across each visit for safety population.

# 4.3.4 Previous and Concomitant Therapies

Data from "Concomitant Medication" form will be summarized for safety population with descriptive statistics.

Therapies will be coded using the INN-1.0V dictionary. New anti-lymphoma treatment (chemotherapy, radiotherapy, immunotherapy), initiated after the Baseline visit will be presented in summary tables.

Handling of partial dates for prior and concomitant therapies will be performed by TCS, Mumbai, India.

Previous therapy includes any medication stopped before exposure to study drug. The following data will be presented in a unique summary table for previous therapies:

- Total number of patients with at least one treatment (n,%)
- Total number of treatments (n)
- Total number of patients with at least one treatment by ATC class level 2 (n,%)
- Total number of treatments by ATC class level 2 (n)
- Treatments by ATC class level 2 (n,%)

Concomitant therapy consists of any medication taken during the study, including those started before but ongoing at first dose of study drug. The following data will be presented overall in a unique summary table for concomitant therapies:

- Total number of patients with at least one treatment (n,%)
- Total number of treatments (n)
- Total number of patients with at least one treatment by ATC class level 2 (n,%)
- Total number of treatments by ATC class level 2 (n)
- Treatments by ATC class level 2 (n,%)

All previous and concomitant therapies reported over the study will be listed.

## 4.3.5 <u>Viral Serology</u>

Viral serology at screening including HBcAb, HBsAg, HCV antibody, and HIV antibody will be summarized for SAF population with descriptive statistics.

#### 4.4 EFFICACY ANALYSIS

The efficacy analysis will be performed in the ITT analysis set.

Efficacy endpoints include EFS, PFS, OS, DFS, and CR/CRu rate.

Summaries will be presented overall and for patients with DLBCL and patients with FL separately.

Response assessments will be based on the Investigator's assessment, completed according to the IWG response criteria (Cheson et al 1999, see Appendix 2 of Study Protocol) or other country standards. The endpoints of EFS, PFS and OS will be defined and analyzed twice using two different starting points for the time-to-event calculations. The first starting point will be first dose of rituximab IV and the second will be first dose of rituximab SC.

The analysis of endpoints measured as a time-to-event (e.g., EFS, PFS, OS and DFS) is based on the survivor function, which is the probability of remaining event free beyond a certain point in time.

The survivor function will be estimated using Kaplan-Meier methodology and summarized using the range, the 25th and 75th percentiles and median survival along their 95% confidence interval.

Patients who have experienced none of these events at the time of analysis (clinical cutoff) and patients who are lost to follow up will be censored at their last clinical assessment date. Patients without post-baseline tumour assessments will be censored at the time of their baseline visit except if death occurs prior to their first scheduled tumour assessment.

The survivor function will be displayed graphically using a Kaplan-Meier curve.

The number and percentage of the patients with event or censored will be also presented. Analysis will be performed using the SAS procedure Proc Lifetest.

# 4.4.1 **Primary Efficacy Endpoint**

Not applicable.

# 4.4.2 <u>Secondary Efficacy Endpoints</u>

#### **Event-Free Survival (EFS)**

EFS is defined as the time from first dose of rituximab (analysed using both first dose of IV and first dose of SC) to first occurrence of progression or relapse, according to the IWG response criteria (Cheson et al 1999, see Appendix 2 of Study Protocol) or other country standards, or initiation of a non-protocol-specified anti-lymphoma therapy or death, whichever occurs first. Time will be calculated in months as follow:

EFS = (date of event/censor – date of first dose + 1) / 30.4375

## **Progression-Free Survival (PFS)**

PFS is defined as the time from first dose of rituximab (analysed using both first dose of IV and first dose of SC) to the first occurrence of progression or relapse, according to the IWG response criteria (Cheson et al 1999, see Appendix 2 of Study Protocol) or other country standards, or death from any cause. Time will be calculated in months as follow:

PFS = (date of event/censor – date of first dose + 1) / 30.4375

#### Overall Survival (OS)

OS is defined as the time from first dose of rituximab (analysed using both first dose of IV and first dose of SC) until death from any cause. Time will be calculated in months as follow:

OS = (date of event/censor – date of first dose + 1) / 30.4375

#### Disease-Free Survival (DFS)

DFS will be assessed in patients achieving CR/CRu and is defined as the period from the date of the initial CR/CRu until the date of relapse or death from any cause. Time will be calculated in months as follow:

Rituximab - Roche North Africa (Algeria, Morocco & Tunisia) Mabrella ML28964 Daughter Protocol 29/Statistical Analysis Plan ML28964

## Complete Response rate (CR)/Complete Response unconfirmed (CRu)

CR/CRu rate at 4-6 weeks after the last dose of Induction treatment will be summarized and presented with the corresponding 95% two-sided Pearson-Clopper CI by treatment group and overall.

Endpoints resulting in an incidence rate (e.g., CR/CRu) will be summarised with a 95% Clopper-Pearson confidence interval.

## 4.4.3 Exploratory Efficacy Endpoints

Not applicable.

## 4.4.4 Sensitivity Analyses

Not applicable.

# 4.4.5 Subgroup Analyses

Demographics and baseline characteristics (age, ethnicity, height, weight, BMI, IPI score, FLIPI score and Surgery/Procedure History) will be also presented stratified by gender (Male, Female).

- a) PFS and OS results will be reported for the following I subgroups, in addition to the analysis populations described in the document: Gender (Female, Male)
- b) FLIPI score (Low risk, Intermediate risk/High risk) for FL patients only
- c) Grade of FL (1, 2, 3a)

#### 4.5 PHARMACOKINETIC AND PHARMACODYNAMIC ANALYSES

Not applicable.

#### 4.6 PATIENT-REPORTED OUTCOME ANALYSES

Patient satisfaction with administration of treatment will be evaluated using the Rituximab Administration Questionnaire (RASQ) for safety population.

The RASQ is a 20-item questionnaire measuring the impact of the mode of treatment administration on five domains: Physical Impact, Psychological Impact, Impact on Activities of Daily Living, Convenience, and Satisfaction. The Physical Impact domain comprises of 3 items (Pain, swelling, and redness (Q2), Pain experience (Q3), Side effects as expected (Q4)), the Psychological Impact domain contains 5 items (Anxious about injection/IV (Q5), Worry condition will get worse (Q6), Anxious thinking about disease (Q7), Confidence the injection/IV treating disease (Q8), Feeling restricted by injection/IV (Q9)), the Impact on Activities of Daily Living domain contains 3 items (Interference with usual/daily activities (Q14a), Limit daily activities (Q14b), Lost/gained time(Q15)), the Convenience domain contains 3 items (Is it convenient to get injection/IV

Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

(Q10), Length of time to get injection/IV as expected (Q12), Bothered by the amount of time to get injection/IV (Q13)) and the Satisfaction domain includes 2 items (How satisfied or dissatisfied are you with the injection/IV (Q1), Would you recommend the way you received the treatment (Q19). All 16 RASQ items included in the above domains have five response options. Reverse-coded response values will be created for eight of the RASQ items (Q2, Q3, Q5, Q6, Q7, Q9, Q14a, and Q14b).

In addition, there are 4 descriptive questions that are not part of the above domains and are scored separately.

For each domain, if there are no missing responses, the domain will be scored using the formula:

Domain score = [(Sum of completed item responses / Number of completed items) - 1] x 100 / (Maximum possible item response value – Minimum possible item response value)

However, if there are any missing responses within a domain then the domain will not be scored (i.e., a missing value is assigned to the domain).

Since the maximum possible item response value is 5 and the minimum possible response value is 1 for all RASQ items, a simpler way to represent the above formula for the RASQ domains is:

RASQ domain score = (Mean of completed item responses -1) x 25

Descriptive statistics will be computed for the RASQ questions assessing patient responses regarding convenience, satisfaction and preference for rituximab SC as compared to rituximab IV. Specifically, frequencies and percentages will be presented by question and timepoint, for the total sample and for patients with DLBCL and patients with FL separately.

In addition, descriptive statistics will be computed by domain (Physical Impact domain, Psychological Impact domain, Impact on Activities of Daily Living domain, Convenience domain and Satisfaction domain) and timepoint overall and for patients with DLBCL and patients with FL separately.

Listings will present by patient data for individual responses and domain scores.

# 4.7 HEALTHCARE PROFESSIONAL REPORTED OUTCOME ANALYSES

Healthcare Professional (HCP) Questionnaire will be evaluated with descriptive statistics. Frequencies and percentages will be presented.

All data reported in Healthcare Professional (HCP) Questionnaire will be listed.

#### 4.8 SAFETY ANALYSES

All safety analyses will be presented for the Safety population overall and for patients with DLBCL and patients with FL separately.

Safety will be assessed by AEs, AEs of grade  $\geqslant$  3, SAEs, AARs including IIRRs, AEs within the MedDRA SMQ "Anaphylactic reactions" (wide), safety laboratory parameters, vital signs, concomitant medications, premature withdrawal from the study and from study medication due to AEs and ECOG performance status. All clinical AEs and SAEs as well as laboratory abnormalities will be recorded and graded according to the NCI-CTCAE version 4.0.

# 4.8.1 <u>Exposure of Study Medication</u>

Exposure to study treatment (rituximab) and chemotherapy, including the number of cycles administered in induction and maintenance phases, duration of treatment exposure (calculated from date of first treatment date to the last treatment date) and dosing information (e.g., dose interruptions, modifications and delays) will be summarized for the safety population.

New anti-lymphoma treatment (chemotherapy, radiotherapy, immunotherapy), initiated after baseline visit will be presented in summary tables.

Summary analysis will be presented overall and for patients with DLBCL and patients with FL separately.

#### 4.8.2 Adverse Events

The analysis of AEs will focus on treatment-emergent adverse events (TEAEs), i.e., AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose. Non-treatment emergent AEs (i.e., those occurring before commencement of study medication) will only be listed. Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA version 24.1).

Handling of partial dates for AEs will be performed by TCS, Mumbai, India. Where an AE start date is partially or fully missing, and it is unclear as to whether AE started after of the study, it will be assumed to be TEAE (worst case).

The incidence of AARs, AEs, AEs leading to premature discontinuation or interruption of study treatment, SAEs, grade  $\geq$  3 AEs will be computed with 95% Confidence Interval (calculated using either the Clopper-Pearson methodology, or the Poisson distribution, for frequencies below 10%). The incidence of each AE will be summarized according to the primary System Organ Class and by Preferred Term. The incidence of cutaneous and soft tissue AARs will additionally be summarised for those that are defined as localized and those that are defined as non-localized. The incidence of deaths and cause of deaths will be listed and summarized.

Counts and percentages will be presented, by primary SOC and PT, overall and for patients with DLBCL and patients with FL separately.

A patient having more than one adverse event with the same PT will be counted only once in the incidence calculation for that PT. Similarly, if a patient has more than one AE in the same SOC, the patient will be counted only once in the total number of patients with an AE for that SOC.

Where AEs are summarized by relationship or by maximum CTC grade, each patient's maximum CTC grade will be used in the summary. If a patient experiences the same adverse event at more than one CTC grade level, or with more than one relationship to study drug, the most severe rating or the stronger causal relationship to study drug will be used.

Any missing CTC grade, casualty, or outcome will not be imputed but classified as unknown for listing purpose and the worst case will be considered for summarization purpose.

If the severity is missing for a TEAE, the TEAE will be considered as Severe.

If the relationship to study treatment is missing for a TEAE, the TEAE will be considered as related to study treatment.

If CTG grade is missing, the worst CRT grade will be considered.

An overview of number of patients with at least one Treatment Emergent Adverse Event (TEAE), at least one serious TEAE, at least one AE of special interest (AESI), at least one Administration Associated Reaction (AARs), at least one cutaneous and soft tissue AARs (localized), at least one cutaneous and soft tissue AARs (non-localized), at least one grade  $\geq$  3 TEAEs, at least one grade  $\geq$  3 serious TEAEs, at least one grade  $\geq$  3 infusion/injection related reactions, number of TEAEs leading to Rituximab drug interrupted/drug delayed, number of TEAEs leading to Rituximab dose discontinuation, number of TEAEs leading to chemotherapy dose modification, number of TEAEs leading to chemotherapy dose discontinuation and number of TEAEs leading to death will be provided.

The following summary statistical tables including frequencies and percentages, along with the 95% CI of the observed proportions (calculated using either the Clopper-Pearson methodology, or the Poisson distribution, for frequencies below 10%) will be provided:

- Proportion of all TEAEs by Primary SOC and PT;
- Proportion of serious TEAEs by Primary SOC and PT;

- Proportion of localized AARs by Primary SOC and PT;
- Proportion of non-localized AARs by Primary SOC and PT;
- Proportion of grade ≥ 3 TEAEs by Primary SOC and PT;
- Proportion of grade ≥ 3 serious TEAEs by Primary SOC and PT;
- Proportion of grade ≥ 3 AARs by Primary SOC and PT;
- Proportion of TEAEs leading to Rituximab drug interrupted/drug delayed by Primary SOC and PT;
- Proportion of TEAEs leading to Rituximab dose discontinuation by Primary SOC and PT;
- Proportion of TEAEs leading to chemotherapy dose modification by Primary SOC and PT;
- Proportion of TEAEs leading to chemotherapy dose discontinuation by Primary SOC and PT;
- Proportion of TEAEs leading to death by Primary SOC and PT.

The following groups of adverse events will be summarized:

- All TEAEs;
- All Treatment-Emergent SAEs;
- All AESI;
- All AARs:
- All IRRs:
- Grade ≥ 3 TEAEs;
- Grade ≥ 3 Treatment-Emergent SAEs;
- Grade ≥ 3 AESI;
- Grade ≥ 3 AARs:
- Grade ≥ 3 IIRRs;
- TEAEs within the MedDRA SMQ "Anaphylactic reactions" (wide);
- TEAEs leading to dose modification of Rituximab;
- TEAEs leading to dose modification of chemotherapy;
- TEAEs leading to discontinuation of chemotherapy;
- TEAEs leading to death;
- Cutaneous and soft tissue AARs (localized);
- Cutaneous and soft tissue AARs (non-localized);

Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)
Mabrella ML28964 Daughter Protocol
34/Statistical Analysis Plan ML28964

- TEAEs with an incidence ≥ 5 %;
- TEAEs by maximum severity;
- Non TEAEs by strongest relationship;
- Non serious TEAEs with an incidence ≥ 5 %.

These groups will be summarized using the following factors by System Organ Class and Preferred Term:

- total
- event related to Rituximab
- event related to chemotherapy

The following individual data listings will be produced:

- A listing of all AEs;
- A listing of all serious AEs;
- A listing of all AESI;
- A listing of all AARs;
- A listing of all AEs related to Rituximab;
- A listing of grade ≥ 3 AEs;
- A listing of all AEs leading to Rituximab drug interruption/drug delay;
- A listing of all AEs leading to Rituximab drug discontinuation;
- A listing of all AEs leading to chemotherapy dose modification;
- A listing of all AEs leading to chemotherapy dose discontinuation;
- A listing of all AEs within the MedDRA SMQ "Anaphylactic reactions";
- A listing of all Cutaneous and soft tissue AARs (localized);
- A listing of all Cutaneous and soft tissue AARs non-(localized);
- A listing of death
- A listing of all pre-treatment AE.

AEs of special interest (AESI) include AARs, hepatotoxicity (elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined in Section 5.3.5.6 of Study Protocol) and suspected transmission of an infectious agent by the study drug (see Section 5.2.3 of Study Protocol).
## 4.8.3 <u>Laboratory Data</u>

Summary analysis will be performed in the safety population overall and for patients with DLBCL and patients with FL separately.

Actual values and the changes from baseline to each time-point in hematology, biochemistry, coagulation test parameters will be summarized using descriptive statistics.

Shift tables of NCI CTCAE grade at baseline against worst grade recorded during the treatment period will be presented for all laboratory parameters.

A list of laboratory assessments to be included:

- Haematology: hemoglobin, RBC count, WBC count and differential count (neutrophils, eosinophils, basophils, monocytes, lymphocytes, other cells) and platelet count;
- Biochemistry at Screening: sodium, potassium, ALT/SGPT, AST/SGOT, total bilirubin, serum creatinine, alkaline phosphatase, albumin, blood urea nitrogen (BUN), C-reactive protein and LDH. Biochemistry at any further timepoint: sodium, potassium, ALT/SGPT, AST/SGOT, total bilirubin, and serum creatinine;
- Coagulation: International Normalized Ratio (INR), Prothrombin Time (PT), Activated Partial Thromboplastin Time (aPTT).

For each laboratory parameter, where appropriate, the reported values will be converted into SI units and if needed boundary values for reference ranges will be converted.

## 4.8.4 <u>Vital Signs</u>

Analysis of vital signs will be performed in the safety population overall and for patients with DLBCL and patients with FL separately.

Vital signs will include measurements of heart rate, systolic and diastolic blood pressure, and body temperature.

A summary of actual values and changes from baseline over the study will be provided for each vital sign with default descriptive statistics at each time-point.

## 4.8.5 <u>ECOG Performance Status</u>

Eastern Cooperative Oncology Group (ECOG) performance status (Grade 0 – Grade 5) will be summarized by frequency tables over time for the safety population overall and for patients with DLBCL and patients with FL separately.

## 4.9 MISSING DATA

Imputed values will be included in the analysis set(s), but will not change the original clinical database (rawdata).

Missing data in safety parameters will not be replaced except for relationship to study medications and severity of AE and partial date in AE and prior/concomitant treatments (Sections 4.3.4 and 4.8.2).

In all efficacy analyses, missing data handling is specific to the efficacy endpoint and details are given within Section 4.4 for all efficacy endpoints.

For analysis of change from baseline endpoints if no baseline value exists for a patient at a specific time-point, then the patient will be excluded from the analysis of that time-point.

# 4.10 INTERIM ANALYSES

No interim analyses are planned.

| 5. | CHINA SUBGROUP ANALYSIS |
|----------------|-------------------------|
| Not applicable | Э. |

## 6. <u>REFERENCES</u>

Badin F, Hayslip J. Rituximab in the treatment of B-cell non-Hodgkin lymphoma, focus on outcomes and comparative effectiveness. Clinicoecon Outcomes Res 2010;2:37-45.

Bookbinder LH, Hofer A, Haller MF et al. A recombinant human enzyme for

enhanced interstitial transport of therapeutics. J Control Release 2006;114(2):230-41. Bordeleau L, Berinstein NL. Molecular diagnostics in follicular non-Hodgkin's lymphoma: a review. Semin Oncol 2000;27(Suppl 12):42-52.

Boye J, Elter T, Engert A. An overview of the current clinical use of the anti-CD20 monoclonal antibody rituximab. Ann Oncol 2003;14:520-35.

Cairo M, Bishop M. Tumor lysis syndrome: new strategies and classification. Br J Hematol 2004;127(1):3-11.

Cartwright RA. Time trends in incidence of haematological malignancies and related conditions. Br J Haematol 1999;106:281-95.

Cheson BD, Horning SJ, Coiffier B, et al. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol 1999;17(4):1244.

Clarke CA, Glaser SL. Changing incidence of non-Hodgkin's lymphomas in the United States. Cancer 2002;94:2015-23.

Coiffier B, Altman A, Pui CH et al. Guidelines for the management of pediatric and adult tumor lysis syndrome: an evidence-based review. J Clin Oncol. 2008 Jun 1;26(16):2767-78.

Coiffier B, Lepage E, Briere J et al. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med 2002;346(4):235-42.

Coiffier B, Thieblemont C, Van Den Neste E et al. Long-term outcome of patients in the LNH-98.5 trial, the first randomized study comparing rituximab-CHOP to standard CHOP chemotherapy in DLBCL patients: a study by the Groupe d'Etudes des Lymphomes de l'Adulte. Blood 2010;116(12):2040-5.

Cunningham D, Smith P, Mouncey P et al. R-CHOP14 versus R-CHOP21: Result of a randomized phase III trial for the treatment of patients with newly diagnosed diffuse large B-cell non-Hodgkin lymphoma. J Clin Oncol 2011;29(15, suppl):abstr 8000.

Davis TA, Grillo-Lopez AJ, White CA et al. Rituximab anti-CD20 monoclonal antibody therapy in non-Hodgkin's lymphoma: safety and efficacy of re-treatment. J Clin Oncol 2000;18(17):3135-43.

Davis TA, White CA, Grillo-Lopez AJ et al. Single-agent monoclonal antibody efficacy in bulky non-Hodgkin's lymphoma: results of a phase II trial of rituximab. J Clin Oncol 1999;17(6):1851-7.

Delarue R, Tilly H, Salles G et al. R-CHOP-14 compared to R-CHOP-21 in elderly patients with diffuse large B-cell lymphoma (DLBCL): Results of the second interim analysis of the LNH03-6B GELA study. Ann Oncol 2011;22(suppl 4):117 abstract 106.

Del Nagro CJ, Mao CP, Brovarney M et al. Comparison of B cell depletion mediated by intravenous (IV) Rituxan(R) and Rituxan given subcutaneous (SC) in cynomolgus monkeys. Blood (ASH Annual Meeting Abstracts) 2010;116(21): abstract 3980.

Demidem A, Lam T, Alan S et al. Chimeric anti-CD20 (IDEC-C2B8) monoclonal antibody sensitizes a B cell lymphoma cell line to cell killing by cytotoxic drugs. Cancer Biother Radiopharm 1997;12:177-86.

Eltom MA, Jemal A, Mbulaiteye SM et al. Trends in Kaposi's sarcoma and non-Hodgkin's lymphoma incidence in the United States from 1973 through 1998. J Natl Cancer Inst. 2002;94:1204-10.

Ferlay J, Autier P, Boniol M et al. Estimates of the cancer incidence and mortality in Europe in 2006. Ann Oncol 2007;18:581-92.

Feugier P, Van Hoof A, Sebban C et al. Long-term results of the R-CHOP study in the treatment of elderly patients with diffuse large B-cell lymphoma: a study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol 2005;23:4117-26.

Fisher RI, Gaynor ER, Dahlberg S et al. Comparison of a standard regimen (CHOP) with three intensive chemotherapy regimens for advanced non-Hodgkin's lymphoma. New Engl J Med 1993;328:1002-6.

Fisher RI, LeBlanc M, Press OW et al: New treatment options have changed the survival of patients with follicular lymphoma. J Clin Oncol 2005;23:8447-52.

Friedberg JW. Treatment of follicular non-Hodgkin's lymphoma: the old and the new. Semin Hematol 2008;45(3 suppl 2):S2-6.

Friedberg JW, Taylor MD, Cerhan JR et al. Follicular lymphoma in the United States: first report of the national LymphoCare study. J Clin Oncol 2009;27(8):1202-8.

Frost GI. Recombinant human hyaluronidase (rHuPH20): an enabling platform for subcutaneous drug and fluid administration. Expert Opin Drug Deliv 2007;4(4):427-40.

Habermann TM. Antibody therapy in aggressive lymphomas. Hematology Am Soc Hematol Educ Program 2007:257-64.

Habermann TM, Weller EA, Morrison VA et al. Rituximab-CHOP versus CHOP alone or with maintenance rituximab in older patients with diffuse large B-cell lymphoma. J Clin Oncol 2006;24(19):3121-7.

Herold M, Dölken G, Fiedler F et al. Ongoing clinical studies – randomized phase III study for the treatment of advanced indolent NHL and MCL: chemotherapy versus chemotherapy plus Rituximab. Ann Hematol 2003;82:77-9.

Herold M, Haas A, Srock S et al. Rituximab added to first-line mitoxantrone, chlorambucil, and prednisolone chemotherapy followed by interferon maintenance prolongs survival in patients with advanced follicular lymphoma: An East German study group hematology and oncology study. J Clin Oncol 2007;25(15):1986-92.

Hiddemann W, Kneba M, Dreyling M et al: Frontline therapy with rituximab added to the combination of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) significantly improves the outcome for patients with advanced-stage follicular lymphoma compared with therapy with CHOP alone: Results of a prospective randomized study of the German low-grade lymphoma study group.

Blood 2005;106:3725-32.

Horning SJ. Natural history of and therapy for the indolent non-Hodgkin's lymphomas. Semin Oncol 1993;20(Suppl 5):75-88.

Howlader N, Noone AM, Krapcho M et al. (eds). SEER Cancer Statistics Review, 1975-2009 (Vintage 2009 Populations), National Cancer Institute. Bethesda, MD, http://seer.cancer.gov/csr/1975\_2009\_pops09/, based on November 2011 SEER data submission, posted to the SEER web site, 2012.

[ILSG] The Non-Hodgkin's Lymphoma Classification Project. A clinical evaluation of the International Lymphoma Study Group classification of non-Hodgkin's lymphoma. Blood 1997;89:3909-18.

Investigator Brochure MabThera®, Rituxan®, Fifteenth Edition, July 2010 (Rituximab IV), and Second Edition, October 2010 (Rituximab SC).

Jaffe ES, Harris NL, Stein H et al. (eds). World Health Organization classification of tumours. Pathology and genetics of tumours of haematopoietic and lymphoid tissues. Lyon, France: IARC Press; 2001.

Keating GM. Rituximab: a review of its use in chronic lymphocytic leukaemia, low- grade or follicular lymphoma and diffuse large B-cell lymphoma. Drugs 2010;70(11):1445-76.

Kornbrot B, Kobayashi RH, Singer A et al. Hypersensitivity to therapeutic murine monoclonal antibodies. Nebr Med J 1994;79(12):393-8.

Landis SH, Murray T, Bolden S et al. Cancer Statistics, 1999. CA Cancer J Clin 1999;49(1):8-31.

Lenz G, Dreyling M, Hoster E et al. Immunochemotherapy with rituximab and cyclophosphamide, doxorubicin, vincristine, and prednisone significantly improves response and time to treatment failure, but not long-term outcome in patients with previously untreated mantle cell lymphoma: Results of a prospective randomized trial of the German low grade lymphoma study group (GLSG). J Clin Oncol 2005;23(9):1984-92.

Lossos IS. Higher-grade transformation of follicular lymphoma - a continuous enigma. Leukemia 2005;19(8):1331-3.

Mager DE, Jusko WJ. General pharmacokinetic model for drugs exhibiting target-mediated drug disposition. J Pharmacokinet Pharmacodyn. 2001;28(6):507-32.

Maloney D, Smith B, Appelbaum F. The anti-tumor effect of monoclonal anti-CD20 antibody (MAB) therapy includes direct anti-proliferative activity and induction of apopthosis in CD20 positive non-Hodgkin's lymphoma (NHL) cell lines. Blood 1996;88:637a.

Marcus R, Imrie K, Belch A et al. CVP chemotherapy plus rituximab compared with CVP as first-line treatment for advanced follicular lymphoma. Blood 2005;105:1417- 23.

Marcus R, Imrie K, Solal-Celigny P et al. Phase III study of R-CVP compared with cyclophosphamide, vincristine, and prednisone alone in patients with previously untreated advanced follicular lymphoma. J Clin Oncol 2008;26(28):4579-86.

McLaughlin P, Grillo-López AJ, Link BK et al. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: half of patients respond to a four-dose treatment program. J Clin Oncol 1998;16:2825-33.

Michallet AS, Coiffier B. Recent developments in the treatment of aggressive non-Hodgkin lymphoma. Blood Rev 2009;23(1):11-23.

Moreau P, Pylypenko H, Grosicki S et al. Subcutaneous versus intravenous administration of bortezomib in patients with relapsed multiple myeloma: a randomised, phase 3, non-inferiority study. Lancet Oncol 2011;12(5):431-40. Morton LM, Wang SS, Devesa SS et al. Lymphoma incidence patterns by WHO subtype in the United States, 1992-2001. Blood 2006;107(1):265–76.

Nathwani BN, Harris NL, Weisenburger D et al. Follicular lymphoma. In Jaffe ES, Harris NL, Stein H et al. (eds). World Health Organization classification of tumors. Pathology and genetics of tumors of haematopoietic and lymphoid tissues. IARC Press: Lyon 2001;162-7.

National Cancer Center Network Guidelines, v3 2011 (www.nccn.org)

Niitsu N. Current treatment strategy of diffuse large B-cell lymphomas. Int J Hematol 2010;92(2):231-7.

Pettengell R, Linch D. Position paper on the therapeutic use of rituximab in CD20-positive diffuse large B-cell non-Hodgkin's lymphoma. Br J Haematol 2003;121(1):44-8.

Pfreundschuh M, Schubert J, Ziepert M et al. German high-grade non-Hodgkin lymphoma study group (DSHNHL). Six versus eight cycles of bi-weekly CHOP-14 with or without rituximab in elderly patients with aggressive CD20+ B-cell lymphomas: a randomised controlled trial (RICOVER-60). Lancet Oncol 2008;9(2):105-16.

Pfreundschuh M, Trümper L, Osterborg A et al. MabThera international trial group. CHOP-like chemotherapy plus rituximab versus CHOP-like chemotherapy alone in young patients with good-prognosis diffuse large-B-cell lymphoma: a randomised controlled trial by the MabThera international trial (MInT) group. Lancet Oncol 2006;7(5):379-91.

Pulte D, Gondos A, Brenner H. Ongoing improvement in outcomes for patients diagnosed as having non-Hodgkin's lymphoma from the 1990s to the early 21st century. Arch Intern Med 2008;168:469-76.

Reff ME, Carner K, Chambers KS et al. Depletion of B cells in vivo by a chimeric mouse human monoclonal antibody to CD20. Blood 1994;83:435-45.

Rituximab Summary of Product Characteristics

Salar A, Bouabdallah R, McIntyre C et al. A two-stage phase Ib study to investigate the pharmacokinetics, safety and tolerability of subcutaneous rituximab in patients with follicular lymphoma as part of maintenance treatment. Blood (ASH Annual Meeting Abstracts) 2010;116(21): abstract 2858.

Salar A, et al. Final Results of the BP22333 Study Demonstrate Non-Inferior Pharmacokinetics and Safety of Subcutaneous Administration of Rituximab Compared with Intravenous Administration As Maintenance Therapy in Patients with Follicular Lymphoma (ASH Annual Meeting Abstracts) 2012. Abstract 1641. Full citation pending.

Salles G, Mounier N, de Guibert S et al: Rituximab combined with chemotherapy and interferon in follicular lymphoma patients: Results of the GELA-GOELAMS FL2000 study. Blood 2008;112:4824-31.

Shipp MA, Harrington DP et al. A predictive model for aggressive non-Hodgkin's lymphoma. The international non-Hodgkin's lymphoma prognostic factors project. N Engl J Med 1993;329(14):987-94.

Smith TJ, Khatcheressian J, Lyman GH et al. 2006 update of recommendations for the use of white blood cell growth factors: an evidence-based clinical practice guideline. J Clin Oncol 2006;24(19):3187-205.

Solal-Celigny P, Roy P, Colombat P et al. Follicular lymphoma international prognostic index. Blood 2004;104(5):1258-65.

Sousou T, Friedberg J. Rituximab in indolent lymphomas. Semin Hematol 2010;47(2):133-42.

Stilgenbauer S, Zenz T, Winkler D et al; German chronic lymphocytic leukemia study group. Subcutaneous alemtuzumab in fludarabine-refractory chronic lymphocytic leukemia: Clinical results and prognostic marker analyses from the CLL2H study of the German chronic lymphocytic leukemia study group. J Clin Oncol 2009;27(24):3994-4001.

Swenson WT, Wooldridge JE, Lynch CF et al. Improved survival of follicular lymphoma patients in the United States. J Clin Oncol 2005;23:5019-26.

Swerdlow SH, Campo E, Harris NL et al. WHO classification of tumours of haematopoietic and lymphoid tissues, 4th edition, IARC Press, 2008.

Tedder TF, Engel P. CD20: a regulator of cell-cycle progression of B lymphocytes. Immunol Today 1994;15:450-4.

Tilly H, Dreyling M; ESMO guidelines working group. Diffuse large B-cell non- Hodgkin's lymphoma: ESMO clinical practice guidelines for diagnosis, treatment and follow-up. Ann Oncol 2010;21(suppl 5):v172-4.

Wynne C, Harvey V, Schwabe C et al. The development of a formulation of trastuzumab for subcutaneous administration. Ann Oncol 2010;21(8):viii78–viii95, abstract 218PD.

Yin A, Li J, Hurst D et al. Population pharmacokinetics (PK) and association of PK and clinical outcomes of rituximab in patients with non-Hodgkin's lymphoma. J Clin Oncol 2010;28:(suppl; abstract e13108) [Published in conjunction with the ASCO 2010 Annual Meeting].

SAS Institute Inc., Cary, NC, USA, version 9.

MedDRA – Medical Dictionary for Regulatory Activities. International Federation of Pharmaceutical Manufacturers Associations (IFPMA), c/o TRW, VAR1/8A/MSSO, 12011 Sunset Hills Road, Reston, VA 20190-3285, USA.

WHO – Drug Dictionary. World Health Organization Collaborating Center for International Drug Monitoring, P.O. Box 26, S-751 03 Uppsala, Sweden.

EMEA, ICH Harmonised Guideline (1998), Statistical Principles for Clinical Trials.

Clinical Study Protocol ML28964, version 3.1, 07 February 2016.

# Appendix 1 - Protocol Synopsis

TITLE: AN OPEN-LABEL, MULTINATIONAL, MULTICENTER,

PHASE IIIB STUDY TO ASSESS SAFETY OF RITUXIMAB FOLLOWING SUBCUTANEOUS ADMINISTRATION IN PATIENTS WITH CD20+ DLBCL OR CD20+ FOLLICULAR

**NHL GRADE 1 TO 3A** 

PROTOCOL NUMBER: ML28964

VERSION NUMBER: 3.1

EUDRACT NUMBER: {Number}
IND NUMBER: N/A

**TEST PRODUCT:** Rituximab (RO 45-2294)

PHASE: IIIb

INDICATION: CD20+ diffuse large B-cell lymphoma or CD20+ follicular non-

Hodgkin's lymphoma grade 1 to 3a

**SPONSOR:** Roche Algeria,

**Objectives** 

## **Primary Objective**

- To evaluate the incidence of administration-associated reactions (AARs) following multiple doses of subcutaneous (SC) rituximab during Induction and/or Maintenance therapy in patients with CD20+ follicular non-Hodgkin's lymphoma (NHL) or CD20+ diffuse large B-cell lymphoma (DLBCL) who have previously received at least one dose of intravenous (IV) rituximab.
- AARs are defined as all adverse events (AEs) occurring within 24 hours of rituximab SC administration and which are considered related to study drug. AARs include infusion/injectionrelated reactions (IIRRs), injection-site reactions, administration site conditions and all symptoms thereof.

## **Secondary Objectives**

- To evaluate patient-reported outcomes in terms of Rituximab Administration Questionnaire (RASQ)
- To further evaluate the safety of rituximab SC in terms of:
  - Grade ≥ 3 AEs
  - Grade ≥ 3 AARs
  - Serious adverse events (SAEs)
- To evaluate the efficacy of rituximab SC in terms of:
  - event-free survival (EFS)
  - progression-free survival (PFS)
  - Overall survival (OS).
  - disease-free survival (DFS)
  - complete response (CR) rate, including complete response unconfirmed (CRu), 4 weeks after the last dose of Induction treatment
- To evaluate healthcare professional outcomes in terms of:
  - HCP (Healthcare Professional) Questionnaire

## **Other Objectives**

Not applicable

Study Design

# **Description of Study**

This is an open-label, single-arm study to evaluate the safety of rituximab SC administered during first line treatment for FL (Induction and/or Maintenance therapy plus 24 months of follow up), or DLBCL (treatment plus 24 months of follow-up).

#### Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

Mabrella ML28964 Daughter Protocol 46/Statistical Analysis Plan ML28964

This study will include adult patients with CD20+ DLBCL or CD20+ follicular NHL (grade 1 to 3a; NHL), who have already received at least one full dose of IV rituximab during first-line treatment, induction or maintenance.

During administration of rituximab SC, patients will be assessed for safety and efficacy as detailed in the **Schedule of Assessments** (see **Appendix 1**). The Rituximab Administration Questionnaire (RASQ, **Appendix 6**) will be applied to patients and Healthcare Professional (HCP) Questionnaire (see **Appendix 7**) will be applied to health care professionals at the end of the study.

#### Induction Therapy:

NHL patients receiving Induction therapy prior to entry into the study must be eligible to receive at least four further cycles of rituximab SC (i.e. 4 additional months of Induction treatment). Patients with follicular NHL who will continue into Maintenance therapy (after staging at the end of Induction) can continue to receive rituximab SC during Maintenance (see below).

Maintenance Therapy (patients with follicular NHL):

NHL patients receiving Maintenance therapy prior to entry into the study must be eligible to receive at least six further cycles of rituximab SC (i.e. 12 additional months of Maintenance treatment).

Patients who are continuing into Maintenance therapy following at least 4 (four) cycles of rituximab SC during Induction Therapy must also be eligible to receive at least six cycles of rituximab SC (i.e. 12 additional months of Maintenance treatment).

Figure 1 Study duration: Patients with CD20+ Follicular NHL



Figure 2 Study duration: Patients with CD20+ DLBCL



#### **Number of Patients**

A sample size of 110 patients is deemed sufficient for this study. In this study, all planned statistical analysis will be exploratory in nature as the study will not be powered to address any pre-defined statements and only descriptive statistical evaluations will be carried out primarily for safety (and efficacy) parameters. Additionally, no published reference is available on administration-associated reactions (AARs) following multiple doses of subcutaneous (SC) rituximab during induction and/or maintenance therapy in patients with CD20+ follicular non-Hodgkin's lymphoma (NHL) or CD20+ diffuse large B-cell lymphoma (DLBCL). However, with 110 patients a 95% Clopper-Pearson CI for the incidence of AARs will be no wider than +/- 9.7%. This width of interval is deemed sufficiently precise to draw valid conclusions around the incidence of ARRs. Additionally, enrolment of more than 110 patients within the specified indications could also be difficult in participating countries.

Due to the fact of exploratory nature of the study, drop out patients will not be replaced.

#### **Target Population**

The target population will consist of adults with CD20+ DLBCL or CD20+ follicular NHL grade 1 to 3a, according to the World Health Organization (WHO) classification system.

#### Inclusion Criteria

Patients must meet the following criteria for study entry:

- 1. Signed, written informed consent form
- 2. Age  $\geq$  18 and  $\leq$  80 years at time of enrolment
- 3. Histologically confirmed, CD20+ DLBCL or CD20+ follicular NHL grade 1 to 3a, according to the WHO classification system
- 4. Currently being treated with rituximab IV in the Induction or Maintenance setting, having received at least one full dose of rituximab IV, defined as standard full dose of rituximab IV 375 mg/m² administered without interruption or early discontinuation because of tolerabilityissues
- 5. Expectation and current ability for the patient to receive at least four additional cycles of treatment during the Induction phase and six additional cycles of treatment during the Maintenance phase (patients with follicular NHL)
- 6. Induction only: An International Prognostic Index (IPI) score of 1-4 or IPI score of 0 with bulky disease, defined as one lesion ≥ 7.5 cm, or Follicular Lymphoma International Prognostic Index (FLIPI) (low, intermediate or high risk) (see **Appendix 3**)
- 7. Induction only: At least one bi-dimensionally measurable lesion defined as ≥ 1.5 cm in its largest dimension on computed tomography (CT) scan
- 8. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3 (see Appendix 3)
- 9. Patients with CD20+ DLBCL eligible for R-CHOP regimen
- 10. Patients with LVEF >55%

#### **Exclusion Criteria**

Patients who meet any of the following criteria will be excluded from study entry:

## Cancer-Related Criteria

- 1. Transformed lymphoma (i.e., histologic evidence of transformation to a Burkitt lymphoma) or follicular lymphoma (FL) Grade IIIB
- 2. Primary central nervous system lymphoma, primary effusion lymphoma, primary mediastinal DLBCL, DLBCL of the testis, or primary cutaneous DLBCL
- 3. History of other malignancy that could affect compliance with the protocol or interpretation of results. This includes a malignancy that has been treated but not with curative intent, unless the malignancy has been in remission without treatment for ≥ 5 years prior to dosing. Note: Patients with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix are eligible for the study.

### Prior or Concomitant Treatments

4. On-going corticosteroid use > 30 mg/day of prednisone or equivalent. Note: patients receiving corticosteroid treatment with ≤ 30 mg/day of prednisone or equivalent must be documented to be on a stable dose of at least 4 weeks' duration prior to dosing.

# Laboratory Assessments at Screening

- 5. Inadequate renal function, defined as:
  - Creatinine > 1.5 times the upper limit of normal (ULN) (unless normal creatinine clearance), or calculated creatinine clearance < 40 mL/min (using the Cockcroft-Gault formula)</li>
- 6. Inadequate hematologic function, defined as:
  - Hemoglobin < 9 g/dL
  - Absolute neutrophil count < 1.5 x 109/L
  - Platelet count < 75 x 109/L

- 7. Inadequate hepatic function, defined as:
  - Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN
  - Total bilirubin ≥ 1.5 x ULN. Note: patients with documented Gilbert disease may be enrolled if total bilirubin is ≤ 3.0 x ULN

#### Other Prior or Current Medical Conditions or Treatments

- 8. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
- 9. For patients with FL and DLBCL Contraindication to any of the individual components of CHOP (cyclophosphamide, vincristine, doxorubicin and prednisone), including prior receipt of anthracyclines
- 10. Other serious underlying medical conditions, which, in the Investigator's judgment, could impair the ability of the patient to participate in the study (e.g., significant cardiovascular disease, uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease)
- 11. Recent major surgery (within 4 weeks prior to dosing, other than for diagnosis
- 12. Active and/or severe bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics except if for tumour fever) within 4 weeks prior to dosing
- 13. Active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection (must be ruled out during Screening)
- 14. History of human immunodeficiency virus (HIV) seropositive status

#### General Criteria

- 15. Inability to provide informed consent and comply with protocol requirements.
- 16. Life expectancy of less than 6 months
- 17. A positive serum pregnancy test in women of childbearing potential within 7 days prior to dosing or within 14 days if with a confirmatory urine pregnancy test within 7 days prior to dosing. Women of childbearing potential are defined as pre-menopausal women or women who are < 2 years after the onset of menopause and are not surgically sterile.
- 18. Fertile men or women of childbearing potential who do not agree to use a highly effective measure of contraception (such as oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) throughout the study and for at least 12 months after the last dose of rituximab.

#### **Length of Study**

Assessments of this study will be performed according to the type of lymphoma (either FL or DLBCL). Since assessments for FL patients are expected to be on-study longer, this portion of the study will be determinative for the length of the study. For FL patients the study is estimated to take approximately 6 years (68 months) based on an approximately 12 month of recruitment period, 8 months of induction and 24 months of maintenance treatment and 24 months of follow-up period.

On the other hand, DLBCL patients are expected to be on-study for a shorter period of time (approximately in 4 years), based on approximately 12 month recruitment, 8 months of treatment and 24 months follow up period.

## **End of Study**

The end of the study, defined as last patient last visit (LPLV), will occur 24 months after the last SC rituximab treatment for the last FL or DLBCL patient, whichever comes later.

- FL patients who complete induction treatment will then enter the maintenance phase. Following the last SC rituximab administration, FL patients will be followed up for 24 months.
- DLBCL patients who receive their last SC rituximab treatment will then enter the post-treatment follow-up phase.
- Patients with SD or PD at staging will be withdrawn from study treatment and will only be followed AEs and for survival until the end of the study.
- Patients who do not complete the Induction treatment per protocol will undergo end-oftreatment assessment within 4 weeks after the last dose of Induction treatment and will be followed until the end of the whole study according to local practice for AEs, tumour response / progression (if PD not yet documented), survival, and documentation of any new antilymphoma treatment.

 Patients who complete the study or discontinue from the study early will be asked to return to the clinic (after 28 days or at least 5 half-lives of any non-rituximab IMPs, whichever longer) after the last dose of study drug for a follow-up visit.

#### **Safety Outcome Measures**

Safety outcomes will include AARs (defined as all related AEs occurring within 24 hours of rituximab SC administration including IIRRs, administration site conditions and all symptoms thereof), grade ≥ 3 AEs, and SAEs. Other safety assessments include routine safety laboratory tests, vital signs measurements and changes in concomitant medications. All clinical AEs and SAEs as well as laboratory abnormalities will be recorded regardless of their intensity / grading. Grading will be completed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.

#### **Efficacy Outcome Measures**

Tumour assessments will be done according to the protocol schedule of assessments (See Appendix 1-Appendix 2).

Tumour assessments will be based on CT scans of the neck, chest, abdomen and/or pelvis (if detectable by these techniques) or other diagnostic means (e.g. magnetic resonance imaging [MRI]) where applicable. Other methods (e.g. MRI) are acceptable for patients in whom CT scans are contraindicated. The CT scan used for eligibility assessments may be performed up to 28 days prior to dosing.

Response assessments 4-6 weeks after the last dose of Induction treatment will be based on the Investigator's assessment, completed according to the International Working Group (IWG) response criteria (Cheson et al. 1999, see Appendix 2).

The efficacy of rituximab SC will be evaluated during Induction and/or Maintenance in terms of EFS, PFS, OS, CR/CRu, and DFS.

The endpoints of EFS, PFS and OS will be defined and analysed twice using two different starting points for the time-to-event calculations. The first starting point will be first dose of rituximab IV and the second will be first dose of rituximab SC.

EFS is defined as the time from first dose of rituximab (analysed using both first dose of IV and first dose of SC) to first occurrence of progression or relapse, according to the IWG response criteria (Cheson et al. 1999, see <a href="Appendix 2">Appendix 2</a>) or initiation of a non–protocol-specified anti-lymphoma therapy or death, whichever occurs first.

PFS is defined as the time from first dose of rituximab (analysed using both first dose of IV and first dose of SC) to the first occurrence of progression or relapse, according to the IWG response criteria (Cheson et al. 1999, see **Appendix 2**) or death from any cause.

OS is defined as the time from first dose of rituximab (analysed using both first dose of IV and first dose of SC) to death from any cause.

DFS will be assessed in patients achieving CR/CRu and is defined as the period from the date of the initial CR/CRu until the date of relapse or death from any cause.

CR/CRu is complete response or complete response unconfirmed and is measured 4 weeks after the last dose of Induction treatment.

# **Exploratory Outcome Measures**

Not applicable

#### Pharmacodynamic and Pharmacokinetic Outcome Measures

Not applicable

#### **Pharmacoeconomic Outcome Measures**

Not applicable

#### **Patient-Reported Outcome Measures**

Patient satisfaction with administration of treatment will be evaluated using the RASQ (see **Appendix 6**) after the rituximab IV administration, after last Rituximab SC in induction and after last Rituximab SC in maintenance. The RASQ will be completed immediately after rituximab administration and before chemotherapy administration in case the patient will receive chemotherapy. Patients prematurely discontinuing treatment during the study should complete the questionnaire at time of

discontinuation, as long as they had been administered at least one dose of treatment via both administration routes.

## **Healthcare Professional Reported Outcome Measures**

At the end of the study, healthcare professional (HCP) questionnaire (see Appendix 7) will be applied to healthcare professionals such as hematologists, internists, nurses or other healthcare professionals who administered rituximab SC.

## **Study Drug and Study Treatment**

The term "study drug" will be used throughout the protocol to refer to rituximab SC. The term "study treatment" will be used to refer to protocol-mandated treatment (also including background chemotherapy and/or other pre-medications).

## **Investigational Medicinal ProductsTest Product**

**Rituximab SC** - The rituximab SC dose is 1400 mg for all patients, independent of patient body surface area (BSA). This translates into an injection volume of 11.7 mL.

Each administration will consist of a single SC injection of rituximab 1400 mg independent of BSA.

**Induction therapy:** rituximab SC will always be administered **prior** to the selected chemotherapy regimen (with the exception of the corticosteroid component in CHOP regimens), on average of once a month for a minimum of four cycles.

**Maintenance therapy (patients with follicular NHL)**: rituximab SC will be administered at 2-month intervals for a minimum of six cycles, according to local standards of care.

#### Comparator

Not applicable.

#### **Non-Investigational Medicinal Products**

<u>Background therapy:</u> Commercially available chemotherapy will be used in combination with rituximab SC, as per standard local practice. For further details, see the local prescribing information for CHOP, CVP or FC.

<u>Concomitant therapy:</u> Patients should receive full supportive care, such as granulocyte colony-stimulating factor (G-CSF) support, transfusions of blood and blood products, prophylactic antiviral medication, antibiotics, anti-emetics, or local application of radiotherapy for consolidation after induction, as applicable and according to institutional standards. Mesna (2-Mercapto Ethane Sulfonate sodium) may be used as prophylaxis of haemorrhagic cystitis.

<u>Pre-medication:</u> In order to reduce the incidence and severity of IIRRs, it is recommended that all patients receive the following premedication administered 30-60 minutes prior to each rituximab administration:

- paracetamol (acetaminophen)
- diphenhydramine hydrochloride or alternative antihistamine.

<u>Tumor Lysis Syndrome Prophylaxis:</u> TLS prevention may include hydration and prophylactic rasburicase (recombinant urate oxidase) in high-risk patients, hydration plus allopurinol or rasburicase for intermediate-risk patients, and close monitoring of electrolyte abnormalities for low-risk patients. Primary management of established TLS involves similar recommendations, with the addition of aggressive hydration and diuresis, plus allopurinol or rasburicase for hyperuricemia.

#### **Statistical Methods**

The analysis of this study will be exploratory and will primarily make use of descriptive statistical methods. In addition, exploratory statistical testing and modeling will be used to highlight interesting aspects of the data. All tests will be two-sided and carried out with a 5%  $\alpha$ -error rate without correction for multiplicity.

All enrolled patients who receive at least one dose of study medication will be included in the Safety Population, which will be the primary analysis population for safety parameters. All enrolled patients will be included in the Intent-to-Treat Population, which will be the primary analysis population for efficacy parameters. Other analysis populations may be defined based on more restrictive criteria, such as fulfillment of eligibility criteria or a minimum duration of the observation period.

### **Endpoint and Analysis**

Safety will be assessed on the following safety parameters: AARs, including IIRRs, AEs, AEs of grade ≥ 3, SAEs, routine laboratory parameters, vital signs, concomitant medications, premature withdrawal from the study and from study medication due to AEs or ECOG performance status.

The incidence of AARs AEs, AEs leading to premature discontinuation or interruption of study treatment, SAEs, grade ≥ 3 AEs will be estimated with 95%-Clopper-Pearson confidence intervals. The incidence of each AE will be summarized by the primary system-organ class and by preferred term. The incidence of deaths and cause of deaths will be listed and summarized.

Laboratory parameters will be summarized and selected laboratory parameters may also be displayed graphically.

Vital signs will be summarized over time.

ECOG performance status will be summarized by frequency tables over time and percentage of patients in different categories will be presented by bar charts at different time points.

Concomitant medication will be coded according to the WHO DRUG dictionary and tabulated in summary tables.

All safety analyses will be based on the Safety population.

The analysis of endpoints measured as a time to event (EFS, PFS, OS and DFS) is based on the survivor function, which is the probability of remaining event-free beyond a certain point in time. The survivor function will be estimated using Kaplan-Meier methodology and summarized using the range, the 25th and 75th percentiles and median survival along with a 95% confidence interval for median survival.

Endpoints resulting in an incidence rate (e.g., CR/CRu) will be summarized with a 95% Clopper- Pearson confidence interval.

#### **Determination of Sample Size**

A sample size of 110 patients is deemed sufficient for this study. In this study, all planned statistical analysis will be exploratory in nature as the study will not be powered to address any pre-defined statements and only descriptive statistical evaluations will be carried out primarily for safety (and efficacy) parameters. Additionally, no published reference is available on administration-associated reactions (AARs) following multiple doses of subcutaneous (SC) rituximab during induction and/or maintenance therapy in patients with CD20+ follicular non-Hodgkin's lymphoma (NHL) or CD20+ diffuse large B-cell lymphoma (DLBCL). However, with 110 patients a 95% Clopper-Pearson CI for the incidence of AARs will be no wider than +/- 9.7%. This width of interval is deemed sufficiently precise to draw valid conclusions around the incidence of ARRs. Additionally, enrolment of more than 110 patients within the specified indications could also be difficult in participating countries. Due to the fact of exploratory nature of the study, drop out patients will not be replaced.

## **Interim Analyses**

Not applicable

#### Study procedures

See Schedule of Assessments, Appendix 1 and Appendix 2.

Appendix 2 - Schedule of Assessments

# SCHEDULE OF ASSESSMENTS FOR PATIENTS WITH CD20+ FOLLICULAR NHL

| Study Period | Screening | | | | | , | | | | | | | | | | | , | | | | | I | EOT | F/UP | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | /Baseline | | | Indu | ıctio | n (cy | /cies | 5) | | | | | Ma | ınt | en | anc | e ( | сус | les | ) | | • | 4-6w<br>after | Every 3m<br>(year 1) | End of |
| Timing / Assessments | D -28 to<br>D -1 | 1[a] | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Final<br>Staging | 1 | 2 | 3 | 4 | 5 | 6 7 | ' 8 | 9 | 1 0 | 1 | 12 | | last<br>dose<br>of SC<br>Rit | • Every 6m (year 2) | Study<br>Visit |
| Written informed consent [b] | Х | | | | | | | | | | | | | | | | | | | | | | | | |
| Demographic data | Х | | | | | | | | | | | | | | | | | | П | | | | | | |
| Medical history | х | | | | | | | | | | | | | | | | | | П | | | | | | |
| Follicular NHL diagnosis and WHO Classification [c] | х | | | | | | | | | | | | | | | | | | | | | | | | |
| Documentation of/testing for HIV, active hepatitis and other infections [d] | х | | | | | | | | | | | | | | | | | | | | | | | | |
| Tumour evaluation [e] | х | | | | | | | | | х | | | П | T | 1 | T | T | | П | | | | Х | Х | Х |
| Physical examination, infection assessment, vital signs [f] | X<br>X | | х | х | x | х | х | x | x | х | х | x | x | x | X | x | x | X | X | X | X | | х | х | х |
| Height and weight | Х | | | | | | | | | X | | | П | 1 | 1 | T | T | | П | | | | | | |
| 12-lead ECG | Х | | | | | | | | | | | | П | 1 | 1 | T | T | | П | | | | | | |
| FLIPI score [g] | Х | | | | | | | | | | | | П | 1 | 1 | T | T | | П | | | | | | |
| ECOG performance status [h] | Х | | | | | | | | | | | | П | 1 | 1 | T | T | | П | | | | | | |
| Serum pregnancy test [i] | х | | | | | | | | | | | П | П | 7 | 7 | T | T | T | П | | | | | | |
| Laboratory: Haematology,<br>Biochemistry, Coagulation tests [j] | х | | x | x | x | х | х | x | x | х | X | X | X | X | X | хх | x | X | X | X | X | | X | Х | х |

| Study Period | Screening | | | Indu | ıctio | n (c\ | cles | ;) | | | | ı | Mai | nte | ena | nce | e (c | vc | les | ) | | EOT | F/UP | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Timing / Assessments | D -28 to | 1[a] | | | | | | | 8 | Final<br>Staging | 1 | | | | | | | | ı | | 12 | 4-6w after last dose of SC Rit | Every 3m<br>(year 1)<br>• Every<br>6m<br>(year 2) | End of<br>Study<br>Visit |
| Study Treatment (minimum doses) | Х | | | | | Х | X | Х | Х | | | | T | Т | Ī | X | X | X | X | X | X | | | |
| Adverse event recording [k] | X | | Х | Х | Х | х | Х | х | х | Х | X | X | X Z | x > | ( ) | x | х | X | х | X | Х | х | Х | Х |
| Concomitant treatments & therapies | X | | Х | Х | Х | Х | X | Х | х | Х | X | X | X | x > | ( X | x | X | X | X | X | X | х | Х | Х |
| RASQ [i] | Х | | | | | | | | | Х | | | 1 | T | T | | | П | Ī | | | х | | |
| HCP Questionnaire [m] | | | | | | | | | | | | | 1 | T | Ī | | | П | | | | Х | | |
| Survival | | · | | | | | | | | Х | | | | | | | | | | | | Х | Х | Х |

- a. Patients must have previously received at least one cycle of IV rituximab before enrolment. All Screening/Baseline assessments could have been performed at the IV cycle visit.
- b. Signed informed consent must be obtained prior to any study-required Screening/Baseline assessments.
- c. Diagnosis of follicular NHL before treatment must have included histological diagnosis and initial CD20 expression confirmation.
- d. Patients known to have active hepatitis C, active hepatitis B, history of HIV seropositive status, or signs or symptoms of other active and/or severe infection must not be included in the study. Serology should be performed according to clinical judgment before and during treatment with rituximab. Local guidelines for patient consent to viral testing must be adhered to.
- e. CT and MRI are currently the best available and most reproducible methods for measuring target lesions selected for response assessment. Conventional CT or MRI should be performed according to institutional standards. Tumour assessment will be based on CT scans of the neck, chest, abdomen and pelvis, as applicable. CT scan with contrast is the recommended technique. However, MRIs of the chest, abdomen, and pelvis with a non-contrast CT scan may be used in patients for whom CT scans with contrast are contraindicated (i.e., patients with contrast allergy or impaired renal clearance). Owing to the global nature of this study, and due to limited availability of FDG-PET scanners, an FDG-PET scan cannot be mandated. The CT scan used for eligibility assessment may be performed up to 28 days before first dose of study medication. The end-of-treatment response assessment including radiology/imaging report must be obtained 4 weeks after the last dose of Induction treatment. Response should be determined on the basis of radiographic and clinical evidence of disease according the IWG guidelines (Cheson et al. 1999; see Appendix 2), or if not applicable, institutional standards should be used for tumour evaluation. Disease progression will be evaluated by the Investigator according to the IWG response criteria for NHL (Cheson et al. 1999; see Appendix 2) or other country standards until PD. Subsequent bone marrow assessments are required to confirm any suspected CR in patients with bone marrow involvement at baseline.
- f. As part of physical exam, SC injection sites will be checked at every treatment visit. As part of tumour assessments, physical examinations should also include the evaluation of the presence and degree of enlarged lymph nodes, hepatomegaly, and splenomegaly. Patients should be assessed for presence of active infections throughout the treatment periods. Vital signs assessment includes resting heart rate, body temperature and blood pressure.
- g. FLIPI score determined at Baseline (prior to Cycle 1). Where possible, the baseline FLIPI score should be calculated from the patient notes. Missing FLIPI scores will not preclude enrolment. See Appendix 3.
- h. ECOG performance status needs to be ≤ 3 for inclusion of the patient into the study. See Appendix 3.

## Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

- i. Women of childbearing potential (defined as pre-menopausal women or women who are < 2 years after the onset of menopause and not surgically sterile) must undergo serum pregnancy test within 7 days prior to first dose or within 14 days if with a confirmatory urine pregnancy test within 7 days prior to dosing.
- j. Haematology parameters will include haemoglobin, RBC, WBC count and differential, and platelet count. Biochemistry parameters at Screening will include sodium, potassium, ALT/SGPT, AST/SGOT, total bilirubin, serum creatinine, alkaline phosphatase, albumin, BUN, C-reactive protein and LDH. Biochemistry parameters at any further timepoint during the study will include sodium, potassium, ALT/SGPT, AST/SGOT, total bilirubin, and serum creatinine. Coagulation tests will include: INR, PT, and aPTT. The results from the safety laboratory assessments must be available on treatment days, prior to the rituximab administrations.
- k. After informed consent has been obtained but prior to dosing, only SAEs caused by a protocol-mandated intervention should be reported (e.g. SAEs related to invasive procedures such as biopsies). All clinical and laboratory AEs reported during the study will be documented and graded using the NCI CTCAE criteria, version 4.0. Special attention should be given to any acute infusion-related toxicities. After initiation of study drug, all AEs/SAEs, regardless of relationship to study drug, will be reported until study closure.
- I. Patient reported outcomes: All patients will be required to complete the Rituximab Administration Questionnaire (RASQ, see Appendix 6) at the end of the study. Patients prematurely discontinuing study treatment should complete the questionnaire at time of discontinuation, as long as they had taken at least one dose via each treatment route (IV and SC) post-randomization. RASQ will be completed immediately after rituximab administration and before chemotherapy administration.
- m. Healthcare Professional (HCP) Questionnaire (see Appendix 7) will be completed at the end of the study by healthcare professionals such as haematologists, internists, nurses or other healthcareprofessionals who administered rituximab SC during the study.

## SCHEDULE OF ASSESSMENTS FOR PATIENTS WITH CD20+ DLBCL

| Study Period | Screening / Baseline | | | | | | cles | | | | | | | nent Fo | | р | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Timing / Assessments | D -28 to<br>D -1 | 1[a] | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Final<br>Staging | 1-3 | 3-6 | 6-9 | 9-122 | 12-18 | 18-24 | End of Study Visit |
| Written informed consent [b] | X | | | | | | | | | | | | | | | | |
| Demographic data | Х | | | | | | | | | | | | | | | | |
| Medical history | Х | | | | | | | | | | | | | | | | |
| DLBCL diagnosis and WHO Classification [c] | х | | | | | | | | | | | | | | | | |
| Documentation of/testing for HIV, active hepatitis and other infections [d] | х | | | | | | | | | | | | | | | | |
| Tumour evaluation [e] | х | | | | | | | | | X | Х | Х | Х | Х | Х | Х | х |
| Physical examination, infection assessment, vital signs [f] | X<br>X | | х | x | x | X | х | x | х | х | X | х | х | х | Х | Х | х |
| Height and weight | X<br>X | | | | | | | | | х | | | | | | | |
| 12-lead ECG | Х | | | | | | | | | | | | | | | | |
| IPI score [g] | Х | | | | | | | | | | | | | | | | |
| ECOG performance status [h] | Х | | | | | | | | | X | | | | | | | |
| Serum pregnancy test [i] | Х | | | | | | | | | | | | | | | | |
| Laboratory: Haematology,<br>Biochemistry, Coagulation tests [j] | X<br>X | | X | X | X | X | x | X | x | х | X | X | X | X | | | x |
| Study Treatment | | | | | | X | X | X | X | | | | | | | | |
| Adverse event recording [k] | Х | | X | X | X | X | х | X | Х | x | X | Х | х | Х | | | х |

| Study Period<br>Visit | Screening<br>/ Baseline | | т | reat | mer | nt (cy | cles) | | | Final | | Post | -Treatn | nent Fo | llow-U | p | End of Study Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timing / Assessments | D -28 to<br>D -1 | 1[a] | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Staging | 1-3 | 3-6 | 6-9 | 9-122 | 12-18 | 18-24 | |
| Concomitant treatments & therapies | х | | X | x | x | X | X | x | x | х | x | X | х | X | X | Х | х |
| RASQ [I] | Х | | | | | | | | | Х | | | | | | | |
| HCP Questionnaire [m] | | | | | | | | | | Х | | | | | | | |
| Survival | | | | | | | | | | X | X | X | X | X | X | Х | х |

- a. Patients must have previously received at least one cycle of IV rituximab before enrolment. All Screening/Baseline assessments could have been performed at the IV cycle visit.
- b. Signed informed consent must be obtained prior to any study-required Screening/Baseline assessments.
- c. Diagnosis of diffuse large B-cell lymphoma before treatment must have included histological diagnosis and initial CD20 expression confirmation.
- d. Patients known to have active hepatitis C, active hepatitis B, history of HIV seropositive status, or signs or symptoms of other active and/or severe infection must not be included in the study. Serology should be performed according to clinical judgment before and during treatment with rituximab. Local guidelines for patient consent to viral testing must be adhered to.
- e. CT and MRI are currently the best available and most reproducible methods for measuring target lesions selected for response assessment. Conventional CT or MRI should be performed according to institutional standards. Tumour assessment will be based on CT scans of the neck, chest, abdomen and pelvis, as applicable. CT scan with contrast is the recommended technique. However, MRIs of the chest, abdomen, and pelvis with a non-contrast CT scan may be used in patients for whom CT scans with contrast are contraindicated (i.e., patients with contrast allergy or impaired renal clearance). Owing to the global nature of this study, and due to limited availability of FDG-PET scanners, an FDG-PET scan cannot be mandated. The CT scan used for eligibility assessment may be performed up to 28 days before first dose of study medication. The end-of-treatment response assessment including radiology/imaging report must be obtained 4 weeks after the last dose of Induction treatment. Response should be determined on the basis of radiographic and clinical evidence of disease according the IWG guidelines (Cheson et al. 1999; see Appendix 2), or if not applicable, institutional standards should be used for tumour evaluation. Screening/Baseline bone marrow examinations should include biopsy and aspirate for morphology (flow studies are optional) for staging purposes unless it has been performed within 1 month prior to dosingand was done for the purpose of diagnosis and staging of DLBCL. Subsequent bone marrow assessments are required to confirm any suspected CR in patients with bone marrow involvement at baseline.
- f. As part of physical exam, SC injection sites will be checked at every treatment visit. As part of tumour assessments, physical examinations should also include the evaluation of the presence and degree of enlarged lymph nodes, hepatomegaly, and splenomegaly. Patients should be assessed for presence of active infections throughout the treatment periods. Vital signs assessment includes resting heart rate, body temperature and blood pressure.
- g. IPI (according to Shipp et al. 1993) score determined at Baseline (prior to Cycle 1). Where possible, the baseline IPI score should be calculated from the patient notes. Missing IPI scores will not preclude enrolment. See Appendix 3.
- h. ECOG performance status needs to be  $\leq 3$  for inclusion of the patient into the study. See Appendix 3.
- i. Women of childbearing potential (defined as pre-menopausal women or women who are < 2 years after the onset of menopause and not surgically sterile) must undergo serum pregnancy test within 7 days prior to first dose or within 14 days if with a confirmatory urine pregnancy test within 7 days prior to dosing.
- j. Haematology parameters will include haemoglobin, RBC, WBC count and differential, and platelet count. Biochemistry parameters at Screening will include sodium, potassium, ALT/SGPT, AST/SGOT, total bilirubin, serum creatinine, alkaline phosphatase, albumin, BUN, C-reactive protein and LDH. Biochemistry parameters at any

- further timepoint during the study will include sodium, potassium, ALT/SGPT, AST/SGOT, total bilirubin, and serum creatinine. Coagulation tests will include: INR, PT, and aPTT. The results from the safety laboratory assessments must be available on treatment days, prior to the rituximab administrations.
- k. After informed consent has been obtained but prior to dosing, only SAEs caused by a protocol-mandated intervention should be reported (e.g. SAEs related to invasive procedures such as biopsies). All clinical and laboratory AEs reported during the study will be documented and graded using the NCI CTCAE criteria, version 4.0. Specialattention should be given to any acute infusion-related toxicities. After initiation of study drug, all AEs/SAEs, regardless of relationship to study drug, will be reported until study closure.
- I. Patient reported outcomes: All patients will be required to complete the Rituximab Administration Questionnaire (see Appendix 6) at the end of the study. Patients prematurely discontinuing study treatment should complete the questionnaire at time of discontinuation, as long as they had taken at least one dose via each treatmentroute (IV and SC) post-randomization. RASQ will be comleted immediately after rituximab administration and before chemotherapy administration.
- m. Healthcare Professional (HCP) Questionnaire (see **Appendix 7**) will be completed at the end of the study by healthcare professionals such as haematologists, internists, nurses or other healthcare professionals who administered rituximab SC during the study.

Rituximab - Roche North Africa (Algeria, Morocco & Tunisia) Mabrella ML28964 Daughter Protocol 59/Statistical Analysis Plan ML28964

| Appendix 3 - Table and Listing Shells |
|---------------------------------------|

TABLE 14.1.1) ENROLLED BY COUNTRY AND SITE (ITT POPULATION)

| | All Patients<br>(N=xxx) |
|---------|-------------------------|
| Country | |
| Algeria | xx (x.x%) |
| Morocco | xx (x.x%) |
| Tunisia | xx (x.x%) |
| Site | |
| Site #1 | xx (x.x%) |
| Site #2 | xx (x.x%) |
| Site #3 | xx (x.x%) |
| Site | xx (x.x%) |
| Site n | xx (x.x%) |

TABLE 14.1.2) SUMMARY OF PATIENT DISPOSITION (ITT POPULATION)

| | Statistic | All Patients<br>(N=xx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|
| Intent-to-treat Population | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Safety Population | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Reason for Discontinuation treatment | | | | |
| Progression of Disease | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Adverse Event | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Pregnancy | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Patient request/Withdraw consent | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Investigator decision | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Lack of compliance | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Lost to Follow-up | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Death | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number of subjects who Continued to Maintenance Phase | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note(s): Percentages for the reasons for discontinuation are based on the number of subjects who discontinued. Other percentages are calculated based on number of subjects in ITT population.

TABLE 14.1.3) SUMMARY OF PROTOCOL DEVIATIONS (ITT POPULATION)

| Category Subcategory | Statis | stic | | atients<br>(N=xxx) | | DLBCL<br>(N=xx) | | FL<br>(N=xx) |
|---|---|---|---|---|---|---|---|---|
| Number of patients with at least one Protocol Deviation | n | (%) | xx | (xx.x%) | xx | (xx.x%) | xx | (xx.x% |
| Protocol Deviations | n | (용) | xx | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Reason 1 | n | (%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Reason 2 | n | (%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Reason 3 | n | (%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Number of patients with at least one major Protocol Deviation | n | (%) | XX | (xx.x%) | xx | (xx.x%) | xx | (xx.x% |
| Major Protocol Deviations | n | (%) | xx | (xx.x%) | XX | (xx.x%) | XX | (xx.x% |
| Reason 1 | n | (%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Reason 2 | n | (%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Reason 3 | n | (%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x% |
| Number of patients with at least one COVID-19 related Protocol Devia | tion n | (왕) | xx | (xx.x%) | xx | (xx.x%) | xx | (xx.x% |
| COVID-19 Protocol Deviations | n | (왕) | xx | (xx.x%) | XX | (xx.x%) | XX | (xx.x% |
| Reason 1 | n | (%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Reason 2 | n | (%) | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x% |
| Reason 3 | n | (%) | xx | (xx,x%) | XX | (xx.x%) | XX | (xx.x% |

Note(s): Percentages for the protocol deviations are based on the number of patients in ITT population in each group. Patients with multiple protocol deviations within the same category are counted only once under those categories. The same patient experiencing multiple protocol deviation criterion are counted under each criterion.

TABLE 14.1.4) SUMMARY OF DEMOGRAPHICS (ITT POPULATION)

| | | Statistic | All Patients (N=xxx) | DLBCL (N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|---|
| Age (Ye | ears) | | | | |
| 9- (- | , | n | XXX | XX | XX |
| | | Mean | XX.X | XX.X | xx.x |
| | | SD | xx.xx | XX.XX | x.xx |
| | | Minimum | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Maximum | XX.X | XX.X | XX.X |
| Sex | | | | | |
| Jen | Male | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Female | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ethnic | ity | | | | |
| | Hispanic (latino) | n (%) | xx (x.x%) | xx (x.x%) | xx (x.x%) |
| | Not Hispanic (non-latino)<br>Not Applicable as | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | per local regulations | n (%) | xx (x.x%) | xx (x.x%) | xx (x.x%) |
| | Other | n (%) | xx (x.x%) | xx (xx.x%) | xx (x.x%) |
| Childb | earing potential | | | | |
| | Yes | n (%) | xx (x.x%) | xx (x.x%) | xx (x.x%) |
| | No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Source: xxx.sas Run DDMMMYYYY

### Programming note:

This table (age and ethnicity variables) to be repeated stratified by sex (Male, Female).

TABLE 14.1.5) SERUM PREGNANCY TEST AT SCREENING (SAFETY POPULATION)

| | Statistic | All Patients<br>(N=xxx) | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Was the serum pregnancy test performed? | , | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Pregnancy test result# | | | | |
| Negative | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of patients in SAF population.

# Percentages are calculated relative to the total number of SAF patients who performed a serum pregnancy test at screening visit.

Source: XXXX.SAS, Run on DDMMMYYYY

TABLE 14.1.6) SUMMARY OF BASELINE CHARACTERISTICS - PART #1 (ITT POPULATION)

| | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|
| Height (cm) | | | | |
| - 3 - (- , | n | XXX | XX | XX |
| | Mean | XXX.X | xxx.x | xxx.x |
| | SD | x.xx | x.xx | x.xx |
| | Minimum | XXX.X | xxx.x | xxx.x |
| | Median | XXX.X | xxx.x | xxx.x |
| | Maximum | XXX.X | xxx.x | xxx.x |
| Weight (Kg) | | | | |
| | n | XXX | XX | XX |
| | Mean | XX.X | XX.X | xx.x |
| | SD | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Maximum | XXX.X | XXX.X | XXX.X |
| BMI (Kg/m^2) | | | | |
| | n | XXX | XX | xx |
| | Mean | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX |
| | Minimum | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Maximum | XX.X | XX.X | xx.x |

Source: xxx.sas Run DDMMMYYYY

#### Programming note:

This table to be repeated stratified by sex (Male, Female).

TABLE 14.1.7) SUMMARY OF BASELINE CHARACTERISTICS - PART #2 (ITT POPULATION)

\_\_\_\_\_

| | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|
| IPI Score | | | | |
| Low risk | n (%) | xx (xx.x%) | xx (xx.x%) | |
| Low intermediate risk | n (%) | xx (x.x%) | xx (xx.x%) | |
| High intermediate risk | n (%) | xx (xx.x%) | xx (xx.x%) | |
| High risk | n (%) | xx (x.x%) | xx (xx.x%) | |
| FLIPI Score | | | | |
| Low risk | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Intermediate risk | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| High risk | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Surgery/Procedure History | | | | |
| General | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lymphoma related | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Both | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Reproductive Status | | | | |
| Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note(s): Percentages for reproductive status are based on the number of female patients in that particular group.

Source: xxx.sas Run DDMMMYYYY

### Programming note:

This table (IPI Score, FLIPI Score, Surgery/Procedure history variables) to be repeated stratified by sex (Male, Female).

TABLE 14.1.8) DLBCL DIAGNOSIS (SAFETY POPULATION)

| | Statistic | DLBCL<br>(N=xxx) |
|---|---|---|
| How was the histological diagnosis obtained? | | |
| Fine needle aspiration | n (%) | xxx (xx.x%) |
| ore needle biopsy | n (%) | xxx (xx.x%) |
| Excisional/incisional biopsy of peripheral lymph node | n (%) | xxx (xx.x%) |
| CD20+ expression# | | |
| Jegative Tegative | n (%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of patients in SAF population.
# Percentages are calculated relative to the number of patients with a diagnosis obtained by means of a Fine Needle Aspiration method.

Source: XXXX.SAS, Run on DDMMMYYYY

TABLE 14.1.9) FOLLICULAR LYMPHOMA DIAGNOSIS (SAFETY POPULATION)

| | Statistic | FL<br>(N=xxx) |
|---|---|---|
| How was the histological diagnosis obtained? | | |
| Fine needle aspiration | n (%) | xxx (xx.x%) |
| Core needle biopsy | n (%) | xxx (xx.x%) |
| Excisional/incisional biopsy of peripheral lymph node | n (%) | xxx (xx.x%) |
| Grade of FL | | |
| Grade 1 | n (%) | xxx (xx.x%) |
| Grade 2 | n (%) | xxx (xx.x%) |
| Grade 3a | n (%) | xxx (xx.x%) |
| CD20+ expression | | |
| Negative | n (%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of patients in SAF population.

Source: XXXX.SAS, Run on DDMMMYYYY

TABLE 14.1.10) SUMMARY OF BONE MARROW AT BASELINE (ITT POPULATION)

| | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|
| Bone marrow assessment done | | | | |
| Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bone marrow assessment using aspirate | | | | |
| Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bone marrow assessment using aspirate result | | | | |
| Positive | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bone marrow assessment using biopsy | | | | |
| Yes | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bone marrow assessment using biopsy result | | | | |
| Positive | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Negative | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |

Percentages are calculated relative to the total number of patients in ITT population.

TABLE 14.1.11) LEAD ECG AT SCREENING (SAFETY POPULATION)

| | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Was 12-lead ECG performed? | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Overall evaluaton of ECG tracing# | | | | |
| Normal | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Abnormal, NCS | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Abnormal, CS | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

CS = Clically Significant.

NCS = Not Clinically Significant.

Percentages are calculated relative to the total number of patients in SAF population.

# Percentages are calculated relative to the total number of SAF patients who performed ECG at screening visit.

Source: XXXX.SAS, Run on DDMMMYYYY
TABLE 14.1.12) VIRAL SEROLOGY AT SCREENING (SAFETY POPULATION)

| | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Was the viral serology sample collected? | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Hepatitis B core antibody (HBcAb) | | | | |
| Negative | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not done | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Hepatitis B surface antigen (HBsAg) | | | | |
| Negative | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not done | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| HCV antibody | | | | |
| Negative | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not done | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| HCV antibody | | | | |
| Negative | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not done | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Does the patient have an active viral | | | | |
| infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)? | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of patients in SAF population.
# Percentages are calculated relative to the total number of SAF patients who performed a viral serology test at screening visit.

TABLE 14.1.13) SUMMARY OF PREVIOUS DISEASE (ITT POPULATION)

| System Organ Class<br>MedDRA Preferred Term | All Patients (N=xxx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|
| Number of patients with at least one previous disease | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| <pre><primary soc=""></primary></pre> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pre><primary soc=""></primary></pre> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pre><primary soc=""></primary></pre> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |

### Notes:

Percentages are calculated relative to the total number of patients in the ITT population. Medical History terms were coded using MedDRA thesaurus version 24.1.

Previous diseases are those not flagged as "Ongoing at study entry" in the CRF form. Patients can have more than one previous disease.

TABLE 14.1.14) SUMMARY OF CONCOMITANT DISEASE (ITT POPULATION)

| System Organ Class<br>MedDRA Preferred Term | All Patients<br>(N=xxx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|
| Number of patients with at least one concomitant disease | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| <pre><primary soc=""></primary></pre> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pre><primary soc=""></primary></pre> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pre><primary soc=""></primary></pre> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |
| <pt></pt> | xx (xx.x%) | xx (xx.x%) | x (xx.x%) |

### Notes:

Percentages are calculated relative to the total number of patients in the ITT population.

Medical History terms were coded using MedDRA thesaurus version 24.1.

Concomitant diseases are those flagged as "Ongoing at study entry" in the CRF form.

Patients can have more than one concomitant disease.

TABLE 14.1.15) SUMMARY OF PHYSICAL EXAMINATION (SAFETY POPULATION)

| Visit | Body System | All Patients (N=xxx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|
| xxx | Head Ears Eyes Nose Throat | | | |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, not clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Not applicable | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Cardiovascular system | | | |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, not clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Not applicable | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Dermatological | | | |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, not clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Not applicable | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Musculoskeletal system | | | |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, not clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Not applicable | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Respiratory system | | | |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, not clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Abnormal, clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Not applicable | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Genitourinary system | | | |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Gastrointestinal system | | | |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Nervous system | | | |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Other | | | |
| | Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note(s): Percentages are based on the number of patients in safety population at the specific visit.

Source: xxx.sas Run DDMMMYYYY

# Rituximab - Roche North Africa (Algeria, Morocco & Tunisia) Mabrella ML28964 Daughter Protocol 75/Statistical Analysis Plan ML28964

TABLE 14.1.16) SUMMARY OF PREVIOUS THERAPIES (SAFETY POPULATION)

| ATC Class Level 2<br>Other Treatment | Statistic | All Patients (N=xxx) | FL<br>(N=xxx) | DLBCL (N=xxx) |
|---|---|---|---|---|
| Total number of patients with at least one treatment | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total number of treatments | n | xxx | XXX | XXX |
| Class 1 | | | | |
| Total number of patients with at least one treatment | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total number of treatments | n | xxx | XXX | XXX |
| Other treatment 1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other treatment 2 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Class 2 | | | | |
| Total number of patients with at least one treatment | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total number of treatments | n | xxx | XXX | XXX |
| Other treatment 1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

### Notes:

Treatments are coded using the INN-1.0V dictionary.

Treatments can appear under multiple classes.

Multiple uses of a specific medication for a patient were counted once in the frequency for the medication. Likewise, multiple uses within a specific medication class for a patient were counted once in the frequency for the medication class.

For frequency counts in "Total number of treatments", multiple uses of the same medication for a patient were counted separately.

Patients can have more than one previous therapy. Previous therapy includes any medication stopped before exposure to study drug.

TABLE 14.1.17) SUMMARY OF CONCOMITANT THERAPIES (SAFETY POPULATION)

| ATC Class Level 2<br>Other Treatment | Statistic | All Patients (N=xxx) | FL<br>(N=xxx) | DLBCL<br>(N=xxx) |
|---|---|---|---|---|
| Total number of patients with at least one treatment | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total number of treatments | n | xxx | XXX | XXX |
| Class 1 | | | | |
| Total number of patients with at least one treatment | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total number of treatments | n | XXX | XXX | XXX |
| Other treatment 1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other treatment 2 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Class 2 | | | | |
| Total number of patients with at least one treatment | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total number of treatments | n | xxx | XXX | XXX |
| Other treatment 1 | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

### Notes:

Treatments are coded using the INN-1.0V dictionary.

Treatments can appear under multiple classes.

Multiple uses of a specific medication for a patient were counted once in the frequency for the medication. Likewise, multiple uses within a specific medication class for a patient were counted once in the frequency for the medication class.

For frequency counts in "Total number of treatments", multiple uses of the same medication for a patient were counted separately.

Patients can have more than one concomitant therapy. Concomitant therapy consists of any medication taken during the study, including those started before but ongoing at first dose of study drug.

TABLE 14.1.18) SUMMARY OF PREVIOUS IV RITUXIMAB DOSE FOR DLBCL (SAFETY POPULATION)

| | Statistic | DLBCL (N=xxx) |
|-------------------------------------------------|-----------|---------------|
| Number of previous IV rituximab treatment cycle | es | |
| One | n (%) | xxx (xx.x%) |
| Two | n (%) | xxx (xx.x%) |
| Three | n (%) | xxx (xx.x%) |
| Four | n (%) | xxx (xx.x%) |
| Dose of most recent IV rituximab cycle | | |
| | n | XXX |
| | Mean (SD) | xx.x (xx.x) |
| | Median | xx.x |
| | Min, Max | XX,XX |

TABLE 14.1.19) SUMMARY OF PREVIOUS IV RITUXIMAB DOSE FOR FL (SAFETY POPULATION)

| | Statistic | FL<br>(N=xxx) |
|---|---|---|
| What phase of IV Rituximab was the patient on for their most recent IV cycle? | | |
| Induction phase | n (%) | xxx (xx.x%) |
| Maintenance phase | n (%) | xxx (xx.x%) |
| Number of previous IV rituximab treatment cycles | | |
| One | n (%) | xxx (xx.x%) |
| Two | n (%) | xxx (xx.x%) |
| Three | n (%) | xxx (xx.x%) |
| Four | n (%) | xxx (xx.x%) |
| Five | n (%) | xxx (xx.x%) |
| Six | n (%) | xxx (xx.x%) |
| Seven | n (%) | xxx (xx.x%) |
| Eight | n (%) | xxx (xx.x%) |
| Dose of most recent IV rituximab cycle | | |
| | n | XXX |
| | Mean (SD) | xx.x (xx.x) |
| | Median | XX.X |
| | Min,Max | xx,xx |
| Which treatment phase is the subject eligible to enter the study? | | |
| Induction phase | n (%) | xxx (xx.x%) |
| Maintenance phase | n (%) | xxx (xx.x%) |

TABLE 14.1.20) EXPOSURE TO RITUXIMAB SC - ADMINISTRATION SUMMARY (SAFETY POPULATION)

| | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|
| Induction Cycle* | | | | |
| Induction Cycle 1 | n (%) | x (x.x%) | | x (x.x%) |
| Induction Cycle 2 | n (%) | x (x.x%) | | x (x.x%) |
| Induction Cycle | n (%) | x (x.x%) | | x (x.x%) |
| Induction Cycle n | n (%) | x (x.x%) | | x (x.x%) |
| Maintenance Cycle* | | | | |
| Maintenance Cycle 1 | n (%) | x (x.x%) | | x (x.x%) |
| Maintenance Cycle 2 | n (%) | x (x.x%) | | x (x.x%) |
| Maintenance Cycle | n (%) | x (x.x%) | | x (x.x%) |
| Maintenance Cycle n | n (%) | x (x.x%) | | x (x.x%) |
| Treatment Cycle* | | | | |
| Treatment Cycle 1 | n (%) | x (x.x%) | x (x.x%) | |
| Treatment Cycle 2 | n (%) | x (x.x%) | x (x.x%) | |
| Treatment Cycle | n (%) | x (x.x%) | x (x.x%) | |
| Treatment Cycle n | n (%) | x (x.x%) | x (x.x%) | |
| Total number of cycles | | | | |
| | n | XXX | XX | XX |
| | Mean | X.X | X . X | X.X |
| | SD | X.XX | X.XX | X.XX |
| | Minimum | X.X | X . X | X.X |
| | Median | X.X | X . X | X.X |
| | Maximum | xx.x | X.X | x.x |

Note(s): \*Number of Rituximab SC cycles exposure. Denominator for calculating the percentage is N (Safety population).

TABLE 14.1.21) EXPOSURE TO RITUXIMAB SC - ADMINISTRATION DETAILS (SAFETY POPULATION)

| | Statistic | All Patients DLBCL (N=xx) | FL<br>(N=xx) |
|---|---|---|---|
| Full Doses | | | |
| Overall | n (%) | xx (xx.x%) xx (xx.x%) | xx (xx.x%) |
| Full Doses in Induction Cycle | | | |
| Induction Cycle 1 | n (%) | x (x.x%) | x (x.x%) |
| Induction Cycle 2 | n (%) | x (x.x%) | x (x.x%) |
| Induction Cycle | n (%) | x (x.x%) | x (x.x%) |
| Induction Cycle n | n (%) | x (x.x%) | x (x.x%) |
| Full Doses in Maintenance Cycle | | | |
| Maintenance Cycle 1 | n (%) | x (x.x%) | x (x.x%) |
| Maintenance Cycle 2 | n (%) | x (x.x%) | x (x.x%) |
| Maintenance Cycle | n (%) | x (x.x%) | x (x.x%) |
| Maintenance Cycle n | n (%) | x (x.x%) | x (x.x%) |
| Full Doses in Treatment Cycle | | | |
| Treatment Cycle 1 | n (%) | x (x.x%) x (x.x%) | |
| Treatment Cycle 2 | n (%) | x (x.x%) x (x.x%) | |
| Treatment Cycle | n (%) | x (x.x%) x (x.x%) | |
| Treatment Cycle n | n (%) | x (x.x%) x (x.x%) | |

TABLE 14.1.22) EXPOSURE TO RITUXIMAB SC - ADMINISTRATION DETAILS (SAFETY POPULATION)

| | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|
| Ouration of Injection | | | | |
| | n | XXX | XXX | XXX |
| | Mean | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX |
| | Minimum | X.X | X.X | X.X |
| | Median | X.X | X.X | X.X |
| | Maximum | XX.X | xx.x | xx.x |
| ose Injected | | | | |
| xxxx mg | n (%) | xxxx (xx.x%) | xxx (xx.x%) | xxxx (xx.x%) |
| xxxx mg | n (%) | xxxx (xx.x%) | xxx (xx.x%) | xxxx (xx.x%) |
| xxxx mg | n (%) | xxxx (xx.x%) | xxx (xx.x%) | xxxx (xx.x%) |
| Interruption Duration* # | | | | |
| • | n | XXX | XXX | XXX |
| | Mean | x.x | x.x | x.x |
| | SD | x.xx | x.xx | x.xx |
| | Minimum | X.X | X.X | x.x |
| | Median | x.x | x.x | x.x |
| | Maximum | XX.X | XX.X | xx.x |

Note(s): #Interruption due to Serious Adverse Event/ Adverse Event of Special Interest.

TABLE 14.1.23) TYPE OF CHEMOTHERAPY (SAFETY POPULATION)

| Type of chemotherapy | Statistic | All Patients (N=xxx) | DLBCL (N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|
| CHOP-14 X 6 | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| CHOP-14 X 8 | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| CHOP-21 X 6 | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| CHOP-21 X 8 | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| CVP-21 X 8 | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| FC-28 X 6 | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| Other | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |

Note(s): Denominator for calculating the percentage is N (Safety population).

TABLE 14.1.24) EXPOSURE TO CHEMOTHERAPY (SAFETY POPULATION)

| Туре | | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|---|
| CHOP-14 X 6 | Induction Cycle | | | | |
| | 1 Induction Cycle | n (%) | x (x.x%) | | x (x.x%) |
| | 2 Induction Cycles | n (%) | x (x.x%) | | x (x.x%) |
| | n Induction Cycles | n (%) | x (x.x%) | | x (x.x%) |
| | Total number of cycles | | | | |
| | | n | xx | | XX |
| | | Mean | x.x | | X.X |
| | | SD | X.XX | | X.XX |
| | | Minimum | X.X | | X.X |
| | | Median | X.X | | X.X |
| | | Maximum | x.x | | x.x |

Note(s): Denominator for calculating the percentage is N (Safety population).

Source: xxx.sas Run DDMMMYYYY

## Programming note:

This table should be also presented for all chemotherapy regimen patient is taking.

TABLE 14.1.25) EXPOSURE TO NEW ANTI - LYMPHOMA TREATMENT CHEMO/IMMUNO THERAPY (SAFETY POPULATION)

| Туре | Statistic | All Patients<br>(N=xxx) | DLBCL<br>(N=xx) | FL<br>(N=xx) | |
|---|---|---|---|---|---|
| Chemo/Immuno Therapy | Total Number of Cycles | | | | |
| | 1 Cycle | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | 2 Cycles | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | n Cycles | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | Total number of cycles | | | | |
| | - | n | XX | XX | XX |
| | | Mean | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | x.xx |
| | | Minimum | X.X | X.X | X.X |
| | | Median | X.X | X.X | X.X |
| | | Maximum | XX.X | х.х | xx.x |
| | Duration of Exposure (days) | | | | |
| | | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XXX.X |
| | | SD | XX.XX | XX.XX | XX.XX |
| | | Minimum | X.X | X.X | XX.X |
| | | Median | XX.X | XX.X | XXX.X |
| | | Maximum | xxx.x | xxx.x | xxx.x |
| | Response | | | | |
| | CR | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | CRu | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | PR | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | SD | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | PD | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | Unable to assess | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |

Note(s): Denominator for calculating the percentage is  ${\tt N}$  (Safety population).

TABLE 14.1.26) INITIAL CHOP REGIMEN DOSAGE (SAFETY POPULATION)

| Study Treatment | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Cyclophosphamide (mg/m^2) | | | | |
| | n | xxx | xxx | xxx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | xx.x | xx.x | xx.x |
| | Min,Max | XX,XX | xx,xx | xx,xx |
| Doxorubicin (mg/m^2) | | | | |
| | n | XXX | xxx | XXX |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | xx.x | XX.X |
| | Min,Max | xx,xx | xx,xx | xx,xx |
| Vincristine (mg/m^2) | | | | |
| | n | XXX | xxx | XXX |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | xx.x | XX.X |
| | Min,Max | XX,XX | xx,xx | xx,xx |
| Prednisone/prednisolone (mg/m^2) | | | | |
| | n | xxx | xxx | xxx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | xx.x | XX.X |
| | Min,Max | xx,xx | xx,xx | xx,xx |

TABLE 14.1.27) INITIAL CVP REGIMEN DOSAGE (SAFETY POPULATION)

| Study Treatment | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL (N=xxx) |
|---|---|---|---|---|
| Cyclophosphamide (mq/m^2) | | | | |
| | n | xxx | xxx | xxx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | xx.x | xx.x |
| | Min,Max | XX,XX | XX,XX | XX,XX |
| Vincristine (mg/m^2) | | | | |
| | n | xxx | xxx | xxx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | xx.x | xx.x |
| | Min,Max | XX,XX | XX,XX | XX,XX |
| Prednisone/prednisolone (mg/m^2) | | | | |
| | n | XXX | xxx | xxx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | xx.x | XX.X | xx.x |
| | Min,Max | xx,xx | xx,xx | xx,xx |

TABLE 14.1.28) INITIAL FLUDARABINE DOSAGE (SAFETY POPULATION)

| Study Treatment | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Fludarabine (mg/m^2) | | | | |
| | n | xxx | xxx | xxx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | xx.x | xx.x | xx.x |
| | Min, Max | XX,XX | xx,xx | XX,XX |
| Cyclophosphamide (mg/m^2) | | | | |
| | n | xxx | xxx | xxx |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | xx.x | xx.x | xx.x |
| | Min,Max | xx,xx | xx,xx | xx,xx |

TABLE 14.1.29) EXPOSURE TO NEW ANTI - LYMPHOMA TREATMENT RADIOTHERAPY (SAFETY POPULATION)

| Туре | | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|---|
| Radiotherapy | Irradiation Site | | | | |
| 1.1 | Neck | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | Chest | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | Abdomen | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | Pelvis | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | Other | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | Cumulative Dose of Radiation (Gy) | | | | |
| | xx.xx Radiation | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | Cumulative Dose of Radiation (Gy) | Cumulative Dose of Radiation (Gy) | | | |
| | | n | XX | XX | XX |
| | | Mean | XX.XX | XX.XX | XX.XX |
| | | SD | X.XX | X.XX | X.XX |
| | | Minimum | XX.XX | XX.XX | XX.XX |
| | | Median | XX.XX | XX.XX | XX.XX |
| | | Maximum | XX.XX | xx.xx | xx.xx |
| | Duration of Exposure (days) | | | | |
| | | n | XX | XX | XX |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | X.XX | X.XX | X.XX |
| | | Minimum | XX.X | XX.X | XX.X |
| | | Median | XX.X | XX.X | XX.X |
| | | Maximum | XX.X | XX.X | XX.X |
| | Response | | | | |
| | CR | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | CRu | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | PR | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | SD | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | PD | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |
| | Unable to assess | n (%) | x (x.x%) | x (x.x%) | x (x.x%) |

Note(s): Denominator for calculating the percentage is N (Safety population).

TABLE 14.2.1) OVERALL SUMMARY OF PATIENTS EXPERIENCING EACH CLASS OF TREATMENT EMERGENT ADVERSE EVENT (SAFETY POPULATION)

| Events | Statistic | All Patients (N=xxx) | DLBCL (N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|
| Treatment Emergent Adverse Events | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| reatment Emergent Serious Adverse Events | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| dverse Events of Special Interest | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| dministration Associated Reactions | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| utaneous and soft tissue AARs (Localized) | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| utaneous and soft tissue AARs (Non-Localized) | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| rade >=3+ Treatment-Emergent Adverse Events | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| rade >=3+ Treatment-Emergent Serious Adverse Events | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| rade >=3+ Administration Associated Reactions | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| rade >=3+ Infusion/Injection-Related Reactions | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| EAEs leading to rituximab drug interrupted/drug delayed | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| EAEs leading to rituximab dose discontinuation | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| EAEs leading to chemotherapy dose modification | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| EAEs leading to chemotherapy dose discontinuation | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| EAEs leading to death | n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note(s): A patient experiencing multiple occurrences of an adverse event was counted, at most, once per Event.

TEAE = Treatment-Emergent Adverse Event.

TABLE 14.2.2) PROPORTION OF TREATMENT EMERGENT ADVERSE EVENT BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Number of patients with | | | | |
| Treatment Emergent Adverse<br>Event | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x,xx-%x,xx xxx xx,x%-xx,x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xx.xx) xxx | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x% | xxx (xx.x%) xxx xx.xx-xx.x% |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx,x%) xxx xx,x%-xx,x% | xxx (xx,x%) xxx xx,x%-xx,x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx,x%) xxx xx,x%-xx,x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%. Each patient is counted at most once within each SOC and PT.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.3) PROPORTION OF SERIOUS TREATMENT EMERGENT ADVERSE EVENT BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Number of patients with serious<br>Treatment Emergent Adverse | | | | |
| Event | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| (Primary SOC> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| (Primary SOC> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%. Each patient is counted at most once within each SOC and PT.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.4) PROPORTION OF LOCALIZED ADMINISTRATION ASSOCIATED REACTIONS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL (N=xxx) |
|---|---|---|---|---|
| Number of patients with | | | | |
| Localized AARs | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | *xxx (*x.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |

Note(s): MedDRA = Medical Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%.

Each patient is counted at most once within each SOC and PT.

TABLE 14.2.5) PROPORTION OF NON-LOCALIZED ADMINISTRATION ASSOCIATED REACTIONS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Number of patients with | | | | |
| Non-localized AARs | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.xx) xxx xx.xx-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.xx) xxx xx.xx-xx.xx | xxx (xx.x%) xxx xx.x%-xx.x% |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%. Each patient is counted at most once within each SOC and PT.

TABLE 14.2.6) PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ AES BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Number of patients with grade >=3+ TEAEs | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| 3 | , , | , | | |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.xx) xxx xx.xx-xx.xx |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.xx) xxx xx.xx-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.xx) xxx xx.xx-xx.xx |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.xx) xxx xx.xx-xx.xx | xxx (xx.x%) xxx xx.x%-xx.x% |

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%. Each patient is counted at most once within each SOC and PT.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.7) PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ SAES BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL (N=xxx) |
|---|---|---|---|---|
| Number of patients with | | | | |
| grade >=3+ serious TEAEs | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <pre><primary soc=""></primary></pre> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| Primary SOC> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| Primary SOC> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | *xx (*x.x*) xxx xx.x*-xx.x* |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%. Each patient is counted at most once within each SOC and PT.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.8) PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ AARS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL (N=xxx) |
|---|---|---|---|---|
| Number of patients with | | | | |
| grade >=3+ AARs | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.xx) | ***.xx (**.xx) **** |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.xx) | ***.xx (**.xx) **** |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%. Each patient is counted at most once within each SOC and PT.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.9) PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO RITUXIMAB DRUG INTERRUPTED/DRUG DELAYED BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL (N=xxx) |
|---|---|---|---|---|
| Number of patients with TEAE<br>leading to drug<br>Interruption/drug delayed | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | **.xx-**.xx | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | *xxx (*x.x*) xxx xx.x*-xx.x* | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | *xxx (*x.x*) xxx xx.x*-xx.x* | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x,xx-%x,xx xxx xx,x%-xx,x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.xx) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | *xxx (*x.x*) xxx xx.x*-xx.x* | *xx (*x.x*) xxx xx.x*-xx.x* |

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%. Each patient is counted at most once within each SOC and PT.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.10) PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO RITUXIMAB DOSE DISCONTINUATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients<br>(N=xxx) | DLBCL (N=xxx) | FL (N=xxx) |
|---|---|---|---|---|
| Number of patients with TEAE | | | | |
| leading to dose discontinuation | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | ** xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt> 1</pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%. Each patient is counted at most once within each SOC and PT.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.11) PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO CHEMOTHERAPY DOSE MODIFICATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL (N=xxx) |
|---|---|---|---|---|
| Number of patients with TEAE<br>leading to chemotherapy dose<br>modification | n (%) | xxx (%x.x%) | xxx (xx.x%) | xxx (%x.x%) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.xx) xxx xx.xx-xx.xx |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.xx) xxx xx.xx-xx.x% |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.xx) xxx xx.xx-xx.x% |
| <pre><primary soc=""></primary></pre> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%. Each patient is counted at most once within each SOC and PT.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.12) PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO CHEMOTHERAPY DOSE DISCONTINUATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Number of patients with TEAE<br>leading to chemotherapy dose<br>discontinuation | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pre><primary soc=""></primary></pre> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | *xx (*x.x*) xxx xx.x*-xx.x |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pre><primary soc=""></primary></pre> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | %x,xx-%x,xx xx,x%-xx,x% |

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%. Each patient is counted at most once within each SOC and PT.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.13) PROPORTION OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO DEATH BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| System Organ Class<br>Preferred Term | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL (N=xxx) |
|---|---|---|---|---|
| Number of patients with TEAE | | | | |
| leading to death | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | %x.xx-%x.xx xxx (%x.xx) xxx |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx,x%) xxx xx,x%-xx,x% | %x.xx-%x.xx xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx,x%) xxx xx,x%-xx,x% | %x.xx-%x.xx xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | **.xx (**.xx) |
| <primary soc=""></primary> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | %xxx (%x.x%) xxx xx.x%-xx.x% | xxx (xx.x%) xxx xx.x%-xx.x% |
| <pt></pt> | n (%) E 95% CI | xxx (xx.x%) xxx xx.x%-xx.x% | *xxx (*x.xx) xxx xx.x*-xx.x | xxx (xx.x%) xxx xx.x%-xx.x% |

N = number of patients, % = Observed percentage, E = number of events, CI = Confidence Interval.

Percentages are calculated relative to the total number of patients in the SAF population.

95% CI of the observed percentage calculated using the Clopper-Pearson methodology, or the Poisson distribution for frequencies below 10%. Each patient is counted at most once within each SOC and PT.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.14) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLE<br>(N=x | | | FL<br>(N=xx) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of E | vents | | | Num | mber of Eve | ents | | Number of Ev | rents |
| Preferred Term | n(%) | Total TR Rituximab TR Chemotherapy | | n(% | ) Tot | al TR | Rituximab | TR Chemotherapy | n(%) Total | TR Rituximak | TR Chemotherapy | |
| Number of patients with | | | | | | | | | | | | |
| Treatment-Emergent | xx (xx.x%) | XXX | xxx | xxx | xx ( | xx.x%) | XXX | xxX | XXX | xx (xx.x%) xx | x xxx | xxx |
| Adverse Events | | | | | | | | | | | | |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx ( | xx.x%) | XXX | XXX | xxx | xx (xx.x%) x | xx xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx ( | xx.x%) | XXX | XXX | XXX | xx (xx.x%) xx | XXX XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx ( | xx.x%) | XXX | XXX | XXX | xx (xx.x%) xx | XXX XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | XX ( | xx.x%) | XXX | XXX | XXX | xx (xx.x%) xx | XX XXX | XXX |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx ( | xx.x%) | xxx | xxX | xxx | xx (xx.x%) x | xx xxx | xxx |
| < PT > | xx (xx.x%) | XXX | xxx | xxx | xx ( | xx.x%) | XXX | xxX | XXX | xx (xx.x%) xx | xx xxx | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx ( | xx.x%) | XXX | XXX | XXX | xx (xx.x%) xx | xx xxx | XXX |
| < PT > | xx (xx.x%) | xxx | xxx | xxx | xx ( | xx.x%) | XXX | xxX | XXX | xx (xx.x%) xx | xx xxx | xxx |

Note(s): n=number of patients with an event. TR=treatment related.

MedDRA = Medical Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.15) SUMMARY OF SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | All Patients<br>(N=xxx) | | | | | DLBCL<br>(N=xx) | | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of H | Events | Number of Events | | | | | | | Nι | umber of Eve | ents |
| Preferred Term | n(% | Total | TR Rituxi | mab TR Chemotherapy | n (%) | Tot | tal TR | Rituximab 1 | R Chemotherapy | n | n(%) Tot | al TE | Rituximab | TR Chemotherap |
| Number of patients with serious | | | | | | | | | | | | | | |
| Treatment-Emergent | xx (xx.x | k) xxx | XXX | xxx | xx (xx | (.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX |
| Adverse Events | | | | | | | | | | | | | | |
| Primary SOC> | xx (xx.x | k) xxx | XXX | xxx | xx (xx | (.x%) | XXX | xxX | xxx | XX | (xx.x%) | XXX | xxx | xxx |
| < PT > | xx (xx.x | k) xxx | XXX | XXX | xx (xx | (.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX |
| < PT > | xx (xx.x | s) xxx | XXX | xxx | xx (xx | (.x%) | XXX | xxX | XXX | XX | (xx.x%) | XXX | XXX | XXX |
| < PT > | xx (xx.x | k) xxx | xxx | xxx | xx (xx | κ.x%) | XXX | XXX | xxx | XX | (xx.x%) | XXX | XXX | xxx |
| rimary SOC> | xx (xx.x | k) xxx | xxx | xxx | xx (xx | κ.χ%) | xxx | xxX | xxx | xx | (xx.x%) | xxx | xxx | xxx |
| < PT > | xx (xx.x | k) xxx | xxx | xxx | xx (xx | (.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | xxx | xxx |
| < PT > | xx (xx.x | b) xxx | XXX | xxx | xx (xx | (.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX |
| < PT > | xx (xx.x | k) xxx | xxx | xxx | xx (xx | (.x%) | XXX | xxX | XXX | xx | (xx.x%) | XXX | XXX | XXX |

Note(s): n=number of patients with an event. TR=treatment related.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.16) SUMMARY OF ADVERSE EVENTS OF SPECIAL INTEREST BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | All Patients<br>(N=xxx) | | | | | DLBCL<br>(N=xx) | | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Ev | ents | | Number of Events | | | | | | Num | ber of Eve | ents |
| Preferred Term | n(%) | Total | TR Rituxim | ab TR Chemotherapy | n(%) | Total | TR | Rituximab TR | Chemotherapy | n | n(%) Total | l TR | Rituximab | TR Chemotherapy |
| Number of patients with | | | | | | | | | | | | | | |
| Adverse Event of | xx (xx.x%) | XXX | XXX | XXX | xx (xx. | x%) x | XX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX |
| Special interest | | | | | | | | | | | | | | |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | x%) x | XX | xxX | xxx | XX | (xx.x%) | XXX | xxx | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx. | x%) x | XX | XXX | XXX | XX | (xx.x%) | KXX | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx. | x%) x | XX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx. | x%) x | XXX | XXX | XXX | XX | (xx.x%) | XXX | xxx | xxx |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | x%) x | XX | xxX | xxx | xx | (xx.x%) | xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | xxx | xxx | xx (xx. | x%) x | XX | xxX | xxx | | (xx.x%) | | xxx | XXX |
| < PT > | xx (xx.x%) | XXX | xxx | xxx | xx (xx. | x%) x | XX | xxX | xxx | XX | (xx.x%) | XXX | xxx | XXX |
| < PT > | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | x%) x | XX | xxX | XXX | XX | (xx.x%) | кхх | XXX | XXX |

Note(s): n=number of patients with an event. TR=treatment related.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.17) SUMMARY OF ADMINISTRATION ASSOCIATED REACTIONS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | DLBCL<br>(N=xx) | | | | | | FL<br>(N=xx) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Even | ts | | | N- | umber of Eve | ents | | | Jumber of Eve | nts |
| Preferred Term | n(%) | Total | TR Rituximab | TR Chemotherapy | n ( | %) T | otal T | R Rituximab | TR Chemotherapy | n | (%) Total T | 'R Rituximab | TR Chemotherapy |
| Number of patients with | | | | | | | | | | | | | |
| Administration Associated Reactions | xx (xx.x%) | XXX | xxx | XXX | XX | (xx.x% | ) xxx | xxX | xxx | XX | (xx.x%) xxx | xxx | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | XX | (xx.x% | ) xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | XX | (xx.x% | ) xxx | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | XX | (xx.x% | ) xxx | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | xxx | xxx | XX | (xx.x% | ) xxx | xxX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx | (xx.x% | ) xxx | xxX | xxx | XX | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | xxx | XXX | XX | (xx.x% | ) xxx | xxX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | XXX | xxx | XXX | XX | (xx.x% | ) xxx | xxX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx | (xx.x% | ) xxx | xxX | XXX | XX | (xx,x%) xxx | xxx | XXX |

Note(s): n=number of patients with an event. TR=treatment related.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TABLE 14.2.18) SUMMARY OF INFUSION/INJECTION-RELATED REACTIONS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | All Patients<br>(N=xxx) | | | | | DLE<br>(N=x | | | FL<br>(N=xx) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Eve | ents | Number of Events | | | | | | Nur | mber of Eve | nts |
| Preferred Term | n(%) | Total | TR Rituxima | ab TR Chemotherapy | n (%) | Tot | al TR | Rituximab T | TR Chemotherapy | n | (%) Total TR | Rituximab | TR Chemotherapy |
| Number of patients with | | | | | | | | | | | | | |
| Infusion/Injection-Related Reaction | xx (xx.x%) | XXX | xxx | XXX | xx ( | xx.x%) | XXX | XXX | xxx | XX | (xx.x%) xxx | xxx | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx | x.x%) | xxx | xxX | xxx | XX | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | xxx | XXX | xx (xx | x.x%) | XXX | XXX | xxx | XX | (xx.x%) xxx | xxx | XXX |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx | x.x%) | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | xxx | XXX | xx (xx | x.x%) | XXX | xxX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx (xx | x.x%) | XXX | xxX | XXX | XX | (xx.x%) xxx | XXX | XXX |

Note(s): n=number of patients with an event. TR=treatment related.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.
TABLE 14.2.19) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ AES BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLE<br>(N=x | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Ever | nts | | | Num | ber of Ever | nts | | | Number of Eve | nts |
| Preferred Term | n(%) | Total | TR Rituximak | TR Chemotherapy | n (% | ) To | tal TR | Rituximab T | 'R Chemotherapy | r | n(%) Total | TR Rituximab | TR Chemotherapy |
| Number of patients with grade | | | | | | | | | | | | | |
| >=3+ Treatment Emergent | | | | | | | | | | | | | |
| Adverse Event | xx (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | xxX | XXX | XX | (xx.x%) xx | xxx xxx | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx | (xx.x%) | xxx | xxX | xxx | xx | (xx.x%) xx | xx xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) xx | xxx xxx | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) xx | xxx xxx | XXX |
| < PT > | xx (xx.x%) | XXX | xxx | xxx | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) xx | xxx xxx | xxx |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx | (xx.x%) | xxx | xxX | xxx | xx | (xx.x%) xx | x xxx | xxx |
| < PT > | xx (xx.x%) | XXX | xxx | XXX | | (xx.x%) | XXX | xxX | XXX | | (xx.x%) xx | | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | xxX | XXX | хx | (xx.x%) xx | xxx xxx | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | | (xx.x%) | XXX | xxX | XXX | ХX | (xx.x%) xx | xxx xxx | XXX |

MedDRA = Medical Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.20) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ SAES BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLE<br>(N=) | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Ever | nts | | | Nun | mber of Ever | nts | | Nu | mber of Eve | nts |
| Preferred Term | n(%) | Total | TR Rituximak | TR Chemotherapy | n (% | t) To | tal TR | Rituximab 1 | R Chemotherapy | n | n(%) Total TR | Rituximab | TR Chemotherapy |
| Number of patients with grade | | | | | | | | | | | | | |
| >=3+ Treatment-Emergent Serious<br>Adverse Events | xx (xx.x%) | xxx | xxx | xxx | XX | (xx.x%) | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| Drimary COCX | xx (xx.x%) | | | | | (xx.x%) | xxx | xxX | | | (xx.x%) xxx | | |
| Primary SOC> < PT > | xx (xx.x%) | XXX | XXX | XXX | | (xx.x%) | XXX | XXX | XXX | | (xx.x%) xxx<br>(xx.x%) xxx | XXX | XXX<br>XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | | (xx.x%) | XXX | XXX | XXX | | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | xxx | xxx | xxx | | (xx.x%) | | xxX | XXX | | (xx.x%) xxx | xxx | XXX |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx | (xx.x%) | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | xxx | xxx | | (xx.x%) | XXX | xxX | xxx | | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | xxX | xxx | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | XX | (xx.x%) | XXX | xxX | XXX | XX | (xx.x%) xxx | XXX | XXX |

MedDRA = Medical Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.21) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ AESI BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DL: | BCL<br>xx) | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Ev | ents | | | Nu | mber of Even | its | | | Nui | mber of Ever | nts |
| Preferred Term | n(%) | Total | TR Rituxim | ab TR Chemotherapy | n (% | t) To | tal TR | Rituximab T | 'R Chemotherapy | r | n(%) Tota | al TR | Rituximab 1 | R Chemotherapy |
| Number of patients with grade | | | | | | | | | | | | | | |
| >=3+ Treatment-Emergent AESI | xx (xx.x%) | xxx | xxx | xxx | XX | (xx.x%) | xxx | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx | (xx.x%) | xxx | xxX | xxx | xx | (xx.x%) | xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | xxX | XXX | XX | (xx.x%) | XXX | XXX | xxx |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx | (xx.x%) | xxx | xxX | xxx | XX | (xx.x%) | xxx | xxx | xxx |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX |
| < PT > | xx (xx,x%) | XXX | XXX | xxx | XX | (xx.x%) | XXX | xxX | XXX | XX | (xx.x%) | XXX | XXX | XXX |

Note(s): n=number of patients with an event. TR=treatment related.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.22) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ AARS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLI<br>(N=: | BCL<br>xx) | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Eve | ents | | | Nui | mber of Eve | nts | | Nı | umber of Eve | ents |
| Preferred Term | n(%) | Total | TR Rituxima | ab TR Chemotherapy | n (%) | To | tal TR | Rituximab | TR Chemotherapy | n | (%) Total TI | R Rituximab | TR Chemotherapy |
| Number of patients with grade | | | | | | | | | | | | | |
| >=3+ Treatment-Emergent AARS | xx (xx.x%) | XXX | XXX | xxx | xx (x | x.x%) | XXX | XXX | xxx | XX | (xx.x%) xxx | XXX | xxx |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (x | x.x%) | xxx | xxX | xxx | XX | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (x | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (x | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | xxx | XXX | xx (x | x.x%) | XXX | xxX | xxx | XX | (xx.x%) xxx | XXX | XXX |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (x | x.x%) | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | xxx | xxx | xx (x | x.x%) | XXX | xxX | XXX | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (x | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx (x | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | xxx | XXX |

Note(s): n=number of patients with an event. TR=treatment related.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.23) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH GRADE >=3+ IIRRS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLB<br>(N=x | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Eve | nts | | | Num | ber of Even | ts | | Nur | mber of Eve | nts |
| Preferred Term | n(%) | Total | TR Rituxima | b TR Chemotherapy | n (%) | Tot | al TR | Rituximab T | R Chemotherapy | n | (%) Total TR | Rituximab | TR Chemotherapy |
| Number of patients with grade >=3+ Treatment-Emergent IIRRS | xx (xx.x%) | xxx | xxx | xxx | xx ( | (xx.x%) | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (x | (x.x% | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (x | (x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (x | (x.x% | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (x | (x.x%) | XXX | XXX | xxx | XX | (xx.x%) xxx | XXX | XXX |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (x | (x.x%) | xxx | xxX | xxx | XX | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (x | (x.x% | XXX | xxX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (x | (x.x% | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx (x | (x.x% | XXX | xxX | XXX | XX | (xx.x%) xxx | XXX | XXX |

MedDRA = MedIcal Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.24) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITHIN THE MEDDRA SMQ `ANAPHYLACTIC REACTIONS' (WIDE) BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | (N= | BCL<br>xx) | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Eve | nts | | | Nu | mber of Even | ts | | N | umber of Eve | nts |
| Preferred Term | n(%) | Total | TR Rituximal | o TR Chemotherapy | n (% | ) To | otal TR | Rituximab T | R Chemotherapy | r | n(%) Total T | R Rituximab | TR Chemotherapy |
| Number of patients with SMQ | | | | | | | | | | | | | |
| Anaphylactic reactions | xx (xx.x%) | XXX | XXX | XXX | xx ( | XX.X%) | ) xxx | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx ( | xx.x% | ) xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx ( | xx.x% | xxx | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx ( | xx.x% | ) xxx | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx ( | xx.x%) | ) xxx | xxX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx ( | xx.x% | ) xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | xxx | XXX | | xx.x% | | xxX | xxx | XX | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx ( | xx.x% | xxx | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx ( | xx.x% | xxx | xxX | XXX | XX | (xx.x%) xxx | XXX | XXX |

Note(s): n=number of patients with an event. TR=treatment related.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.25) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO RITUXIMAB DRUG INTERRUPTED/DRUG DELAYED BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLB<br>(N=x | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Eve | nts | | | Num | ber of Eve | nts | | Nı | umber of Ever | nts |
| Preferred Term | n(%) | Total | TR Rituxima | b TR Chemotherapy | n(%) | Tota | 1 TR | Rituximab | TR Chemotherapy | n | (%) Total TI | R Rituximab 1 | TR Chemotherap |
| Number of patients with<br>Treatment-Emergent Adverse Event<br>Leading to Rituximab<br>Drug interrupted/delayed | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | x%) : | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | x%) : | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | x%) : | XXX | xxX | xxx | XX | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx (xx. | x%) : | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx. | x%) : | XXX | XXX | xxx | XX | (xx.x%) xxx | xxx | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | x%) : | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | x%) : | XXX | XXX | xxx | XX | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx (xx. | x%) : | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx. | x%) : | XXX | xxX | xxx | xx | (xx.x%) xxx | XXX | XXX |

MedDRA = Medical Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.26) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO RITUXIMAB DOSE DISCONTINUATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLE<br>(N=> | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Even | ts | | | Nun | mber of Even | ts | | Nu | mber of Eve | nts |
| Preferred Term | n(%) | Total | TR Rituximab | TR Chemotherapy | n(%) | Tota | al TR | Rituximab T | R Chemotherapy | n | (%) Total TR | Rituximab | TR Chemotherapy |
| Number of patients with<br>Treatment-Emergent Adverse Event<br>Leading to Rituximab | | | | | | | | | | | | | |
| Dose discontinuation | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | . x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | xxx | xxx |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | . x%) | XXX | xxX | xxx | XX | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx. | .x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx. | .x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx. | . x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | .x%) | xxx | xxX | XXX | XX | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx. | .x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx. | .x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx (xx. | x%) | XXX | xxX | XXX | XX | (xx.x%) xxx | XXX | XXX |

MedDRA = Medical Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.27) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO CHEMOTHERAPY DOSE MODIFICATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLI<br>(N=2 | BCL<br>kx) | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Even | ts | | | Nur | mber of Event | S | | Nı | umber of Eve | nts |
| Preferred Term | n (%) | Total | TR Rituximab | TR Chemotherapy | n (%) | То | tal TR | Rituximab TR | Chemotherapy | n | n(%) Total Ti | R Rituximab | TR Chemotherapy |
| Number of patients with<br>Treatment-Emergent Adverse Event<br>Leading to Chemotherapy | | | | | | | | | | | | | |
| Dose modification | xx (xx.x%) | XXX | xxx | xxx | xx (: | (x.x%) | xxx | XXX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (: | xx.x%) | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx ( | (x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx ( | (x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx ( | (x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (: | (x.x%) | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx ( | (x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx ( | (x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | xxx | xxx | xx ( | (x.x%) | XXX | xxX | XXX | XX | (xx.x%) xxx | XXX | xxx |

MedDRA = Medical Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.28) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO CHEMOTHERAPY DOSE DISCONTINUATION BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DL<br>(N= | BCL<br>xx) | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Ever | nts | | | Nu | mber of Eve | nts | | | Numb | er of Ever | nts |
| Preferred Term | n(%) | Total | TR Rituximab | TR Chemotherapy | n (9 | ð) To | tal TR | Rituximab | TR Chemotherapy | n | n(%) Total | L TR R | ituximab 1 | R Chemotherapy |
| Number of patients with Treatment-Emergent Adverse Event Leading to Chemotherapy Dose discontinuation | xx (xx.x%) | xxx | xxx | xxx | xx | (xx.x%) | xxx | xxX | XXX | xx | (xx.x%) > | «×× | xxx | xxx |
| | (, | | | | | (, | | | | | ( | | | |
| Primary SOC> | xx (xx.x%) | XXX | xxx | XXX | XX | (xx.x%) | XXX | xxX | xxx | XX | (xx.x%) x | XXX | xxx | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) x | КХХ | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) x | XXX | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) > | XXX | XXX | XXX |
| Primary SOC> | xx (xx.x%) | xxx | XXX | xxx | xx | (xx.x%) | xxx | xxX | xxx | XX | (xx.x%) x | кхх | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) > | XXX | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX | | (xx.x%) > | | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) | XXX | XXX | XXX | XX | (xx.x%) x | XXX | XXX | XXX |

MedDRA = Medical Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.29) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS LEADING TO DEATH BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLE<br>(N=x | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Eve | nts | | | Num | ber of Ever | nts | | Nun | ber of Eve | nts |
| Preferred Term | n(%) | Total | TR Rituxima | b TR Chemotherapy | n (%) | Tot | al TR | Rituximab 1 | 'R Chemotherapy | n | n(%) Total TR | Rituximab | TR Chemotherapy |
| Number of patients with | | | | | | | | | | | | | |
| reatment-Emergent Adverse Event | | | | | | | | | | | | | |
| eading to death | xx (xx.x%) | XXX | XXX | XXX | xx (x | (x.x% | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (x | x.x%) | xxx | xxX | xxx | XX | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | xxx | xxx | xxx | xx (x | x.x%) | XXX | xxX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | xxx | xxx | xxx | xx (x | x.x%) | XXX | xxX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (x | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (x | x.x%) | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | XXX | xxx | xxx | xx (x | x.x%) | XXX | xxX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | XXX | xxx | XXX | xx (x | x.x%) | XXX | xxX | xxx | XX | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx (x | x.x%) | XXX | xxX | XXX | XX | (xx.x%) xxx | xxx | XXX |

MedDRA = Medical Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.30) SUMMARY OF CUTANEOUS AND SOFT TISSUE AARS (LOCALIZED) BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLB<br>(N=x | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Eve | nts | | | Num | ber of Ever | nts | | Nui | mber of Eve | nts |
| Preferred Term | n(%) | Total | TR Rituxima | b TR Chemotherapy | n (%) | Tot | al TR | Rituximab ' | TR Chemotherapy | n | (%) Total TR | Rituximab | TR Chemotherapy |
| Number of patients with | | | | | | | | | | | | | |
| ARS localized | xx (xx.x%) | XXX | XXX | xxx | xx (x | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (x | x.x%) | xxx | xxX | xxx | XX | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (x | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (x | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (x | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | xxx | XXX |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (x | x.x%) | xxx | xxX | xxx | XX | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (x | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (x | x.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx (x | x.x%) | XXX | xxX | xxx | XX | (xx.x%) xxx | XXX | XXX |

Note(s): n=number of patients with an event. TR=treatment related.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TABLE 14.2.31) SUMMARY OF CUTANEOUS AND SOFT TISSUE AARS (NON-LOCALIZED) BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLB<br>(N=x | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Eve | ents | | | Num | ber of Eve | nts | | 1 | Number of Ev | ents |
| Preferred Term | n(%) | Total | TR Rituxima | ab TR Chemotherapy | n(%) | Tot | al TR | Rituximab | TR Chemotherapy | r | n(%) Total ' | R Rituximab | TR Chemotherap |
| Number of patients with<br>Cutaneous and soft tissue<br>AARS non-localized | xx (xx. | x%) x | xx xxx | xxx | xx | x (xx. | x%) x | xx xxX | xxx | | xx (xx.x%) | xxx xxx | xxx |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx | x.x%) | xxx | xxX | xxx | xx | (xx.x%) xx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx | (.x%) | XXX | XXX | XXX | XX | (xx.x%) xx | xxx | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx | (.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx | (.x%) | XXX | XXX | xxx | XX | (xx.x%) xx | xxx | xxx |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx | x.x%) | xxx | xxX | xxx | XX | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | xxx | xxx | xx (xx | | XXX | xxX | xxx | XX | (xx.x%) xx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx | (.x%) | XXX | XXX | XXX | XX | (xx.x%) xx | xxx | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx (xx | ( %x · | XXX | xxX | XXX | xx | (xx.x%) xx | xxx | XXX |

MedDRA = Medical Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TABLE 14.2.32) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS WITH AN INCIDENCE OF >=5% BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DL<br>(N= | BCL<br>xx) | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Eve | nts | | | Nu | mber of Event | .s | | Nu | mber of Eve | nts |
| Preferred Term | n(%) | Total | TR Rituximal | b TR Chemotherapy | n(% | ) To | otal TR | Rituximab TF | Chemotherapy | n | (%) Total TR | Rituximab | TR Chemotherap |
| Number of patients with Treatment-Em | nergent | | | | | | | | | | | | |
| Adverse Events with Incidence >=5% | xx (xx.x%) | XXX | XXX | xxx | xx ( | xx.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx ( | xx.x%) | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx ( | xx.x%) | XXX | XXX | XXX | ХX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx ( | xx.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx ( | xx.x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx ( | xx.x%) | xxx | xxX | xxx | хх | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | xxx | xxx | xxx | xx ( | xx.x%) | XXX | xxX | XXX | хх | (xx.x%) xxx | xxx | XXX |
| < PT > | xx (xx.x%) | XXX | xxx | XXX | | xx.x%) | | xxX | xxx | хх | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx ( | xx.x%) | xxx | xxX | XXX | XX | (xx,x%) xxx | XXX | XXX |

Note(s): n=number of patients with an event. TR=treatment related.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.33) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM AND MAXIMUM SEVERITY (SAFETY POPULATION)

| | | | | All Patients (N=xxx) | | | | DLB( | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Maximum | System Organ Class | | | Number of Eve | <br>ents | | | Numbe | er of Ever | ts | Numbe | er of Eve | <br>nts |
| Severity | Preferred Term | n (%) | Total | TR Rituximak | o TR Chemotherapy | n(%) | Total | TR Rit | tuximab TF | Chemotherapy | n(%) Total TR Rit | uximab T | R Chemotherapy |
| rade x | Number of patients with<br>Treatment-Emergent Adverse | | | | | | | | | | | | |
| | Event (Max Grade) | xx (xx.x% | ) xxx | XXX | xxx | xx | (xx.x%) | xxx | XXX | XXX | xx (xx.x%) xxx | XXX | XXX |
| | Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx ( | (xx.x%) | xxx | xxX | xxx | xx (xx.x%) xxx | xxx | xxx |
| | < PT > | xx (xx.x%) | xxx | XXX | xxx | xx ( | (xx.x%) | XXX | XXX | XXX | xx (xx.x%) xxx | xxx | XXX |
| | < PT > | xx (xx.x%) | xxx | XXX | xxx | xx ( | (xx.x%) | XXX | XXX | XXX | xx (xx.x%) xxx | XXX | XXX |
| | < PT > | xx (xx.x%) | XXX | xxx | XXX | XX ( | (xx.x%) | XXX | xxx | XXX | xx (xx.x%) xxx | xxx | XXX |
| | Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx ( | (xx.x%) | xxx | xxX | xxx | xx (xx.x%) xxx | xxx | xxx |
| | < PT > | xx (xx.x%) | xxx | xxx | xxx | XX | (xx.x%) | XXX | XXX | XXX | xx (xx.x%) xxx | xxx | XXX |
| | < PT > | xx (xx.x%) | xxx | XXX | xxx | XX ( | (xx.x%) | XXX | XXX | XXX | xx (xx.x%) xxx | xxx | XXX |
| | < PT > | xx (xx.x%) | XXX | XXX | xxx | xx ( | (xx.x%) | XXX | XXX | xxx | xx (xx.x%) xxx | XXX | xxx |
| rade x | Number of patients with<br>Treatment-Emergent Adverse | | | | | | | | | | | | |
| | Event (Max Grade) | xx (xx.x% | ) xxx | xxx | XXX | XX | (xx.x%) | XXX | XXX | XXX | xx (xx.x%) xxx | xxx | XXX |
| | Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx | (xx.x%) | xxx | xxX | xxx | xx (xx.x%) xxx | xxx | xxx |
| | < PT > | xx (xx.x%) | XXX | XXX | XXX | XX ( | (xx.x%) | XXX | xxX | XXX | xx (xx.x%) xxx | XXX | XXX |
| | < PT > | xx (xx.x%) | XXX | XXX | XXX | XX ( | (xx.x%) | XXX | xxX | XXX | xx (xx.x%) xxx | xxx | XXX |
| | < PT > | xx (xx.x%) | XXX | XXX | XXX | xx ( | (xx.x%) | XXX | XXX | XXX | xx (xx.x%) xxx | XXX | xxx |
| | Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | | (xx.x%) | xxx | xxX | xxx | xx (xx.x%) xxx | xxx | xxx |
| | < PT > | xx (xx.x%) | XXX | XXX | XXX | | (xx.x%) | XXX | xxX | XXX | xx (xx.x%) xxx | XXX | XXX |
| | < PT > | xx (xx.x%) | XXX | XXX | XXX | | (xx.x%) | XXX | xxX | XXX | xx (xx.x%) xxx | XXX | XXX |
| | < PT > | xx (xx.x%) | XXX | XXX | XXX | XX ( | (xx.x%) | XXX | XXX | XXX | xx (xx.x%) xxx | XXX | XXX |

Note(s): n=number of patients with an event. TR=treatment related.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.34) SUMMARY OF TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM AND STRONGEST RELATIONSHIP (SAFETY POPULATION)

| | | | | Patients<br>xxx) | | | | DLBC | | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Strong | gest System Organ Class | | | Number of | Events | | | Nu | umber of E | lvents | | | Number of Ev | ents |
| relat | ionship Preferred Term | n(%) | Total | TR Ritux | ximab TR Chemotherapy | n (%) | Tot | tal TF | R Rituxima | ab TR Chemother | rapy | n(%) Total | TR Rituximab | TR Chemotherap |
| Yes | Number of patients with | | | | | | | | | | | | | |
| | Treatment-Emergent Advers | е | | | | | | | | | | | | |
| | Event (Max Grade) | xx (xx.x%) | xxx | XXX | XXX | xx (xx | x%) | xxx | XXX | XXX | XX | x (xx.x%) xxx | XXX | XXX |
| | Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx.: | (%) x | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| | < PT > | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | (%) > | xxx | xxX | XXX | xx | (xx.x%) xxx | xxx | XXX |
| | < PT > | xx (xx.x%) | XXX | xxx | xxx | xx (xx. | | XXX | xxX | XXX | XX | (xx.x%) xxx | xxx | xxx |
| | < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx. | (용) > | XXX | XXX | xxx | XX | (xx.x%) xxx | xxx | xxx |
| | Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | (왕) > | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| | < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx. | (용) > | XXX | xxX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| | < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx. | (용) > | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| | < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx. | (응) > | XXX | XXX | xxx | XX | (xx.x%) xxx | XXX | XXX |
| No | Number of patients with Treatment-Emergent Advers | e | | | | | | | | | | | | |
| | Event (Max Grade) | xx (xx.x%) | xxx | XXX | XXX | xx (xx | x%) | xxx | XXX | XXX | XX | x (xx.x%) xxx | XXX | XXX |
| | Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | ·8) s | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| | < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx. | , | XXX | xxX | XXX | | (xx.x%) xxx | XXX | XXX |
| | < PT > | xx (xx.x%) | xxx | xxx | xxx | xx (xx.: | | xxx | xxX | XXX | | (xx.x%) xxx | xxx | XXX |
| | < PT > | xx (xx.x%) | xxx | xxx | XXX | xx (xx. | (%) > | XXX | XXX | xxx | | (xx.x%) xxx | xxx | XXX |
| | Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx. | (용) > | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| | < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx. | (응) > | XXX | xxX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| | < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx. | (용) > | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| | < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx. | (%) > | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |

Note(s): n=number of patients with an event. TR=treatment related.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.35) SUMMARY OF NON-SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS WITH AN INCIDENCE OF >=5% BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAFETY POPULATION)

| | | | ll Patients<br>N=xxx) | | | | DLE<br>(N=2 | BCL<br>xx) | | | | FL<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | Number of Ever | nts | | | Nur | mber of Eve | ents | | Nu | umber of Eve | ents |
| Preferred Term | n(%) | Total | TR Rituximak | TR Chemotherapy | n(%) | Tot | al TR | Rituximab | TR Chemotherapy | n | n(%) Total TF | R Rituximab | TR Chemotherapy |
| Number of patients with Treatment-Em | ergent | | | | | | | | | | | | |
| Adverse Events with Incidence >=5% | xx (xx.x%) | XXX | xxx | xxx | xx (xx | .x%) | XXX | XXX | xxx | XX | (xx.x%) xxx | xxx | XXX |
| Primary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx | .x%) | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx | .x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | XXX | xxx | xx (xx | .x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | XXX | xxx | xxx | xx (xx | .x%) | XXX | XXX | xxx | XX | (xx.x%) xxx | xxx | xxx |
| rimary SOC> | xx (xx.x%) | xxx | xxx | xxx | xx (xx | .x%) | xxx | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | xxx | XXX | xx (xx | .x%) | XXX | xxX | xxx | xx | (xx.x%) xxx | xxx | xxx |
| < PT > | xx (xx.x%) | XXX | XXX | XXX | xx (xx | .x%) | XXX | XXX | XXX | XX | (xx.x%) xxx | XXX | XXX |
| < PT > | xx (xx.x%) | xxx | XXX | xxx | xx (xx | .x%) | XXX | xxX | XXX | XX | (xx.x%) xxx | XXX | XXX |

MedDRA = MedIcal Dictionary for Regulatory Activities. SOC and PT are from the MedDRA dictionary, version 24.1.

A patient experiencing multiple occurrences of an adverse event was counted, at most, once per System Organ Class and Preferred Term.

TEAEs are AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose.

TABLE 14.2.36) SUMMARY OF PATIENTS DEAD OVER THE STUDY (SAFETY POPULATION)

| | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Total number of patients dead | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Primary cause of death | | | | |
| Progression of disease | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Adverse event | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Unknown | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| If cause of death is AE, was the underlying cancer a contributing factor#? | | | | |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Is there reasonable suspected casual relationship to study medication? | | | | |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Was an autopsy performed? | | | | |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of patients in the SAF population.

# Percentages are calculated relative to the total number of patients with primary cause of death = "AE".

TABLE 14.3.1) SUMMARY OF HEMATOLOGY PARAMETERS OVER THE STUDY (SAFETY POPULATION)

| | | | Patients | | DLBCL | | _ FL |
|---|---|---|---|---|---|---|---|
| Hemoglobin (g/L) | | (1 | N=xxx) | | (N=xx) | | (N=xx) |
| | Statistic | Value | Change from<br>Screening | Value | Change from<br>Screening | Value | Change from<br>Screening |
| Screening Visit | n | xxx | | xx | | xx | |
| | Mean (SD) | xxx.x (xx.xx) | | xxx.x (xx.xx) | | xxx.x (xx.xx) | |
| | Median | xxx.x | | XXX.X | | xxx.x | |
| | Min/Max | xx.x/xxx.x | | xx.x/xxx.x | | xx.x/xxx.x | |
| Cycle 1 Induction | n | xx | xx | | | XX | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (x.xx) | | | xxx.x (xx.xx) | x.x (x.xx) |
| | Median | xxx.x | X.X | | | xxx.x | X.X |
| | Min/Max | xxx.x/xxx.x | xx.x/x.x | | | xxx.x/xxx.x | xx.x/x.x |
| Cycle 2 Induction | n | XX | XX | | | XX | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (xx.xx) | | | xxx.x (xx.xx) | x.x (xx.xx) |
| | Median | xxx.x | x.x | | | XXX.X | X.X |
| | Min/Max | xx.x/xxx.x | xx.x/xx.x | | | xx.x/xxx.x | xx.x/xx.x |
| Cycle x Induction | n | xx | XX | | | xx | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (xx.xx) | | | xxx.x (xx.xx) | x.x (xx.xx) |
| | Median | xxx.x | X.X | | | xxx.x | X.X |
| | Min/Max | xx.x/xxx.x | xx.x/xx.x | | | xx.x/xxx.x | xx.x/xx.x |

Change from Screening values includes only those patients with both a screening value and a value for summarized time period. n represents number of patients contributing to summary statistics.

Source: XXXX.SAS, Run on DDMMMYYYY

## Programming note:

This table to be repeated for all hematology parameters for each visit of induction and maintenance phases. Data must be presented according to the International System of Units (SI).

TABLE 14.3.2) SUMMARY OF BLOOD CHEMISTRY PARAMETERS OVER THE STUDY (SAFETY POPULATION)

| | | | Patients | | DLBCL | | FL |
|---|---|---|---|---|---|---|---|
| Sodium (mmol/L) | | (N: | =xxx) | ( | (N=xx) | ( | N=xx) |
| | Statistic | Value | Change from<br>Screening | Value | Change from<br>Screening | Value | Change from<br>Screening |
| Screening Visit | n | xxx | | xx | | xx | |
| | Mean (SD) | xxx.x (xx.xx) | | xxx.x (xx.xx) | | xxx.x (xx.xx) | |
| | Median | xxx.x | | xxx.x | | xxx.x | |
| | Min/Max | xx.x/xxx.x | | xx.x/xxx.x | | xx.x/xxx.x | |
| Cycle 1 Induction | n | XX | xx | | | xx | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (x.xx) | | | xxx.x (xx.xx) | x.x (x.xx) |
| | Median | xxx.x | X.X | | | xxx.x | х.х |
| | Min/Max | xxx.x/xxx.x | xx.x/x.x | | | xxx.x/xxx.x | xx.x/x.x |
| Cycle 2 Induction | n | xx | xx | | | XX | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (xx.xx) | | | xxx.x (xx.xx) | x.x (xx.xx) |
| | Median | xxx.x | x.x | | | xxx.x | х.х |
| | Min/Max | xx.x/xxx.x | xx.x/xx.x | | | xx.x/xxx.x | xx.x/xx.x |
| Cycle x Induction | n | xx | XX | | | xx | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (xx.xx) | | | xxx.x (xx.xx) | x.x (xx.xx) |
| | Median | xxx.x | X.X | | | xxx.x | X.X |
| | Min/Max | xx.x/xxx.x | xx.x/xx.x | | | xx.x/xxx.x | xx.x/xx.x |

Change from Screening values includes only those patients with both a screening value and a value for summarized time period. n represents number of patients contributing to summary statistics.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table to be repeated for all blood chemistry parameters for each visit of induction and maintenance phases. Data must be presented according to the International System of Units (SI).

TABLE 14.3.3) SUMMARY OF COAGULATION TESTS OVER THE STUDY (SAFETY POPULATION)

| D. ( ) | | | Patients | | DLBCL | | FL |
|---|---|---|---|---|---|---|---|
| PT (sec) | | (N | =xxx) | | (N=xx)<br>Change from | | (N=xx) |
| | Statistic | Value | Change from<br>Screening | Value | Screening | Value | Change from<br>Screening |
| Screening Visit | n | xxx | | xx | | xx | |
| - | Mean (SD) | xxx.x (xx.xx) | | xxx.x (xx.xx) | | xxx.x (xx.xx) | |
| | Median | xxx.x | | xxx.x | | xxx.x | |
| | Min/Max | xx.x/xxx.x | | xx.x/xxx.x | | xx.x/xxx.x | |
| Cycle 1 Induction | n | xx | xx | | | xx | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (x.xx) | | | xxx.x (xx.xx) | x.x (x.xx) |
| | Median | xxx.x | X . X | | | xxx.x | X.X |
| | Min/Max | xxx.x/xxx.x | xx.x/x.x | | | xxx.x/xxx.x | xx.x/x.x |
| Cycle 2 Induction | n | xx | xx | | | xx | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (xx.xx) | | | xxx.x (xx.xx) | x.x (xx.xx) |
| | Median | xxx.x | X.X | | | xxx.x | X.X |
| | Min/Max | xx.x/xxx.x | xx.x/xx.x | | | xx.x/xxx.x | xx.x/xx.x |
| ••• | | | | | | | |
| Cycle x Induction | n | xx | xx | | | xx | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (xx.xx) | | | xxx.x (xx.xx) | x.x (xx.xx) |
| | Median | xxx.x | X.X | | | xxx.x | X.X |
| | Min/Max | xx.x/xxx.x | xx.x/xx.x | | | xx.x/xxx.x | xx.x/xx.x |

Change from Screening values includes only those patients with both a screening value and a value for summarized time period. n represents number of patients contributing to summary statistics.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table to be repeated for all blood chemistry parameters for each visit of induction and maintenance phases. Data must be presented according to the International System of Units (SI).

TABLE 14.3.4) SHIFT TABLE OF HEMATOLOGY PARAMETERS ACCORDING TO NCI CTCAE WORST GRADE RECORDED DURING THE TREATMENT PERIOD (SAFETY POPULATION)

| | | | | NCI CTC | AE Worst Grade | During Treatment | t Period | |
|---|---|---|---|---|---|---|---|---|
| | | Statistic | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Not Done | All |
| DLBCL | Screening | | | | | | | |
| | Grade 1 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Grade 2 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Grade 3 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Grade 4 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx,x) | xxx (xx.x) |
| | Not Done | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | All | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| L | Screening | | | | | | | |
| | Grade 1 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Grade 2 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Grade 3 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Grade 4 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Not Done | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | All | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| All Patients | Screening | | | | | | | |
| | Grade 1 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Grade 2 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Grade 3 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Grade 4 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Not Done | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | All | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Percentage are calculated relative to the total number of patients in the SAF population (row percentages).

Source: XXXX.SAS, Run on DDMMMYYYY

## Programming note:

This table to be repeated for all hematology parameters.

TABLE 14.3.5) SHIFT TABLE OF BLOOD CHEMISTRY PARAMETERS ACCORDING TO NCI CTCAE WORST GRADE RECORDED DURING THE TREATMENT PERIOD (SAFETY POPULATION)

| | | | NCI CTC | AE Worst Grade | During Treatment | t Period | |
|---|---|---|---|---|---|---|---|
| | Statistic | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Not Done | All |
| Screening | | | | | | | |
| _ | n (%) | vvv (vv v) | vvv (vv v) | vvv (vv v) | vvv (vv v) | vvv (vv v) | xxx (xx.x) |
| | | , , | , , | , , | , , | , , | xxx (xx.x) |
| | | , , | , , | , , | , , | | xxx (xx.x) |
| | | , , | , , | | , , | | xxx (xx.x) |
| | | , , | , , | , , | , , | | xxx (xx.x) |
| | | , , | , , | , , | , , | | xxx (xx.x) |
| VII | 11 (0) | AAA (AA.A) | AAA (AA.A) | AAA (AA.A) | AAA (AA.A) | AAA (AA.A) | AAA (AA.A) |
| Screening | | | | | | | |
| Grade 1 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Grade 2 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Grade 3 | | xxx (xx,x) | xxx (xx.x) | xxx (xx.x) | | xxx (xx.x) | xxx (xx.x) |
| Grade 4 | | xxx (xx,x) | xxx (xx.x) | xxx (xx.x) | | xxx (xx.x) | xxx (xx.x) |
| Not Done | | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | | xxx (xx.x) | xxx (xx.x) |
| | | , , | , , | , , | , , | , , | xxx (xx.x) |
| | , | , , | , , | , , | , , | , , | , , |
| Screening | | | | | | | |
| Grade 1 | n (%) | xxx (xx,x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Grade 2 | | xxx (xx,x) | xxx (xx.x) | | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Grade 3 | | | | | | | xxx (xx.x) |
| | | , , | , , | , , | , , | | xxx (xx.x) |
| | | , , | , , | , , | , , | , , | xxx (xx.x) |
| | | , , | , , | , , | , , | , , | xxx (xx.x) |
| | Grade 2<br>Grade 3<br>Grade 4<br>Not Done<br>All<br>Screening<br>Grade 1 | Screening Grade 1 | Screening Grade 1 | Statistic Grade 1 Grade 2 | Statistic Grade 1 Grade 2 Grade 3 | Screening Grade 1 | Screening Grade 1 |

Percentage are calculated relative to the total number of patients in the SAF population (row percentages).

Source: XXXX.SAS, Run on DDMMMYYYY

# Programming note:

This table to be repeated for all blood chemistry parameters.

TABLE 14.3.6) SHIFT TABLE OF COAGULATION TESTS ACCORDING TO NCI CTCAE WORST GRADE RECORDED DURING THE TREATMENT PERIOD (SAFETY POPULATION)

NCI CTCAE Worst Grade During Treatment Period Statistic Grade 1 Grade 2 Grade 3 Not Done All Grade 4 DLBCL Screening Grade 1 n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) Grade 2 n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) Grade 3 n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) Grade 4 n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx,x) Not Done n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) All n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) FLScreening Grade 1 n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) Grade 2 xxx (xx.x) n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) Grade 3 n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) Grade 4 n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) Not Done n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) All n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) All Patients Screening Grade 1 n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) Grade 2 n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) Grade 3 n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) Grade 4 n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) Not Done n (%) xxx (xx.x) xxx (xx.x) xxx (xx,x) xxx (xx.x) xxx (xx.x) xxx (xx.x) All n (%) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x) xxx (xx.x)

Notes:

Percentage are calculated relative to the total number of patients in the SAF population (row percentages).

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table to be repeated for all coagulation tests.

TABLE 14.3.7) SUMMARY OF VITAL SIGNS OVER THE STUDY (SAFETY POPULATION)

| | | | Patients | | DLBCL | | FL |
|---|---|---|---|---|---|---|---|
| Heart Rate (bpm) | | (N: | =xxx) | ( | (N=xx) | (1 | N=xx) |
| | Statistic | Value | Change from<br>Screening | Value | Change from<br>Screening | Value | Change from<br>Screening |
| | Statistic | value | | value | | value | Screening |
| Screening Visit | n | xxx | | xx | | xx | |
| | Mean (SD) | xxx.x (xx.xx) | | xxx.x (xx.xx) | | xxx.x (xx.xx) | |
| | Median | xxx.x | | xxx.x | | xxx.x | |
| | Min/Max | xx.x/xxx.x | | xx.x/xxx.x | | xx.x/xxx.x | |
| Cycle 1 Induction | n | xx | xx | | | XX | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (x.xx) | | | xxx.x (xx.xx) | x.x (x.xx) |
| | Median | xxx.x | X.X | | | xxx.x | X.X |
| | Min/Max | xxx.x/xxx.x | xx.x/x.x | | | xxx.x/xxx.x | xx.x/x.x |
| Cycle 2 Induction | n | XX | XX | | | xx | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (xx.xx) | | | xxx.x (xx.xx) | x.x (xx.xx) |
| | Median | xxx.x | X.X | | | xxx.x | X.X |
| | Min/Max | xx.x/xxx.x | xx.x/xx.x | | | xx.x/xxx.x | xx.x/xx.x |
| Cycle x Induction | n | xx | xx | | | xx | xx |
| | Mean (SD) | xxx.x (xx.xx) | x.x (xx.xx) | | | xxx.x (xx.xx) | x.x (xx.xx) |
| | Median | xxx.x | X.X | | | xxx.x | X.X |
| | Min/Max | xx.x/xxx.x | xx.x/xx.x | | | xx.x/xxx.x | xx.x/xx.x |

Change from Screening values includes only those patients with both a screening value and a value for summarized time period. n represents number of patients contributing to summary statistics.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table to be repeated for Systolic Blood Pressure, Diastolic Blood Pressure, Body Weight and Body Temperature.

TABLE 14.3.8) ECOG PERFORMANCE STATUS (SAFETY POPULATION)

| | | All Pa | tients<br>xxx) | DLB( | | FI<br>(N=x | |
|---|---|---|---|---|---|---|---|
| Cycle/Visit | ECOG-PS | n | % | n (iv- | %<br>% | n | % |
| Screening Visit | Grade 1 | xxx | х.х | xx | х.х | xx | х.х |
| - | Grade 2 | XXX | x.x | xx | x.x | XX | х.х |
| | Grade 3 | XXX | X.X | xx | x.x | XX | х.х |
| | Grade 4 | XXX | X.X | XX | x.x | XX | х.х |
| | Grade 5 | XXX | X.X | XX | x.x | XX | х.х |
| | Missing | XXX | х.х | XX | х.х | | х.х |
| Final Staging | Grade 1 | xxx | x.x | xx | х.х | xx | х.х |
| | Grade 2 | XXX | X.X | XX | x.x | XX | х.х |
| | Grade 3 | XXX | X.X | XX | x.x | XX | х.х |
| | Grade 4 | XXX | X.X | XX | x.x | XX | х.х |
| | Grade 5 | XXX | X.X | XX | X.X | XX | х.х |
| | Missing | XXX | x.x | XX | x.x | XX | х.х |

TABLE 14.4.1) TARGET LESION ASSESSMENT AT SCREENING (PART #1) (SAFETY POPULATION)

| | Statistic All Patients (N=xxx) | | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Were any target lesions identified? | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx,x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Location of lesion | | | | |
| Neck | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Chest | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Abdomen | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Pelvis | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| CT with contrast | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| CT result | | | | |
| Negative | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not assessed | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| CT without contrast | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| /es | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| CT w/o contrast result | | | | |
| Negative | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not assessed | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| MRI | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| /es | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| MRI result | | | | |
| Negative | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not assessed | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of patients in SAF population.

TABLE 14.4.2) TARGET LESION ASSESSMENT AT SCREENING (PART #2) (SAFETY POPULATION)

| | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Clinical assessment | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Clinical assessment result | | | | |
| Negative | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not assessed | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| FDG-PET | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| FDG-PET result | | | | |
| Negative | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not assessed | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other assessment | | | | |
| No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Other assessment | | | | |
| Negative | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Positive | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not assessed | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of patients in SAF population.

TABLE 14.4.3) POST-SCREENING TARGET LESION ASSESSMENT (PART #1) (SAFETY POPULATION)

| | | Statistic | All Patients (N=xxx) | DLBCL (N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|---|
| Study Visit <xxx></xxx> | Was a target lesions assessment done at this visit? | | | | |
| Study VISIT (XXX) | No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | 163 | 11 (0) | AAA (AA.A0) | AAA (AA.A0) | AAA (AA.A0) |
| | Were there any changes in the Target Lesions since | | | | |
| | the previous visit assessment? | | | | |
| | No | | | | |
| | Yes | | | | |
| | Not applicable | | | | |
| | Location of lesion | | | | |
| | Neck | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Chest | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Abdomen | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Pelvis | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Other | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | CT with contrast | | | | |
| | No | n (%) | / ) | xxx (xx.x%) | |
| | | . , | xxx (xx.x%) | , , | xxx (xx.x%) |
| | Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | CT result | | | | |
| | Increased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Decreased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No change | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | CT without contrast | | | | |
| | No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | CT w/o contrast result | | | | |
| | Increased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Decreased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No change | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | MRI | | | | |
| | No. | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | 163 | 11 (-0) | AAA (AA.A%) | AAA (AA.A°) | AAA (AA.X8) |
| | MRI result | (0) | | | , |
| | Increased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Decreased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No change | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of patients in SAF population performing the study visit.

# Programming note:

This table should be also presented for all post-screening visits.

Source: XXXX.SAS, Run on DDMMMYYYY

# Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

Mabrella ML28964 Daughter Protocol 136/Statistical Analysis Plan ML28964

TABLE 14.4.4) POST-SCREENING TARGET LESION ASSESSMENT (PART #2) (SAFETY POPULATION)

| | | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|---|
| Study Visit <xxx></xxx> | Clinical assessment | | | | |
| | No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Clinical assessment result | | | | |
| | Increased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Decreased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No change | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | FDG-PET | | | | |
| | No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | FDG-PET result | | | | |
| | Increased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Decreased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No change | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Other assessment | | | | |
| | No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Other assessment | | | | |
| | Increased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Decreased | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No change | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Change in lesion since first assessed /previous visit | | | | |
| | Enlarged | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | No change | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Reduced in size | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Not visible/too small | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Not applicable | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx,x%) |

Percentages are calculated relative to the total number of patients in SAF population performing the study visit.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table should be also presented for all post-screening visits.

TABLE 14.4.5) OVERALL LESION ASSESSMENT (SAFETY POPULATION)

| | | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|---|
| Study Visit <xxx></xxx> | Response of target lesions | | | | |
| | Complete response (CR) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Complete response unconfirmed (CRu) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Partial response (PR) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Stable disease (SD) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Progressive disease (PD) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Unable to assess (UA) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not applicable | Not applicable | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Are there any new lesions? | | | | |
| | No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Yes | Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x% |
| | Investigator's overall assessment of | | | | |
| | response at this visit | | | | |
| | Complete response (CR) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x% |
| | Complete response unconfirmed (CRu) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x% |
| | Partial response (PR) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x% |
| | Stable disease (SD) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x% |
| | Progressive disease (PD) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x% |
| | Unable to assess (UA) | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x% |
| | Not applicable | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x% |

Percentages are calculated relative to the total number of patients in SAF population performing the study visit.

Source: XXXX.SAS, Run on DDMMMYYYY

## Programming note:

This table should be also presented for all post-screening visits.

TABLE 14.5.1) OVERALL SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV (ITT POPULATION)

| | Statistic | All Patients<br>(N=xxx) | DLBCL<br>(N=xxx) | FL (N=xxx) |
|---|---|---|---|---|
| Time to event (months) | 25th (95% CI)<br>Median (95% CI)<br>75th (95% CI) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) |
| Number of patients Events | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Censored | n (%) | xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |

Percentages are calculated on the number of patients in the ITT population.

Overall survival(months) was estimated using Kaplan-Meier method.

Patients who are not reported as having died at the time of analysis will be censored at the last contact date.

Patients who do not have post-baseline information will be censored at the date of initiation of study treatment. Patients enrolled but not treated will be assigned time = 0.

•

### Programming note:

This table should be also presented from the first dose of Rituximab SC. This table should be also presented stratified by:

a) Gender (Female, Male)

- b) FLIPI score (Low risk, Intermediate risk/High risk) for FL patients only
- c) Grade of FL (1, 2, 3a)

TABLE 14.5.2) OVERALL SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION (ITT POPULATION)

| Time<br>(months) | Censoring<br>Indicator | Distribution<br>Function<br>Estimate | Failure | Survival<br>Standard<br>Error | Number<br>Failed | SDF Lower<br>Confidence<br>Limit | SDF Upper<br>Confidence<br>Limit |
|---|---|---|---|---|---|---|---|
| XXX | X | x.xxxx | X | X.XXXX | XXX | X.XXXX | x.xxx |
| XXX | X | x.xxx | X | x.xxxx | XXX | X.XXXX | X.XXXX |
| XXX | X | x.xxxx | X | X.XXXX | XXX | X.XXXX | x.xxxx |
| XXX | X | x.xxxx | X | X.XXXX | XXX | X.XXXX | x.xxxx |
| XXX | Х | X.XXXX | Х | x.xxxx | XXX | X.XXXX | X.XXXX |
| XXX | X | x.xxx | X | x.xxxx | XXX | X.XXXX | X.XXXX |

Data derived from Kaplan-Meier curve.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table should be presented for All Patients, DLBCL and FL groups. This table should be also presented from the first dose of Rituximab SC. This table should be also presented stratified by:

- a) Gender (Female, Male)
- b) FLIPI score (Low risk, Intermediate risk/High risk) for FL patients only
- c) Grade of FL (1, 2, 3a)

TABLE 14.5.3) OVERALL SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION CURVE FOR ALL SUBJECTS (ITT POPULATION)



Data derived from Kaplan-Meier curve.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table should be also presented from the first dose of Rituximab SC. This table should be also presented stratified by:

- a) Gender (Female, Male)
- b) FLIPI score (Low risk, Intermediate risk/High risk) for FL patients only
- c) Grade of FL (1, 2, 3a)

# Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

Mabrella ML28964 Daughter Protocol 141/Statistical Analysis Plan ML28964



Data derived from Kaplan-Meier curve.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table should be also presented from the first dose of Rituximab SC. This table should be also presented stratified by:

- a) Gender (Female, Male)
- b) FLIPI score (Low risk, Intermediate risk/High risk) for FL patients only
- C) Grade of FL (1, 2, 3a)

# Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

Mabrella ML28964 Daughter Protocol 142/Statistical Analysis Plan ML28964

TABLE 14.5.5) PROGRESSION FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV (ITT POPULATION)

| | Statistic | All Patients<br>(N=xxx) | DLBCL (N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Time to event (months) | 25th (95% CI)<br>Median (95% CI)<br>75th (95% CI) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) |
| Number of patients<br>Events<br>Censored | n (%)<br>n (%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |

Percentages are calculated on the number of patients in the ITT population.

PFS (months) was estimated using Kaplan-Meier method.

PFS is defined as the time from first dose of rituximab to the first occurrence of progression or relapse, or death from any cause, whichever occurs first.

Patients who have not experienced disease progression or death at the time of analysis and patients who are lost to follow up will be censored at their last clinical assessment date. Patients without post-baseline tumour assessments will be censored at the time of their baseline visit except if death occurs prior to their first scheduled tumour assessment.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table should be also presented from the first dose of Rituximab SC. This table should be also presented stratified by:

- d) Gender (Female, Male)
- e) FLIPI score (Low risk, Intermediate risk/High risk) for FL patients only
- f) Grade of FL (1, 2, 3a)
TABLE 14.5.6) PROGRESSION FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION (ITT POPULATION)

| Time (months) | Censoring<br>Indicator | Distribution<br>Function<br>Estimate | Failure | Survival<br>Standard<br>Error | Number<br>Failed | SDF Lower<br>Confidence<br>Limit | SDF Upper<br>Confidence<br>Limit |
|---|---|---|---|---|---|---|---|
| XXX | X | X.XXXX | X | X.XXXX | XXX | x.xxxx | x.xxxx |
| XXX | X | x.xxxx | X | X.XXXX | XXX | X.XXXX | X.XXXX |
| XXX | X | x.xxxx | X | X.XXXX | XXX | X.XXXX | X.XXXX |
| XXX | X | X.XXXX | X | x.xxxx | XXX | X.XXXX | X.XXXX |
| XXX | X | X.XXXX | X | x.xxxx | XXX | X.XXXX | X.XXXX |
| XXX | X | x.xxxx | X | x.xxxx | XXX | X.XXXX | x.xxxx |

Data derived from Kaplan-Meier curve.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table should be presented for All Patients, DLBCL and FL groups. This table should be also presented from the first dose of Rituximab SC. This table should be also presented stratified by:

- a) Gender (Female, Male)
- b) FLIPI score (Low risk, Intermediate risk/High risk) for FL patients only
- c) Grade of FL (1, 2, 3a)



Data derived from Kaplan-Meier curve.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table should be also presented from the first dose of Rituximab SC. This table should be also presented stratified by:

- a) Gender (Female, Male)
- b) FLIPI score (Low risk, Intermediate risk/High risk) for FL patients only
- c) Grade of FL (1, 2, 3a)

# Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

Mabrella ML28964 Daughter Protocol 145/Statistical Analysis Plan ML28964

TABLE 14.5.8) PROGRESSION FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION CURVE by TYPE OF LYMPHOMA (ITT POPULATION)



Data derived from Kaplan-Meier curve.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table should be also presented from the first dose of Rituximab SC. This table should be also presented stratified by:

- a) Gender (Female, Male)
- b) FLIPI score (Low risk, Intermediate risk/High risk) for FL patients only
- c) Grade of FL (1, 2, 3a)

# Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

Mabrella ML28964 Daughter Protocol 146/Statistical Analysis Plan ML28964

TABLE 14.5.9) DISEASE FREE SURVIVAL (ITT POPULATION)

| | Statistic | All Patients<br>(N=xxx) | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Time to event (months) | 25th (95% CI)<br>Median (95% CI)<br>75th (95% CI) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) |
| Number of patients | | | | |
| Events | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Censored | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Percentages are calculated on the number of patients in the ITT population.

DFS (months) was estimated using Kaplan-Meier method.

DFS will be assessed in patients achieving CR/CRu and is defined as the period from the date of the initial CR/CRu until the date of relapse or death from any cause. Patients who have not experienced disease progression or death at the time of analysis and patients who are lost to follow up will be censored at their last clinical assessment date.

TABLE 14.5.10) DISEASE FREE SURVIVAL: DISTRIBUCTION FUNCTION (ITT POPULATION)

| Time<br>(months) | Censoring<br>Indicator | Distribution<br>Function<br>Estimate | Failure | Survival<br>Standard<br>Error | Number<br>Failed | SDF Lower<br>Confidence<br>Limit | SDF Upper<br>Confidence<br>Limit |
|---|---|---|---|---|---|---|---|
| xxx | х | x.xxxx | х | x.xxxx | xxx | x.xxxx | x.xxxx |
| XXX | X | x.xxxx | X | x.xxxx | XXX | x.xxxx | x.xxxx |
| XXX | X | x.xxxx | X | x.xxxx | XXX | X.XXXX | x.xxxx |
| XXX | X | X.XXXX | X | x.xxxx | XXX | X.XXXX | X.XXXX |
| XXX | X | X.XXXX | X | X.XXXX | XXX | X.XXXX | X.XXXX |
| XXX | X | X.XXXX | X | X.XXXX | XXX | X.XXXX | X.XXXX |

Data derived from Kaplan-Meier curve.

Source: XXXX.SAS, Run on DDMMMYYYY

## Programming note:

This table should be presented for All Patients, DLBCL and FL groups.

TABLE 14.5.11) DISEASE FREE SURVIVAL: DISTRIBUCTION FUNCTION CURVE FOR ALL SUBJECTS (ITT POPULATION)



Data derived from Kaplan-Meier curve.

TABLE 14.5.12) DISEASE FREE SURVIVAL: DISTRIBUCTION FUNCTION CURVE BY TYPE OF LYMPHOMA (ITT POPULATION)



Data derived from Kaplan-Meier curve.

Source: XXXX.SAS, Run on DDMMMYYYY

Mabrella ML28964 Daughter Protocol 150/Statistical Analysis Plan ML28964

TABLE 14.5.13) EVENT FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV (ITT POPULATION)

| | Statistic | All Patients<br>(N=xxx) | DLBCL (N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| Time to event (months) | 25th (95% CI)<br>Median (95% CI)<br>75th (95% CI) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) | xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x)<br>xxx.x (xxx.x,xxx.x) |
| Number of patients<br>Events<br>Censored | n (%)<br>n (%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |

Percentages are calculated on the number of patients in the ITT population.

EFS (months) was estimated using Kaplan-Meier method.

EFS is defined as the time from first dose of rituximab to first occurrence of progression or relapse, or initiation of a non-protocol-specified anti-lymphoma therapy or death, whichever occurs first.

Patients who have not experienced disease progression or relapse or initiation of a non-protocol-specified anti-lynphoma therapy or death at the time of analysis and patients who are lost to follow up will be censored at their last clinical assessment date.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table should be also presented from the first dose of Rituximab SC.

TABLE 14.5.14) EVENT FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION (ITT POPULATION)

| Time<br>(months) | Censoring<br>Indicator | Distribution<br>Function<br>Estimate | Failure | Survival<br>Standard<br>Error | Number<br>Failed | SDF Lower<br>Confidence<br>Limit | SDF Upper<br>Confidence<br>Limit |
|---|---|---|---|---|---|---|---|
| xxx | х | x.xxxx | х | x.xxxx | xxx | x.xxxx | x.xxxx |
| XXX | X | x.xxxx | X | x.xxxx | XXX | x.xxxx | x.xxxx |
| XXX | X | x.xxxx | X | x.xxxx | XXX | X.XXXX | x.xxxx |
| XXX | X | X.XXXX | X | x.xxxx | XXX | X.XXXX | X.XXXX |
| XXX | X | X.XXXX | X | X.XXXX | XXX | X.XXXX | X.XXXX |
| XXX | X | X.XXXX | X | X.XXXX | XXX | X.XXXX | X.XXXX |

Data derived from Kaplan-Meier curve.

Source: XXXX.SAS, Run on DDMMMYYYY

## Programming note:

This table should be presented for All Patients, DLBCL and FL groups. This table should be also presented from the first dose of Rituximab SC.

TABLE 14.5.15) EVENT FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION CURVE FOR ALL SUBJECTS (ITT POPULATION)



Data derived from Kaplan-Meier curve.

Source: XXXX.SAS, Run on DDMMMYYYY

### Programming note:

This table should be also presented from the first dose of Rituximab SC.

TABLE 14.5.16) EVENT FREE SURVIVAL FROM FIRST DOSE OF RITUXIMAB IV: DISTRIBUCTION FUNCTION CURVE BY TYPE OF LYMPHOMA (ITT POPULATION)



Data derived from Kaplan-Meier curve.

Source: XXXX.SAS, Run on DDMMMYYYY

## Programming note:

This table should be also presented from the first dose of Rituximab SC.

# Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

TABLE 14.5.17) SUMMARY OF COMPLETE RESPONSE OR COMPLETE RESPONSE UNCONFIRMED (ITT POPULATION)

| | Statistic | All Patients<br>(N=xxx) | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|
| CR | n/N1 (%) - 95% CI | xx/XXX (xx.x%) - xx.x,xx.x | xx/XXX (xx.x%) - xx.x,xx.x | xx/XXX (xx.x%) - xx.x,xx.x |
| CRu (unconfirmed)<br>CR/CRu | n/N1 (%) - 95% CI<br>n/N1 (%) - 95% CI | xx/XXX (xx.x%) - xx.x,xx.x<br>xx/XXX (xx.x%) - xx.x,xx.x | xx/XXX (xx.x%) - xx.x,xx.x<br>xx/XXX (xx.x%) - xx.x,xx.x | xx/XXX (xx.x%) - xx.x,xx.x<br>xx/XXX (xx.x%) - xx.x,xx.x |

CR = Complete Response. CRu = Complete Response Unconfirmed.

N1=Number of patients have evaluable overall lesion assessment data.

Two-sided Clopper-Pearson confidence interval.

Tumour assessment measured four weeks after the end of the Induction treatment.

Number of patients performing the tumour assessment was used as denominator.

TABLE 14.6.1) RITUXIMAB IV ADMINISTRATION SATIFICATION QUESTIONNAIRE - ITEMS FREQUENCY ANALYSIS (SAFETY POPULATION)

| | | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|---|
| Study Visit <xxx></xxx> | Was the RASQ questionnaire completed? | | | | |
| ocuay vibic (xxx) | No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | 1. Thinking about the Rituximab IV infusion, how satisfied or | | | | |
| | dissatisfied are you with the IV infusion? | | | | |
| | Very satisfied | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Satisfied | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Neither satisfied nor dissatisfied | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Dissatisfied | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Very dissatisfied | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Patient did not answer question | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | 2. Thinking about the Rituximab IV infusion, how do you rate the | | | | |
| | pain, swelling or redness you experienced at the site of the drug | | | | |
| | infusion? | | | | |
| | None | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Mild | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Moderate | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Severe | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Very severe | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Patient did not answer question | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of patients in SAF population performing the RASQ questionnaire for Rituximab IV administration.

Source: XXXX.SAS, Run on DDMMMYYYY

## Programming note:

All items of RASQ questionnaire for Rituximab IV administration must be presented.

TABLE 14.6.2) RITUXIMAB SC ADMINISTRATION SATIFICATION QUESTIONNAIRE - ITEMS FREQUENCY ANALYSIS (SAFETY POPULATION)

| | | Statistic | All Patients (N=xxx) | DLBCL<br>(N=xxx) | FL<br>(N=xxx) |
|---|---|---|---|---|---|
| Study Visit <xxx></xxx> | Was the RASQ questionnaire completed? | | | | |
| | No | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Yes | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | 1. Thinking about the Rituximab SC injection, how satisfied or | | | | |
| | dissatisfied are you with the SC injection? | | | | |
| | Very satisfied | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx,x%) |
| | Satisfied | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Neither satisfied nor dissatisfied | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Dissatisfied | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Very dissatisfied | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Patient did not answer question | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | 2. Thinking about the Rituximab SC injection, how do you rate the | | | | |
| | pain, swelling or redness you experienced at the site of the drug | | | | |
| | infusion? | | | | |
| | None | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Mild | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Moderate | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Severe | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Very severe | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | Patient did not answer question | n (%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of patients in SAF population performing the RASQ questionnaire for Rituximab SC administration.

Source: XXXX.SAS, Run on DDMMMYYYY

## Programming note:

All items of RASQ questionnaire for Rituximab SC administration must be presented.

TABLE 14.6.3) SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE IV MEAN SCORES (SAFETY POPULATION)

| | | All Patients | DLBCL | FL |
|----------|-----------|--------------|--------------|-------------|
| | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | xx.x | XX.X | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |

TABLE 14.6.4) SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE IV MEAN SCORES (SAFETY POPULATION)

| Psychological Im | pact domain | | | |
|---|---|---|---|---|
| | Statistic | All Patients (N=xx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
| | | (N AA) | (N AA) | |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |

TABLE 14.6.5) SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE IV MEAN SCORES (SAFETY POPULATION)

Impact on Activities of Daily Living domain All Patients FLDLBCL Statistic (N=xx)(N=xx)(N=xx)Visit xx Mean (SD) xx.x (xx.xx) xx.x (xx.xx)xx.x (xx.xx) Median XX.X XX.X XX.X Min/Max xx.x/xx.x xx.x/xx.x xx.x/xx.x Visit xx Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median XX.X XX.X XX.X Min/Max xx.x/xx.x xx.x/xx.x xx.x/xx.x Visit xx XX XX XX Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median XX.X XX.X XX.X Min/Max xx.x/xx.x xx.x/xx.x xx.x/xx.x

TABLE 14.6.6) SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE IV MEAN SCORES (SAFETY POPULATION)

Convenience domain All Patients DLBCL FL Statistic (N=xx) (N=xx) (N=xx)Visit xx Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x XX.X Min/Max xx.x/xx.x Visit xx Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median XX.X XX.X XX.X Min/Max xx.x/xx.x xx.x/xx.x xx.x/xx.x Visit xx XX Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median xx.x XX.X XX.X Min/Max xx.x/xx.x xx.x/xx.x xx.x/xx.x

TABLE 14.6.7) SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE IV MEAN SCORES (SAFETY POPULATION)

| Satisfaction domain | | All Patients | DLBCL | FL |
|---------------------|-----------|--------------|--------------|--------------|
| | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Visit xx | n | xx | xx | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | xx.x | xx.x | xx.x |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |

TABLE 14.6.8) SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE SC MEAN SCORES (SAFETY POPULATION)

| | | All Patients | DLBCL | FL |
|----------|-----------|--------------|--------------|--------------|
| | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | XX | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | XX | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |

TABLE 14.6.9) SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE SC MEAN SCORES (SAFETY POPULATION)

| Psychological Impa | act domain | | | |
|---|---|---|---|---|
| | Statistic | All Patients<br>(N=xx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | xx.x |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |

TABLE 14.6.10) SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE SC MEAN SCORES (SAFETY POPULATION)

Impact on Activities of Daily Living domain All Patients FLDLBCL Statistic (N=xx) (N=xx)(N=xx)Visit xx Mean (SD) xx.x (xx.xx) xx.x (xx.xx)xx.x (xx.xx) Median XX.X XX.X XX.X Min/Max xx.x/xx.x xx.x/xx.x xx.x/xx.x Visit xx Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median XX.X XX.X XX.X Min/Max xx.x/xx.x xx.x/xx.x xx.x/xx.x Visit xx XX XX XX Mean (SD) xx.x (xx.xx) xx.x (xx.xx) xx.x (xx.xx) Median XX.X XX.X XX.X Min/Max xx.x/xx.x xx.x/xx.x xx.x/xx.x

TABLE 14.6.11) SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE SC MEAN SCORES (SAFETY POPULATION)

| Convenience domain | | All Patients | DLBCL | FI. |
|--------------------|-----------|--------------|--------------|--------------|
| | Statistic | (N=xx) | (N=xx) | (N=xx) |
| Visit xx | n | xx | xx | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | xx.x | XX.X | xx.x |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |

TABLE 14.6.12) SUMMARY OF RITUXIMAB ADMINISTRATION SATISFACTION QUESTIONNAIRE SC MEAN SCORES (SAFETY POPULATION)

| Satisfaction domain | Statistic | All Patients (N=xx) | DLBCL<br>(N=xx) | FL<br>(N=xx) |
|---|---|---|---|---|
| Visit xx | n | XX | XX | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | XX | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |
| Visit xx | n | xx | XX | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | XX.X |
| | Min/Max | xx.x/xx.x | xx.x/xx.x | xx.x/xx.x |

TABLE 14.6.13) HEALTHCARE PROFESSIONAL QUESTIONNAIRE (PART #1)

| | | All Healthcare<br>Professionals<br>(N=xxx) |
|---|---|---|
| Was the HCP questionnaire completed? | | |
| No | n (%) | xxx (xx.x%) |
| Yes | n (%) | xxx (xx.x%) |
| 1.Did you personally administer the SC Rituximab in the study? | | |
| Always | n (%) | xxx (xx.x%) |
| Sometimes | n (%) | xxx (xx.x%) |
| Never | n (%) | xxx (xx.x%) |
| 1a. If never, who did administer the SC Rituximab in the study? | | |
| Other hematologist | n (%) | xxx (xx.x%) |
| Other internist | n (%) | xxx (xx.x%) |
| Oncology/chemo nurse | n (%) | xxx (xx.x%) |
| Other | n (%) | xxx (xx.x%) |
| 2. How many minutes preparation time was required after receiving the Rituximab vial from the pharmacy? | | |
| <5 | n (%) | xxx (xx.x%) |
| 6-10 | n (%) | xxx (xx.x%) |
| 11-15 | n (%) | xxx (xx.x%) |
| 16-20 | n (%) | xxx (xx.x%) |
| >20 | n (%) | xxx (xx.x%) |
| Not sure | n (%) | xxx (xx.x%) |
| 3. How many minutes in total did it usually take to administer the Rituximab subcutaneously using the hand held syringe? | | |
| <5 | n (%) | xxx (xx.x%) |
| 6-15 | n (%) | xxx (xx.x%) |
| 16-30 | n (%) | xxx (xx.x%) |
| 31-60 | n (%) | xxx (xx.x%) |
| 61-90 | n (%) | xxx (xx.x%) |
| >90 | n (%) | xxx (xx.x%) |
| Not sure | n (%) | xxx (xx.x%) |
| 4. How long do you think the SC sessions usually lasted from patients' arrival until departure | | |
| <2 hours | n (%) | xxx (xx.x%) |
| >2 but <3 hours | n (%) | xxx (xx.x%) |
| >3 but <4 hours | n (%) | xxx (xx.x%) |
| 5. How anxious do you think the SC treatment made patients feel? | | |
| Not al all | n (%) | xxx (xx.x%) |
| Fairly | n (%) | xxx (xx.x%) |
| Very | n (%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of healthcare professional performing the HCP questionnaire.

Source: XXXX.SAS, Run on DDMMMYYYY

# Rituximab - Roche North Africa (Algeria, Morocco & Tunisia)

Mabrella ML28964 Daughter Protocol 168/Statistical Analysis Plan ML28964

TABLE 14.6.14) HEALTHCARE PROFESSIONAL QUESTIONNAIRE (PART #2)

| | Statistic | |
|---|---|---|
| 6. How reliable was using the hand held syringe to give Rituximab | | |
| subcutaneously? | | |
| Not at all | n (%) | xxx (xx.x%) |
| Fairly | n (%) | xxx (xx.x%) |
| Very | n (%) | xxx (xx.x%) |
| Extremely | n (%) | xxx (xx.x%) |
| 7.Overall how easy did you/your staff find giving Rituximab subcutaneously using the hand held syringe? | | |
| Not at all | n (%) | xxx (xx.x%) |
| Fairly | n (%) | xxx (xx.x%) |
| Very | n (%) | xxx (xx.x%) |
| Extremely | n (%) | xxx (xx.x%) |
| 8. How likely would you be to offer or recommend SC administration of Rituximab via a hand held syringe to your patients in the future? | | |
| Not at all | n (%) | xxx (xx,x%) |
| Fairly | n (%) | xxx (xx.x%) |
| Very | n (%) | xxx (xx.x%) |
| Extremely | n (%) | xxx (xx.x%) |
| 9.In general how would you describe your experience regarding the Rituximab SC treatment? | | |
| Satisfactory | n (%) | xxx (xx.x%) |
| Unsatisfactory | n (%) | xxx (xx.x%) |

Percentages are calculated relative to the total number of healthcare professional performing the HCP questionnaire.

LISTING 16.2.1)1. ANALYSIS SETS

| Site | Intent-To-Treat<br>Population | Safety<br>Population | Reason for Exclusion<br>from Safety<br>Population | Type of<br>Lymphoma |
|---|---|---|---|---|
| XXXX | XXX | XXX | XXX | XXX |
| XXXX | XXX | XXX | XXX | XXX |
| XXXX | XXX | XXX | XXX | XXX |
| XXXX | XXX | XXX | XXX | XXX |
| XXXX | XXX | XXX | XXX | XXX |
| XXXX | XXX | XXX | XXX | XXX |
| XXXX | xxx | XXX | XXX | XXX |
| | XXXX<br>XXXX<br>XXXX<br>XXXX | XXXX XXX<br>XXXX XXX<br>XXXX XXX<br>XXXX XXX<br>XXXX XXX | XXXX | Population |

LISTING 16.2.1)2. INCLUSION/EXCLUSION CRITERIA VIOLATED

| Patient | Type of<br>Lymphoma | Failed Criteria |
|---------|---------------------|-----------------|
| xxxx | xxxx | xxx |
| XXXX | XXXX | xxx |
| XXXX | XXXX | xxx |
| XXXX | XXXX | XXX |

Only I/E criteria failed are reported in this line listing.

LISTING 16.2.2)1. MAJOR PROTOCOL DEVIATIONS

| Patient | Type of<br>Lymphoma | Category | Description of Deviation |
|---------|---------------------|----------|--------------------------|
| xxxx | xxxx | xxxxx | xxxxx<br>xxxxx |
| xxxx | xxxx | xxxxx | xxxxx |
| xxxx | xxxx | xxxxx | xxxxx |

LISTING 16.2.2)2. MINOR PROTOCOL DEVIATIONS

| Patient | Type of<br>Lymphoma | Category | Description of Deviations |
|---------|---------------------|----------|---------------------------|
| xxxx | xxxx | xxxxx | XXXXX |
| xxxx | xxxx | xxxxx | xxxxx |
| xxxx | xxxx | xxxxx | xxxxx |

LISTING 16.2.2)3. COVID-19 RELATED PROTOCOL DEVIATIONS

| Patient | Type of<br>Lymphoma | Category | Description of Deviations |
|---------|---------------------|----------|---------------------------|
| xxxx | xxxx | xxxxx | xxxx<br>xxxx |
| xxxx | xxxx | xxxxx | xxxxx |
| xxxx | xxxx | xxxxx | xxxxx |

LISTING 16.2.3)1. STUDY DRUG DISCONTINUATION

| Patient | Type of<br>Lymphoma | Study Drug<br>Discontinued? | Date of Trt<br>Discontinuation | Primary Reason If Other, for trt Specify Discontinuation | | Date of Last<br>Rituximab Dose | Date of Last<br>Chemotherapy<br>Dose | Will the Patient<br>Proceed the FUP? |
|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | DDMMMYYYY | xxx | xxx | DDMMMYYYY | DDMMMYYYY | xxx |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | DDMMMYYYY | DDMMMYYYY | XXX |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | DDMMMYYYY | DDMMMYYYY | xxx |
| xxxx | xxxx | XXXX | DDMMMYYYY | XXX | xxx | DDMMMYYYY | DDMMMYYYY | xxx |

LISTING 16.2.4)1. INFORMED CONSENT & DEMOGRAPHY

| Patient | Type of<br>Lymphoma | Was IC<br>Obtained? | Date of<br>Consent | Date of<br>Birth | Age<br>(yrs) | Sex | If Female,<br>Childbearing<br>Potential | Ethnicity | If Other, Specify | Derived Age from Birth<br>Year and ICF Date | Height<br>(cm) | Weight<br>(Kg) | BMI<br>(Kg/m^2) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | DDMMMYYYY | DDMMMYYYY | xxx | xxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxx | xxx | xxx |
| XXXX | XXXX | XXXX | DDMMMYYYY | DDMMMYYYY | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXX | XXX |
| XXXX | XXXX | XXXX | DDMMMYYYY | DDMMMYYYY | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXX | XXX |
| XXXX | XXXX | XXXX | DDMMMYYYY | DDMMMYYYY | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXX | XXX |

LISTING 16.2.4)2. MEDICAL HISTORY

| Patient | Type of<br>Lymphoma | No. | Medical<br>History<br>Term | LLT | PΤ | SOC | Start Date (DDMMMYYYY) | Stop Date<br>(DDMMMYYYY) | Ongoing at<br>Study Entry? |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | х | Xxxxxxx | xxxx | xxxx | xxxx | DDMMMYYYY | DDMMMYYYY | xxxxxx |
| XXXX | XXXX | x | Xxxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | DDMMMYYYY | XXXXXX |
| XXXX | xxxx | Х | Xxxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | DDMMMYYYY | xxxxxx |
| xxxx | xxxx | х | Xxxxxxx | xxxx | XXXX | xxxx | DDMMMYYYY | DDMMMYYYY | XXXXXX |

LISTING 16.2.4)3. SURGERY AND PROCEDURES HISTORY (CANCER AND NON-CANCER RELATED)

| Patient | Type of<br>Lymphoma | No. | Has patient Any Cancer or Non-Cancer Surgeries? | History Type | Surgery/Procedure | Date of<br>Surgery/Procedure |
|---|---|---|---|---|---|---|
| xxxx | xxxx | х | Xxxxxxx | xxxx | xxxx | DDMMMYYYY |
| XXXX | XXXX | Х | Xxxxxxx | XXXX | xxxx | DDMMMYYYY |
| XXXX | XXXX | Х | Xxxxxxx | XXXX | xxxx | DDMMMYYYY |
| xxxx | XXXX | Х | Xxxxxxx | XXXX | xxxx | DDMMMYYYY |

LISTING 16.2.4)4. DLBCL DIAGNOSIS

| Patient | Type of<br>Lymphoma | Date of<br>Histological<br>Diagnosis | How Was Histological<br>Diagnosis Obtained? | If Fine Needle Aspiration, Provide Details | CD20+ Expression |
|---|---|---|---|---|---|
| xxxx | xxxx | DDMMMYYYY | xxx | XXX | xxxxxx |
| XXXX | xxxx | DDMMMYYYY | xxx | xxx | xxxxxx |
| XXXX | XXXX | DDMMMYYYY | xxx | xxx | XXXXXX |
| xxxx | XXXX | DDMMMYYYY | xxx | XXX | xxxxxx |
LISTING 16.2.4)5. FOLLICULAR LYMPHOMA DIAGNOSIS

| Patient | Type of<br>Lymphoma | Date of<br>Histological<br>Diagnosis | How Was Histological<br>Diagnosis Obtained? | If Fine Needle Aspiration,<br>Provide Details | Grade of FL | CD20+ Expression |
|---|---|---|---|---|---|---|
| xxxx | xxxx | DDMMMYYYY | xxx | xxx | xxxxxx | xxxxxx |
| XXXX | XXXX | DDMMMYYYY | xxx | XXX | XXXXXX | xxxxxx |
| XXXX | XXXX | DDMMMYYYY | xxx | XXX | XXXXXX | xxxxxx |
| XXXX | XXXX | DDMMMYYYY | xxx | XXX | XXXXXX | xxxxxx |

LISTING 16.2.4)6. ECOG PERFORMANCE STATUS, FLIPI AND IPI SCORE

| Patient | Type of<br>Lymphoma | Date of<br>Assessment<br>of ECOG PS | ECOG PS | Date of<br>Assessment<br>of FLIPI<br>Score | FLIPI Score | Date of<br>Assessment<br>of IPI Score | IPI Score |
|---|---|---|---|---|---|---|---|
| xxxx | xxxx | DDMMMYYYY | xxx | DDMMMYYYY | xxx | DDMMMYYYY | XXX |
| XXXX | XXXX | DDMMMYYYY | XXX | DDMMMYYYY | XXX | DDMMMYYYY | XXX |
| XXXX | XXXX | DDMMMYYYY | XXX | DDMMMYYYY | XXX | DDMMMYYYY | XXX |
| XXXX | XXXX | DDMMMYYYY | XXX | DDMMMYYYY | XXX | DDMMMYYYY | XXX |

LISTING 16.2.4)7. VIRAL SEROLOGY AT SCREENING

| Patient | Type of<br>Lymphoma | Was Viral<br>Serology Sample<br>Collected? | Date of Sample<br>Collection | HBcAb | HbsAg | HCV<br>Antibody | HIV<br>Antibody | Viral Infection<br>with HBV or HCV? |
|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | DDMMMYYYY | xxx | xxx | xxx | xxx | xxx |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | xxx |
| XXXX | XXXX | xxxx | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | xxx |

# LISTING 16.2.4)8. CONCOMITANT MEDICATIONS

| Patient | Type of<br>Lymphoma | No. | Medication<br>Name | PT | SOC | Reason for<br>Medication | If Other,<br>Specify | Indication | Start Date (DDMMMYYYY) | Dose | Dose<br>Unit | Freq. | Route | If Other, Specify | Stop Date<br>(DDMMMYYYY) | Ongoing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | х | Xxxxxxx | XXXX | xxxx | xxx | xxx | xxx | DDMMMYYYY | xxx | xxx | XXX | xxxxx | xxxxxx | DDMMMYYYY | xxxxxx |
| XXXX | XXXX | Х | Xxxxxx | XXXX | XXXX | XXX | XXX | XXX | DDMMMYYYY | XXX | XXX | XXX | XXXXXX | xxxxxx | DDMMMYYYY | XXXXXX |
| XXXX | XXXX | х | Xxxxxx | XXXX | XXXX | XXX | XXX | XXX | DDMMMYYYY | XXX | XXX | XXX | XXXXXX | xxxxxx | DDMMMYYYY | XXXXXX |
| XXXX | XXXX | х | Xxxxxx | XXXX | XXXX | XXX | XXX | XXX | DDMMMYYYY | XXX | XXX | XXX | XXXXXX | xxxxxx | DDMMMYYYY | XXXXXX |

LISTING 16.2.5)1. PREVIOUS IV RITUXIMAB DOSE - DLBCL

| Patient | Type of<br>Lymphoma | No. of Previous<br>IV Rituximab<br>Treatment Cycles | Dose of Most<br>Recent IV<br>Rituximab<br>Cycle | Date of 1 <sup>st</sup><br>Rituximab IV<br>Administration | Wich Treatment Cycle is<br>the Subject's First<br>on-Study Cycle? |
|---|---|---|---|---|---|
| xxxx | xxxx | xxx | xxx | DDMMMYYYY | xxx |
| XXXX | XXXX | XXX | XXX | DDMMMYYYY | XXX |
| XXXX | xxxx | XXX | xxx | DDMMMYYYY | xxx |
| XXXX | XXXX | xxx | XXX | DDMMMYYYY | xxx |

LISTING 16.2.5)2. PREVIOUS IV RITUXIMAB DOSE - FL

| Patient | Type of<br>Lymphoma | Phase of IV<br>Rituximab | No. of Cycles<br>of IV<br>Rituximab<br>Recived<br>Previously | Date of 1 <sup>st</sup><br>Rituximab IV<br>Administration | Dose of Most<br>Recent IV<br>Rituximab<br>Cycle | Eligible Phase<br>to Enter the<br>Study | Wich Treatment Cycle is<br>the Subject's First<br>on-Study Cycle? |
|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xxx | xxx | DDMMMYYYY | xxx | xxx | xxx |
| XXXX | XXXX | XXX | XXX | DDMMMYYYY | XXX | XXX | xxx |
| XXXX | XXXX | XXX | XXX | DDMMMYYYY | XXX | XXX | xxx |
| XXXX | XXXX | xxx | xxx | DDMMMYYYY | xxx | xxx | XXX |

LISTING 16.2.5)3. INITIAL CHOP

| Patient | Type of<br>Lymphoma | Start Date<br>of CHOP | Cyclophosphamide<br>Fixed Unit<br>(mg/m^2) | Doxorubicin<br>Fixed Unit<br>(mg/m^2) | Vincristine<br>Fixed Unit<br>(mg/m^2) | Prednisone/Prednisolone<br>Fixed Unit<br>(mg/m^2) |
|---|---|---|---|---|---|---|
| xxxx | xxxx | DDMMMYYYY | xxx | xxx | xxx | xxx |
| XXXX | XXXX | DDMMMYYYY | xxx | XXX | XXX | xxx |
| XXXX | XXXX | DDMMMYYYY | xxx | XXX | XXX | xxx |
| xxxx | xxxx | DDMMMYYYY | xxx | XXX | XXX | xxx |

LISTING 16.2.5)4. SUBSEQUENT CHOP

| Patient | Type of<br>Lymphoma | Cycle | If Patient Receiving Same<br>Regimen as in the Previous<br>Cycle? | Start Date | If No, Specify Regimen Moved Onto |
|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | xxxx | DDMMMYYYY | xxx |
| XXXX | XXXX | XXXX | XXXX | DDMMMYYYY | XXX |
| XXXX | XXXX | XXXX | XXXX | DDMMMYYYY | XXX |
| XXXX | XXXX | XXXX | xxxx | DDMMMYYYY | XXX |

LISTING 16.2.5)5. SUBSEQUENT CVP

| Patient | Type of<br>Lymphoma | Cycle | If Patient Receiving Same<br>Regimen as in the Previous<br>Cycle? | Start Date | If No, Specify Regimen Moved Onto |
|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | xxxx | DDMMMYYYY | xxx |
| XXXX | XXXX | XXXX | xxxx | DDMMMYYYY | XXX |
| XXXX | XXXX | XXXX | xxxx | DDMMMYYYY | XXX |
| XXXX | XXXX | XXXX | xxxx | DDMMMYYYY | XXX |

LISTING 16.2.5)6. SUBSEQUENT FLUDARABINE

| Patient | Type of<br>Lymphoma | Cycle | If Patient Receiving Same<br>Regimen as in the Previous<br>Cycle? | Start Date | If No, Specify Regimen Moved Onto |
|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | xxxx | DDMMMYYYY | xxx |
| XXXX | XXXX | XXXX | XXXX | DDMMMYYYY | XXX |
| XXXX | XXXX | XXXX | XXXX | DDMMMYYYY | XXX |
| XXXX | XXXX | XXXX | xxxx | DDMMMYYYY | XXX |

LISTING 16.2.5)7. SUBSEQUENT CHEMOTHERAPY

| Patient | Type of<br>Lymphoma | Cycle | If Patient Receiving Same<br>Regimen as in the Previous<br>Cycle? | Start Date | If No, Specify Regimen Moved Onto |
|---|---|---|---|---|---|
| xxxx | xxxx | xxxx<br>xxxx<br>xxxx | XXXX<br>XXXX<br>XXXX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | xxx<br>xxx<br>xxx |
| xxxx | xxxx | xxxx<br>xxxx | XXXX<br>XXXX<br>XXXX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | XXX<br>XXX<br>XXX |

LISTING 16.2.5)8. INITIAL CVP

| Patient | Type of<br>Lymphoma | Start Date<br>of CVP | Cyclophosphamide<br>Fixed Unit<br>(mg/m^2) | Vincristine<br>Fixed Unit<br>(mg/m^2) | Prednisone/Prednisolone<br>Fixed Unit<br>(mg/m^2) |
|---|---|---|---|---|---|
| xxxx | xxxx | DDMMMYYYY | xxx | xxx | xxx |
| XXXX | XXXX | DDMMMYYYY | xxx | XXX | xxx |
| XXXX | XXXX | DDMMMYYYY | xxx | XXX | xxx |
| XXXX | XXXX | DDMMMYYYY | xxx | XXX | xxx |

LISTING 16.2.5) 9. INITIAL FLUDARABINE

| Patient | Type of<br>Lymphoma | Start Date | Fludarabine<br>Fixed Unit<br>(mg/m^2) | Cyclophosphamide<br>Fixed Unit<br>(mg/m^2) |
|---|---|---|---|---|
| xxxx | xxxx | DDMMMYYYY | xxx | xxx |
| xxxx | XXXX | DDMMMYYYY | XXX | xxx |
| XXXX | XXXX | DDMMMYYYY | xxx | xxx |
| XXXX | XXXX | DDMMMYYYY | xxx | xxx |

LISTING 16.2.5)10. OTHER CHEMOTHERAPY

| | ype of<br>ymphoma | Chemotherapy Agent | Regimen<br>Start Date | Dose | Unit | Regimen<br>Stop Date |
|---|---|---|---|---|---|---|
| xxxx x | xxx | xxxx | DDMMMYYYY | xxx | xxx | DDMMMYYYY |
| xxxx x | XXXX | xxxx | DDMMMYYYY | XXX | XXX | DDMMMYYYY |
| xxxx x | XXXX | xxxx | DDMMMYYYY | XXX | XXX | DDMMMYYYY |
| xxxx x | XXXX | xxxx | DDMMMYYYY | XXX | XXX | DDMMMYYYY |

LISTING 16.2.5)11. STUDY DRUG ADMINISTRATION

| Patient | Type of<br>Lymphoma | Visit | Was Rituximab<br>Administered? | Start Date | Start<br>Time | Stop Date | Stop<br>Time | Intended<br>Total Dose | Actual<br>Total Dose | Was Full<br>e Dose Given? | If No,<br>Provide<br>Reason | If Other,<br>Specify | If AE, is<br>Grade 3-4<br>IIRR? | Drug<br>Administered<br>on time per<br>Schedule | If No,<br>Specify |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | DDMMMYYYY | le le | DDMMMYYYY | hh:mm | | | | | | | | |
| XXXX | XXXX | XXXX | XXXX | | hh:mm | | | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | | XXXX | XXXX | DDMMMYYYY | hh:mm | DDMMMYYYY | hh:mm | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | | XXXX | XXXX | DDMMMYYYY | hh:mm | DDMMMYYYY | hh:mm | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | | XXXX | XXXX | DDMMMYYYY | hh:mm | DDMMMYYYY | hh:mm | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXXX | XXXX | XXXX | XXXX | DDMMMYYYY | hh:mm | DDMMMYYYY | hh:mm | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | | XXXX | XXXX | DDMMMYYYY | hh:mm | DDMMMYYYY | hh:mm | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | | XXXX | XXXX | DDMMMYYYY | hh:mm | DDMMMYYYY | hh:mm | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | | XXXX | XXXX | DDMMMYYYY | hh:mm | DDMMMYYYY | hh:mm | XXX | XXX | XXX | XXX | xxx | xxx | xxx | xxx |

LISTING 16.2.5)12. ANTI-LYMPHOMA CHEMO/IMMUNO THERAPY TREATMENT

| Patient | Type of<br>Lymphoma | New Chemo/Immuno<br>Therapy for FL | Seq. | Drug Name | Cumulative<br>Dose | Unit | No.<br>Cycles | Start Date | End Date | Response |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xxxxx | xxx | xxx | xxx | xxx | xxx | DDMMMYYYY | DDMMMYYYY | xxx |
| XXXX | XXXX | xxxxx | XXX | XXX | XXX | XXX | XXX | DDMMMYYYY | DDMMMYYYY | XXX |
| XXXX | XXXX | xxxxx | XXX | XXX | XXX | XXX | XXX | DDMMMYYYY | DDMMMYYYY | XXX |
| xxxx | XXXX | xxxxx | XXX | XXX | XXX | xxx | XXX | DDMMMYYYY | DDMMMYYYY | XXX |

LISTING 16.2.5)13. ANTI-LYMPHOMA RADIOTHERAPY TREATMENT

| Patient | Type of<br>Lymphoma | New Radiotherapy<br>for FL | Seq. | Irradiation<br>Site | If Other,<br>Specify | Cumulative<br>Dose | Unit | Start Date | End Date | Response |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | XXXXX<br>XXXXX<br>XXXXX | XXX<br>XXX<br>XXX | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | xxx<br>xxx<br>xxx |

LISTING 16.2.5)14. ANTI-LYMPHOMA TREATMENT

| Patient | Type of<br>Lymphoma | New Non-Protocol Specified<br>Anti-Lymphoma Treatment | Start Date | Anti-Lymphoma<br>Treatment | Radiotherapy | Chemo-Immuno<br>Therapy |
|---|---|---|---|---|---|---|
| xxxx | xxxx | Х | DDMMMYYYY | xxxxx | xxxxx | xxxxx |
| XXXX | XXXX | Х | DDMMMYYYY | XXXXX | XXXXX | xxxxx |
| XXXX | XXXX | Х | DDMMMYYYY | xxxxx | XXXXX | xxxxx |
| XXXX | XXXX | х | DDMMMYYYY | xxxxx | XXXXX | xxxxx |
| ΔΛΛΛ | AAAA | A | DDMMIIIII | ΑΛΛΛΛ | AAAAA | AAAAA |

LISTING 16.2.5)15. CHEMOTHERAPY SELECTION

| Patient | Type of<br>Lymphoma | Chemotherapy<br>Regiment | If Other, Specify |
|---------|---------------------|--------------------------|-------------------|
| xxxx | xxxx | xxxxx | xxxxx |
| XXXX | XXXX | XXXXX | xxxxx |
| XXXX | XXXX | XXXXX | XXXXX |
| XXXX | XXXX | XXXXX | XXXXX |

### LISTING 16.2.6)1. PRE-TREATMENT ADVERSE EVENTS

| Patient | Type of<br>Lymphoma | No. | Description | LLT | PT | SOC | Start Date (DDMMMYYYY) | SAE | Initial<br>Intensity | AESI | AAR | Extreme<br>Intensity | Relation to<br>Chemotherapy | Action<br>Taken with<br>Chemotherapy | AE Required<br>Treatment | Outcome | End Date (DDMMMYYYY) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | х | Xxxxxxx | xxxx | xxxx | xxxx | DDMMMYYYY | xxx | xxx | xxx | xxx | xxx | xxxxxx | xxxxxx | xxx | xxxxxx | DDMMMYYYY |
| XXXX | XXXX | x | Xxxxxxx | XXXX | XXXX | | | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY |
| XXXX | XXXX | х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | xxx | XXX | XXX | XXXXXX | XXXXXX | XXX | xxxxxx | DDMMMYYYY |
| XXXX | XXXX | х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXX | xxxxxx | DDMMMYYYY |

Note:

ARR = Administration-associated reaction.

### LISTING 16.2.6)2. ADVERSE EVENTS

| Patient | Type of<br>Lymphoma | No. | Description | LLT | PΤ | SOC | Start Date (DDMMMYYYY) | SAE | Initial<br>Intensity | AESI | AAR | Extreme<br>Intensity | Relation to<br>Rituximab | Action<br>Taken with<br>Rituximab | Relation to<br>Chemotherapy | Action<br>Taken with<br>Chemotherapy | AE Required<br>Treatment | Outcome | End Date (DDMMMYYYY) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | v | Xxxxxxx | ~~~~ | ~~~~ | ~~~~ | DDMMMYYYY | xxx | vvv | xxx | xxx | xxx | xxxxxx | xxxxxx | xxxxx | xxxxxx | xxx | xxxxxx | DDMMMYYYY |
| AAAA | AAAA | ^ | | | | | | ^^^ | AAA | 222 | ^^^ | AAA | ^^^^ | ^^^^ | ^^^^ | ΑΛΛΑΛΑ | ^^^ | AAAAAA | |
| XXXX | XXXX | X | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY |
| XXXX | XXXX | Х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY |
| XXXX | XXXX | Х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxx | XXXXXX | DDMMMYYYY |

Note:

ARR = Administration-associated reaction.

### LISTING 16.2.6)3. SERIOUS ADVERSE EVENTS

| Patient | Type of<br>Lymphoma | No. | Description | n LLT | PT | SOC | Start Date (DDMMMYYYY) | SAE | Initial<br>Intensity | AESI | AAR | Extreme<br>Intensity | Relation to<br>Rituximab | Action<br>Taken with<br>Rituximab | Relation to<br>Chemotherapy | Action<br>Taken with<br>Chemotherapy | AE Required<br>Treatment | Outcome | End Date (DDMMMYYYY) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXXX | Х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY |
| XXXX | XXXX | Х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | xxxxxx | DDMMMYYYY |
| XXXX | XXXX | Х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | xxxxxx | DDMMMYYYY |
| xxxx | xxxx | Х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | xxxxxx | xxxxxx | xxxxxx | xxxxxx | XXX | XXXXXX | DDMMMYYYY |

Note:

ARR = Administration-associated reaction.

## LISTING 16.2.6)4. ADVERSE EVENTS OF SPECIAL INTEREST (AESI)

| Patient | Type of<br>Lymphoma | No. | Description | LLT | PT | SOC | Start Date (DDMMMYYYY) | SAE | Initial<br>Intensity | AESI | AAR | Extreme<br>Intensity | Relation to<br>Rituximab | Action<br>Taken with<br>Rituximab | Relation to<br>Chemotherapy | Action<br>Taken with<br>Chemotherapy | AE Required<br>Treatment | Outcome | End Date (DDMMMYYYY) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | ** | | | | DDIAGGGGG | | | | | | | | | | | | DDIAGONIN |
| XXXX | XXXX | X | Xxxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY |
| XXXX | XXXX | Х | XxxxxxX | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY |
| XXXX | XXXX | Х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY |
| xxxx | xxxx | Х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | xxxxxx | xxxxxx | XXXXXX | XXXXXX | xxx | xxxxxx | DDMMMYYYY |

Note:

ARR = Administration-associated reaction.

LISTING 16.2.6)5. ADMINISTERED ASSOCIATED REACTIONS

| Patient Type of No. | . Description | n LLT | PT | SOC Start Date (DDMMMYYYY) | SAE | Initial<br>Intensity | AESI | AAR | Extreme<br>Intensity | Relation to<br>Rituximab | Taken with<br>Rituximab | Relation to<br>Chemotherapy | Action<br>Taken with<br>Chemotherapy | AE Required<br>Treatment | Outcome | End Date (DDMMMYYYY) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx xxxx x<br>xxxx xxxx x | Xxxxxx<br>Xxxxxx | xxxx | xxxx | xxxx DDMMMYYYY<br>xxxx DDMMMYYYY | | xxx<br>xxx | xxx | | | xxxxx | xxxxx<br>xxxxx | xxxxxx | xxxxxx | xxx<br>xxx | xxxxxx | DDMMMYYYY<br>DDMMMYYYY |
| XXXX XXXX X | Xxxxxxx | XXXX | XXXX | xxxx DDMMMYYYY<br>xxxx DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY<br>DDMMMYYYY |

ARR = Administration-associated reaction.

# LISTING 16.2.6)6. GRADE 3+ ADVERSE EVENTS

| Patient | Type of<br>Lymphoma | No. | Description | LLT | PT | SOC | Start Date (DDMMMYYYY) | SAE | Initial<br>Intensity | AESI | AAR | Extreme<br>Intensity | Relation to<br>Rituximab | Action<br>Taken with<br>Rituximab | Relation to<br>Chemotherapy | Action<br>Taken with<br>Chemotherapy | AE Required<br>Treatment | Outcome | End Date (DDMMMYYYY) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | ** | | | | DDIAGGGGG | | | | | | | | | | | | DDIAGONIN |
| XXXX | XXXX | X | Xxxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY |
| XXXX | XXXX | Х | XxxxxxX | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY |
| XXXX | XXXX | Х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY |
| xxxx | xxxx | Х | Xxxxxx | XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | xxxxxx | xxxxxx | XXXXXX | XXXXXX | xxx | xxxxxx | DDMMMYYYY |

Note:

ARR = Administration-associated reaction.

LISTING 16.2.6)7. ADVERSE EVENTS LEADING TO RITUXIMAB DRUG INTERRUPTION OR DRUG DELAYED

| Patient Type of No. | . Description | n LLT | PT | SOC Start Date (DDMMMYYYY) | SAE | Initial<br>Intensity | AESI | AAR | Extreme<br>Intensity | Relation to<br>Rituximab | Taken with<br>Rituximab | Relation to<br>Chemotherapy | Action<br>Taken with<br>Chemotherapy | AE Required<br>Treatment | Outcome | End Date (DDMMMYYYY) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx xxxx x<br>xxxx xxxx x | Xxxxxx<br>Xxxxxx | xxxx | xxxx | xxxx DDMMMYYYY<br>xxxx DDMMMYYYY | | xxx<br>xxx | xxx | | | xxxxx | xxxxx<br>xxxxx | xxxxxx | xxxxxx | xxx<br>xxx | xxxxxx | DDMMMYYYY<br>DDMMMYYYY |
| XXXX XXXX X | Xxxxxxx | XXXX | XXXX | xxxx DDMMMYYYY<br>xxxx DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY<br>DDMMMYYYY |

ARR = Administration-associated reaction.

LISTING 16.2.6)8. ADVERSE EVENTS LEADING TO CHEMOTHERAPY DOSE MODIFICATION

| Patient | Type of<br>Lymphoma | No. | Description | LLT | PT | SOC | Start Date (DDMMMYYYY) | SAE | Initial<br>Intensity | AESI | AAR | Extreme<br>Intensity | Relation to<br>Rituximab | Action<br>Taken with<br>Rituximab | Relation to<br>Chemotherapy | Action<br>Taken with<br>Chemotherapy | AE Required<br>Treatment | Outcome | End Date (DDMMMYYYY) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | xxxx | x | Xxxxxxx | xxxx | xxxx | | DDMMMYYYY<br>DDMMMYYYY | xxx | | | | | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxx | xxxxx | DDMMMYYYY<br>DDMMMYYYY |
| xxxx | XXXX<br>XXXX | X<br>X | Xxxxxxx<br>Xxxxxxx<br>Xxxxxxx | XXXX | XXXX | xxxx | DDMMMYYYY<br>DDMMMYYYY | XXX | XXX | XXX | | XXX | xxxxxx<br>xxxxxx | xxxxxx<br>xxxxxx | xxxxxx<br>xxxxxx | XXXXXX<br>XXXXXX | XXX<br>XXX | XXXXXX | DDMMMYYYY<br>DDMMMYYYY |

ARR = Administration-associated reaction.

LISTING 16.2.6)9. ADVERSE EVENTS LEADING TO CHEMOTHERAPY DISCONTINUATION

| Patient Type of No. | . Description | n LLT | PT | SOC Start Date (DDMMMYYYY) | SAE | Initial<br>Intensity | AESI | AAR | Extreme<br>Intensity | Relation to<br>Rituximab | Taken with<br>Rituximab | Relation to<br>Chemotherapy | Action<br>Taken with<br>Chemotherapy | AE Required<br>Treatment | Outcome | End Date (DDMMMYYYY) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx xxxx x<br>xxxx xxxx x | Xxxxxx<br>Xxxxxx | xxxx | xxxx | xxxx DDMMMYYYY<br>xxxx DDMMMYYYY | | xxx<br>xxx | xxx | | | xxxxx | xxxxx<br>xxxxx | xxxxxx | xxxxxx | xxx<br>xxx | xxxxxx | DDMMMYYYY<br>DDMMMYYYY |
| XXXX XXXX X | Xxxxxxx | XXXX | XXXX | xxxx DDMMMYYYY<br>xxxx DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY<br>DDMMMYYYY |

ARR = Administration-associated reaction.

LISTING 16.2.6)10. ADVERSE EVENTS WITHIN THE MEDDRA SMQ ANAPHYLACTIC REACTIONS

| Patient Type of No. | . Description | n LLT | PT | SOC Start Date (DDMMMYYYY) | SAE | Initial<br>Intensity | AESI | AAR | Extreme<br>Intensity | Relation to<br>Rituximab | Taken with<br>Rituximab | Relation to<br>Chemotherapy | Action<br>Taken with<br>Chemotherapy | AE Required<br>Treatment | Outcome | End Date (DDMMMYYYY) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx xxxx x<br>xxxx xxxx x | Xxxxxx<br>Xxxxxx | xxxx | xxxx | xxxx DDMMMYYYY<br>xxxx DDMMMYYYY | | xxx<br>xxx | xxx | | | xxxxx | xxxxx<br>xxxxx | xxxxxx | xxxxxx | xxx<br>xxx | xxxxxx | DDMMMYYYY<br>DDMMMYYYY |
| XXXX XXXX X | Xxxxxxx | XXXX | XXXX | xxxx DDMMMYYYY<br>xxxx DDMMMYYYY | XXX | XXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY<br>DDMMMYYYY |

ARR = Administration-associated reaction.

LISTING 16.2.6)11. INJECTION SITE REACTIONS

| Patient | Type of<br>Lymphoma | Visit | Was an Infection<br>Assessment Done? | Active<br>Infection | Was a Rituximab SC<br>Injection Site<br>Examination Done? | Date of<br>Assessment | Examination<br>Result |
|---|---|---|---|---|---|---|---|
| xxxx | xxxx | х | Xxxxxxx | xxxx | xxxx | DDMMMYYYY | xxx |
| XXXX | XXXX | x | Xxxxxxx | XXXX | XXXX | DDMMMYYYY | XXX |
| XXXX | XXXX | x | Xxxxxxx | XXXX | XXXX | DDMMMYYYY | XXX |
| xxxx | XXXX | х | Xxxxxxx | XXXX | xxxx | DDMMMYYYY | XXX |

LISTING 16.2.6)12. DEATH

| Patient | Type of<br>Lymphoma | Date of<br>Death | Primary Cause of Death | If cause is AE, was<br>Undelying Cancer a<br>Contributing Factor? | If Other, Specify | Suspected Causal<br>Realationship to<br>Study Medication | Was Autopsy<br>Performed? | If Yes,<br>Summarize<br>Findings |
|---|---|---|---|---|---|---|---|---|
| | | DDIAGGUUU | | | | | | |
| XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |
| XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |
| XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXXXX | XXXXX | XXXXXX | XXXXXX |
| XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |

LISTING 16.2.7.1) HEMATOLOGY

| | | | | | | | | Or | iginal uni | t | | SI |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | Type of<br>Lymphoma | Age<br>(yrs) | Gender | Visit | Collection<br>Date<br>(DDMMMYYYY) | Parameter | Value | NRLL | NRUL | Reference to<br>Normal Range | Value | Unit |
| XXXX | XXXX | XXXX | XXXX | XXXX | DDMMMYYYY | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | DDIAAAAAAA | | | | | | | |
| | | XXXX | XXXX | XXXX | DDMMMYYYY | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | DDMMWWW | | | | | | | |
| | | XXXX | XXXX | XXXX | DDMMMYYYY | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | DDMMMYYYY | | | | | | | |
| XXXX | XXXX | XXXX | XXXX | XXXX | DDMMMIII | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |

NRLL: Normal range lower limit. NRUL: Normal range upper limit.

LISTING 16.2.7.2) BIOCHEMISTRY

| | | | | | | | | Or | iginal uni | t | | SI |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | Type of<br>Lymphoma | Age<br>(yrs) | Gender | Visit | Collection<br>Date<br>(DDMMMYYYY) | Parameter | Value | NRLL | NRUL | Reference to<br>Normal Range | Value | Unit |
| xxxx | xxxx | xxxx | xxxx | xxxx | DDMMMYYYY | xxxxxx | xxxx | xxxx | xxxx | xxxxxx | xxxxxx | xxxxxx |
| ^^^ | ^^^ | **** | ^^^^ | ^^^ | DDMMIIII | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | | xxxxxx | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | xxxxxx |
| | | xxxx | xxxx | xxxx | DDMMMYYYY | xxxxxx | xxxx | xxxx | xxxx | xxxxxx | xxxxxx | xxxxxx |
| | | 212121 | mm | nnn | DDIMMITTI | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | | xxxxxx | XXXX | XXXX | XXXX | xxxxxx | xxxxxx | xxxxxx |
| | | xxxx | xxxx | xxxx | DDMMMYYYY | xxxxxx | xxxx | xxxx | xxxx | xxxxxx | xxxxxx | xxxxxx |
| | | | | | | xxxxxx | xxxx | xxxx | xxxx | XXXXXX | xxxxxx | xxxxxx |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX | XXXXXX | XXXXXX |
| | | | | | | xxxxxx | xxxx | xxxx | xxxx | xxxxxx | xxxxxx | xxxxxx |
| | | | | | | xxxxxx | xxxx | xxxx | xxxx | xxxxxx | xxxxxx | xxxxxx |
| xxxx | xxxx | xxxx | xxxx | xxxx | DDMMMYYYY | xxxxxx | xxxx | xxxx | xxxx | xxxxxx | xxxxxx | xxxxxx |
| | | | | | | xxxxxx | xxxx | xxxx | xxxx | XXXXXX | xxxxxx | xxxxxx |
| | | | | | | xxxxxx | xxxx | xxxx | xxxx | xxxxxx | xxxxxx | xxxxxx |
| | | | | | | xxxxxx | xxxx | xxxx | xxxx | XXXXXX | xxxxxx | xxxxxx |
| | | | | | | xxxxxx | xxxx | xxxx | xxxx | xxxxxx | xxxxxx | xxxxxx |

NRLL: Normal range lower limit. NRUL: Normal range upper limit.

LISTING 16.2.7.3) COAGULATION TESTS

| Patient | Type of<br>Lymphoma | Age<br>(yrs) | Gender | Visit | Collection<br>Date<br>(DDMMMYYYY) | Parameter | Value | NRLL | NRUL | Reference to<br>Normal Range |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | DDMMMYYYY | | | | | |
| XXXX | XXXX | XXXX | XXXX | XXXX | DDMMMIIII | XXXXXX | XXXX | xxxx | xxxx | XXXXXX |
| | | | | | | XXXXXX | XXXX | xxxx | XXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX |
| | | xxxx | xxxx | xxxx | DDMMMYYYY | xxxxxx | xxxx | xxxx | xxxx | xxxxxx |
| | | | ******* | ******* | 22 | XXXXXX | XXXX | xxxx | XXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | xxxx | XXXX | XXXXXX |
| | | | | | | XXXXXX | xxxx | xxxx | xxxx | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX |
| | | | | | | ********** | ******* | ****** | ******* | |
| | | xxxx | xxxx | xxxx | DDMMMYYYY | xxxxxx | xxxx | xxxx | xxxx | xxxxxx |
| | | | | | | XXXXXX | XXXX | xxxx | XXXX | xxxxxx |
| | | | | | | XXXXXX | XXXX | xxxx | XXXX | xxxxxx |
| | | | | | | XXXXXX | XXXX | xxxx | XXXX | xxxxxx |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX |
| XXXX | XXXX | XXXX | XXXX | XXXX | DDMMMYYYY | XXXXXX | XXXX | xxxx | XXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | xxxxxx |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX |
| | | | | | | XXXXXX | XXXX | XXXX | XXXX | XXXXXX |

NRLL: Normal range lower limit. NRUL: Normal range upper limit.

LISTING 16.2.8.1) VITAL SIGNS & BODY WEIGHT

| Patient | Type of<br>Lymphoma | Visit | Was Vital Signs<br>Performed? | Date of<br>Assessment | Pulse<br>(bpm) | SBP<br>(mmHg) | DBP<br>(mmHg) | Body<br>Temperature<br>(°C) | Body<br>Weight<br>(Kg) |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | xxxx | DDMMMYYYY | xxx | xxx | xxx | xxx | xxx |
| | | xxxx | xxxx | DDMMMYYYY | xxx | xxx | xxx | XXX | xxx |
| | | xxxx | xxxx | DDMMMYYYY | xxx | xxx | xxx | XXX | xxx |
| | | XXXX | xxxx | DDMMMYYYY | XXX | XXX | XXX | xxx | xxx |
| xxxx | xxxx | xxxx | xxxx | DDMMMYYYY | xxx | xxx | xxx | xxx | xxx |
| | | xxxx | xxxx | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX |
| | | xxxx | xxxx | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX |
| | | xxxx | xxxx | DDMMMYYYY | XXX | XXX | XXX | XXX | XXX |

LISTING 16.2.8.2) SERUM PREGNANCY TEST

| Patient | Type of<br>Lymphoma | Was Serum<br>Pregnancy Test<br>Performed? | Date of<br>Assessment | Test<br>Result |
|---|---|---|---|---|
| xxxx | xxxx | xxxx | DDMMMYYYY | xxx |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXX |
| XXXX | XXXX | xxxx | DDMMMYYYY | XXX |
| xxxx | xxxx | xxxx | DDMMMYYYY | xxx |
LISTING 16.2.8.3) URINE PREGNANCY TEST

| Patient | Type of<br>Lymphoma | Was Urine<br>Pregnancy Test<br>Performed? | Date of Urine<br>Pregnancy Test | Test Result |
|---|---|---|---|---|
| xxxx | xxxx | xxxx | DDMMMYYYY | xxx |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXX |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXX |
| xxxx | XXXX | xxxx | DDMMMYYYY | XXX |

LISTING 16.2.8.4) PHYSICAL EXAMINATION

| Patient | Type of<br>Lymphoma | Visit | Date of<br>Assessment<br>(DDMMMYYYY) | Body System | Result |
|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | DDMMMYYYY | XXXX<br>XXXX<br>XXXX | xxxx<br>xxxx<br>xxxx |
| xxxx | xxxx | xxxx | DDMMMYYYY | xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx |
| xxxx | xxxx | xxxx | DDMMMYYYY | XXXX<br>XXXX<br>XXXX | XXXX<br>XXXX<br>XXXX |

LISTING 16.2.8.5) 12-LEAD ECG

| Patient | Type of<br>Lymphoma | ECG Performed? | ECG Date<br>(DDMMMYYYY) | ECG Result |
|---|---|---|---|---|
| xxxx | xxxx | xxx | DDMMMYYYY | xxxxxxx |
| XXXX | XXXX | xxx | DDMMMYYYY | xxxxxxx |
| XXXX | XXXX | xxx | DDMMMYYYY | xxxxxxx |
| XXXX | XXXX | xxx | DDMMMYYYY | xxxxxxx |

LISTING 16.2.8.6) TARGET LESION ASSESSMENT AT SCREENING (PART #1)

| Patient | Type of<br>Lymphoma | Were Target<br>Lesions<br>Identified? | Location | If Other,<br>Specify | CT with<br>Contrast | Date of<br>CT Scan | CT Scan<br>Result | CT w/o<br>Contrast | Date of CT<br>Scan | Result | MRI | Date of<br>MRI | MRI<br>Result |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | xxxx | xxxx | xxxx | DDMMMYYYY | xxxx | xxxx | DDMMMYYYY | xxx | xxx | DDMMMYYYY | xxx |
| xxxx | xxxx | xxxx | xxxx | xxxx | xxxx | DDMMMYYYY | xxxx | xxxx | DDMMMYYYY | xxx | xxx | DDMMMYYYY | xxx |
| xxxx | XXXX | XXXX | XXXX | XXXX | XXXX | DDMMMYYYY | XXXX | XXXX | DDMMMYYYY | XXX | xxx | DDMMMYYYY | XXX |
| xxxx | XXXX | XXXX | XXXX | XXXX | XXXX | DDMMMYYYY | XXXX | XXXX | DDMMMYYYY | XXX | xxx | DDMMMYYYY | XXX |

LISTING 16.2.8.7) TARGET LESION ASSESSMENT AT SCREENING (PART #2)

| Patient | Type of<br>Lymphoma | Clinical<br>Assessment? | Date of<br>Assessment | Result | FDG-PET | Date of<br>Scan | Result | Other | If Other, Specify | Date of<br>Scan | Result |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | XXX<br>XXX<br>XXX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | xxx<br>xxx<br>xxx<br>xxx |

LISTING 16.2.8.8) TARGET LESION ASSESSMENT SUBSEQUENT (PART #1)

| Patient | Type of<br>Lymphoma | Visit | Were Any<br>Changes? | Location | If Other,<br>Specify | CT with<br>Contrast | Date of<br>CT Scan | CT Scan<br>Result | CT w/o<br>Contrast | Date of<br>CT Scan | Result | MRI | Date of<br>MRI | MRI<br>Result |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | ****<br>**** | xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | xxx<br>xxx<br>xxx |

LISTING 16.2.8.9) TARGET LESION ASSESSMENT SUBSEQUENT (PART #2)

| Patient | Type of<br>Lymphoma | Clinical<br>Assessment? | Date of<br>Assessment | Result | FDG-PET | Date of<br>Scan | Result | Other | If Other, Specify | Date of<br>Scan | Result | Change in Lesion Since<br>First Assessed or<br>Previous Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | DDMMMYYYY | xxxx | xxxx | DDMMMYYYY | xxxx | xxxx | xxx | DDMMMYYYY | xxx | xxx |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXXX | XXXX | DDMMMYYYY | XXXX | XXXX | XXX | DDMMMYYYY | XXX | XXX |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXXX | XXXX | DDMMMYYYY | XXXX | XXXX | xxx | DDMMMYYYY | XXX | xxx |
| XXXX | XXXX | XXXX | DDMMMYYYY | xxxx | XXXX | DDMMMYYYY | xxxx | xxxx | xxx | DDMMMYYYY | XXX | xxx |

LISTING 16.2.8.10) OVERALL LESION ASSESSMENT

| Patient | Type of<br>Lymphoma | Date<br>of Assessment | Response of Target<br>Lesions | New<br>Lesions? | Inv.'s Overall Assessment<br>of Response at This Visit | Date of<br>Progression |
|---|---|---|---|---|---|---|
| xxxx | xxxx | DDMMMYYYY | xxxx | xxx | XXX | DDMMMYYYY |
| xxxx | XXXX | DDMMMYYYY | xxxx | XXX | xxx | DDMMMYYYY |
| XXXX | XXXX | DDMMMYYYY | xxxx | XXX | xxx | DDMMMYYYY |
| XXXX | XXXX | DDMMMYYYY | xxxx | XXX | xxx | DDMMMYYYY |

LISTING 16.2.8.11) SURVIVAL STATUS

| Patient | Type of<br>Lymphoma | Was Survival<br>Assessment<br>Performed? | Date of<br>Assessment | Survival<br>Status | Date of Last<br>Contact | Has the Patient Started<br>New Lymphoma Treatment<br>Since Last Contact? | Start Date |
|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | DDMMMYYYY | xxx | DDMMMYYYY | xxx | DDMMMYYYY |
| xxxx | XXXX | XXXX | DDMMMYYYY | XXX | DDMMMYYYY | xxx | DDMMMYYYY |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXX | DDMMMYYYY | xxx | DDMMMYYYY |
| xxxx | xxxx | XXXX | DDMMMYYYY | XXX | DDMMMYYYY | xxx | DDMMMYYYY |

LISTING 16.2.8.12) BONE MARROW ASSESSMENT

| Patient | Type of<br>Lymphoma | Was Bone Marrow<br>Assesment Done? | Date of BM assessment | Was BM Assessment<br>Done Using Aspirate? | Result | Was BM Assessment<br>Done Using Biopsy? | Result |
|---|---|---|---|---|---|---|---|
| xxxx | xxxx | x | DDMMMYYYY | xxxxx | xxxxx | xxxxx | xxxxx |
| XXXX | XXXX | x | DDMMMYYYY | xxxxx | XXXXX | xxxxx | XXXXX |
| XXXX | XXXX | x | DDMMMYYYY | xxxxx | XXXXX | xxxxx | XXXXX |
| xxxx | XXXX | x | DDMMMYYYY | xxxxx | XXXXX | xxxxx | XXXXX |

LISTING 16.2.8.13) RASQ FOR IV ADMINISTRATION

| Patient | Type of<br>Lymphoma | Was RASQ<br>Completed? | Date of<br>Assessment | Item #1 | Item 1a | | Item 20 | Physical<br>impact<br>domain<br>value | Psychological impact domain value | Impact or<br>ADL<br>Domain<br>value | | Satisfaction<br>Domain<br>value |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx |

LISTING 16.2.8.14) RASQ FOR SC ADMINISTRATION

| | | _ | Date of<br>Assessment | Item #1 | Item 1a | • • | Item 20 | Physical<br>impact<br>domain<br>value | Psychological impact domain value | Impact or<br>ADL<br>Domain<br>value | | Satisfaction<br>Domain<br>value |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| **** *** **** *** **** *** | x 2 | xxxx<br>xxxx<br>xxxx | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | XXX<br>XXX<br>XXX | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx | XXX<br>XXX<br>XXX | xxx<br>xxx<br>xxx<br>xxx | xxx<br>xxx<br>xxx<br>xxx |

LISTING 16.2.8.15) HEALTHCARE PROFESSIONAL QUESTIONNAIRE

| Site | Healthcare<br>professional | Was HPQ<br>Completed? | Date of<br>Assessment | Item #1 | Item 1a | | Item 10 |
|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | DDMMMYYYY | xxx | xxx | xxx | xxx |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX |
| XXXX | XXXX | XXXX | DDMMMYYYY | XXX | XXX | XXX | XXX |